

**Statistical Analysis Plan** Arcutis Biotherapeutics, Inc. ARQ-151-202

Version: 1 Date: 22OCT2020

# STATISTICAL ANALYSIS PLAN

| Protocol Number: | ARQ-151-202 |
|---|---|
| Study Title: | A Phase 2, Multicenter, Open-Label Extension Study of the Long-Term Safety of ARQ-151 Cream 0.3% in Adult Subjects with Chronic Plaque Psoriasis who have Completed Preceding Study ARQ-151-201 Phase 2 Randomized Controlled Trial (Cohort 1) and non-ARQ-151-201 Subjects (Cohort 2) |
| Development Phase of Study: | Phase 2 |
| Sponsor: | Arcutis Biotherapeutics, Inc.<br>2945 Townsgate Road, Suite 110<br>Westlake Village, CA 91361<br>USA |
| Sponsor Contact: | |
| Statistical Analysis Plan based on Protocol Version: | Version 1.0 Amendment 1, 25 March 2019 |
| Statistical Analysis Plan Date:<br>Statistical Analysis Plan Version: | 22OCT2020<br>Version 1 |



Arcutis Biotherapeutics, Inc. ARQ-151-202




Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.



**Statistical Analysis Plan** Arcutis Biotherapeutics, Inc. ARQ-151-202


# SAP Change History

| Version | Date | Summary of Changes | Author |
|---------|-------------|--------------------|--------|
| 1 | 22 OCT 2020 | Original document | |



Statistical Analysis Plan Arcutis Biotherapeutics, Inc. ARQ-151-202


# **TABLE OF CONTENTS**

| 1. | LIS | T OF A | BBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
|---|---|---|---|---|
| 2. | INT | TRODU( | CTION | 6 |
| 3. | STU | U <b>DY O</b> B | BJECTIVES | 7 |
| 4. | STUDY DESIGN | | | |
| | 4.1 | Overal | 1 Study Design | 8 |
| | | 4.1.1 | Schedule of Visits and Assessments | 8 |
| | | 4.1.2 | Method of Assigning Subjects to Treatment Groups | 8 |
| | | 4.1.3 | Blinding | |
| 5. | EFI | FICACY | Y AND SAFETY ENDPOINTS | 8 |
| | 5.1 | Safety | Endpoints | 8 |
| | 5.2 | Efficac | ey Endpoints | 9 |
| 6. | STA | ATISTIC | CAL AND ANALYTICAL PLANS | 11 |
| | 6.1 | Genera | al Methodology | 11 |
| | | 6.1.1 | Statistical Analysis | 11 |
| | | 6.1.2 | Baseline Definition | 11 |
| | | 6.1.3 | Visit Windowing | 12 |
| | | 6.1.4 | Adjustments for Covariates | 12 |
| | | 6.1.5 | Handling of Dropouts or Missing Data | 12 |
| | | 6.1.6 | Interim Analyses and Data Monitoring | 12 |
| | | 6.1.7 | Multicenter Studies | 13 |
| | | 6.1.8 | Multiple Comparisons/Multiplicity | 13 |
| | | 6.1.9 | Use of an Efficacy Subset of Subjects | 13 |
| | | 6.1.10 | Active-Control Studies Intended to Show Equivalence | 13 |
| | | 6.1.11 | Examination of Subgroups | 13 |
| | 6.2 | Dispos | ition of Subjects | 13 |
| | 6.3 | Protoco | ol Deviations | 13 |
| | 6.4 | Data S | ets Analyzed | 13 |
| | | 6.4.1 | Safety Population | 13 |
| | 6.5 | Demog | graphic and Other Baseline Characteristics | 14 |
| | 6.6 | Prior a | nd Concomitant Medications | 14 |
| | 6.7 | Analys | sis of Efficacy | 14 |



Statistical Analysis Plan Arcutis Biotherapeutics, Inc. ARQ-151-202

| | 6.8 | Safety | Evaluation | | 15 |
|---|---|---|---|---|---|
| | | 6.8.1 | | Exposure | |
| | | 6.8.2 | Adverse 1 | Events | 15 |
| | | 6.8.3 | Clinical I | Laboratory Evaluation | 16 |
| | | 6.8.4 | | servations Related to Safety | |
| | | | 6.8.4.1 | 12-Lead Electrocardiogram Measurements | 16 |
| | | | 6.8.4.2 | Vital Signs | |
| | | | 6.8.4.3 | Physical Examination | 17 |
| | | | 6.8.4.4 | Local Tolerance Assessments | |
| | | | 6.8.4.5 | Patient Health Questionnaire Depression Scale | 1′ |
| | | | 6.8.4.6 | Columbia-Suicide Severity Rating Scale | 17 |
| | | | 6.8.4.7 | Prior and Concomitant Medication | |
| 7. | DE | ΓERMI | NATION ( | OF SAMPLE SIZE | 18 |
| 8. | CH | ANGES | IN THE I | PLANNED ANALYSES | 18 |
| 9. | RE | FEREN | CES | | 20 |
| 10. | IND | EX OF | PLANNE | D TABLES | <b>2</b> 1 |
| 11. | INE | EX OF | ' PLANNE | D LISTINGS | 302 |



Arcutis Biotherapeutics, Inc. ARQ-151-202

Version: 1

Date: 22OCT2020

#### 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE(s) adverse event(s)

ATC anatomical therapeutic chemical

cm centimeters

C-SSRS Columbia-Suicide Severity Rating Scale

ECG electrocardiogram

IGA Investigator Global Assessment

I-IGA Intertriginous Investigator Global Assessment

kg kilograms max maximum

MedDRA Medical Dictionary for Regulatory Activities

min minimum

mPASI Modified Psoriasis Area Severity Index

mPASI-75 75% reduction from Baseline of Modified Psoriasis Area Severity Index

n number of observations

N number of subjects (sample size)

PASI-50 50% reduction from Baseline of Psoriasis Area Severity Index PASI-75 75% reduction from Baseline of Psoriasis Area Severity Index

PHQ-8 Patient Health Questionnaire Depression Scale

QST QST Consultations, Ltd. SAE(s) serious adverse event(s)

SAS® Statistical Analysis System (SAS® Institute Inc., Cary, NC)

SD standard deviation SOC system organ class

TEAE(s) treatment-emergent adverse event(s)

US United States

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

#### 2. INTRODUCTION

Roflumilast is a phosphodiesterase 4 (PDE-4) inhibitor approved globally to reduce the risk of exacerbations in patients with severe chronic obstructive pulmonary disease (COPD) associated with chronic bronchitis. Roflumilast and its active metabolite, roflumilast N-oxide, are high



Arcutis Biotherapeutics, Inc. ARQ-151-202


affinity selective inhibitors of PDE-4 (a major cyclic-3',5'-adenosine monophosphate (cyclic AMP)-metabolizing enzyme), whose activity leads to accumulation of intracellular cyclic AMP.

There are four different subtypes of PDE-4: PDE-4a, PDE-4b, PDE-4c, and PDE-4d, each with several isoforms (splicing variants). IC<sub>50</sub> values of both roflumilast and roflumilast N-oxide for the different PDE-4 isoforms and subtypes are mostly sub-nanomolar and single digit nanomolar (Hatzelmann 2010). The PDE-4 family of enzymes are the most prevalent phosphodiesterases in immune cells and inhibition of PDE-4 subtypes has been associated with anti-inflammatory effects in many biological systems.

Psoriasis is a chronic inflammatory skin disease characterized by raised, well-demarcated, erythematous oval plaques with adherent silvery scales. Numerous past reports have suggested a deficiency of cyclic AMP-dependent protein kinases in human psoriatic skin (Brion 1986). More recently, various cytokines produced by Th1 and Th17 cells have been shown to play a crucial role in the pathogenesis of psoriasis. It has been postulated that the anti-inflammatory effects of PDE-4 inhibitors may provide a beneficial therapeutic intervention in the treatment of chronic plaque psoriasis and recently Otezla® (apremilast), a PDE-4 inhibitor, has been approved for the oral treatment of chronic plaque psoriasis.

The past 15 years have witnessed a transformation in the systemic treatment of moderate to severe psoriasis with the advent of biological therapies. However, for patients with milder forms of disease, best treated with topical options, the therapeutic landscape really has not changed in several decades. Topical steroids come in all shapes and forms, but the lower potency steroids are not effective and the higher potency steroids are beset with issues of local skin atrophy and the potential for hypothalamic-pituitary axis suppression when applied over larger body surface areas and for prolonged periods of time. Vitamin D has been the other staple of topical psoriasis treatment but it is irritating, not suitable for use on the face or intertriginous areas, and its efficacy is rather modest. Hence, there is substantial medical need for additional topical approaches in the treatment of psoriasis. The study sponsor is developing a topical formulation of roflumilast for the treatment of chronic plaque psoriasis. Our Phase 2a results suggest that ARQ-151 may be a highly efficacious and well-tolerated topical treatment for psoriasis.

#### 3. STUDY OBJECTIVES

The objective of this study is to assess long-term safety in a multicenter, open-label, 52-week study in subjects treated with ARQ-151 cream 0.3% after completing a 12-week Phase 2b study (ARQ-151-201) Cohort 1 and non ARQ-151-201 subjects (Cohort 2).



Arcutis Biotherapeutics, Inc. ARQ-151-202


#### 4. STUDY DESIGN

### 4.1 Overall Study Design

This is an open-label, long-term safety study of ARQ-151 cream 0.3% in subjects with chronic plaque psoriasis involving between 0 and 25% BSA. Eligible subjects will enroll into the long-term safety study on the same day as the Week 12 visit for the previous study (ARQ-151-201) for Cohort 1 and on Day 1 for non ARQ-151-201 subjects in Cohort 2. Study medication will be applied by the subjects topically once a day for 52 weeks at home.

A total of up to approximately 300 subjects (Cohort 1) and up to approximately 100 non ARQ-151-201 subjects (Cohort 2) will be enrolled at approximately 30 study sites in the United States and Canada. Subjects will be adult (≥18 y/o) males or females with chronic plaque psoriasis. Periodic clinic visits will include assessments for clinical safety, application site reactions evaluated in the clinic using the method of Berger and Bowman (Berger-1982), disease improvement or progression, and investigator global assessment (IGA).

#### 4.1.1 Schedule of Visits and Assessments

The schedule of assessments can be found in Section 5 of the protocol.

# 4.1.2 Method of Assigning Subjects to Treatment Groups

This is an open-label single-arm study. Eligible subjects will receive ARQ-151 cream 0.3%.

#### 4.1.3 Blinding

Not applicable.

#### 5. EFFICACY AND SAFETY ENDPOINTS

#### 5.1 Safety Endpoints

The primary endpoint will be analysis of safety monitored through application site assessments in the clinic using the method of Berger and Bowman, clinical laboratory testing, 12-lead electrocardiograms (ECGs), Patient Health Questionnaire Depression Scale (PHQ-8), Columbia-Suicide Severity Rating Scale (C-SSRS) and adverse events (AEs). Two primary endpoint analyses are planned:

- Occurrence of treatment emergent AEs (TEAEs)
- Occurrence of Serious Adverse Events (SAEs)



Arcutis Biotherapeutics, Inc. ARQ-151-202


Additionally a set of secondary endpoints will be summarized. These include:

- Changes in PHQ-8, C-SSRS, ECG, clinical laboratory parameters, and vital signs over time.
- Incidence of 5% of weight loss or gain from baseline.
- Incidence of shifts from baseline to last, highest and lowest BMI category.
- Incidence of application site reactions assessed by the investigator.

# **5.2** Efficacy Endpoints

The secondary endpoints are related to efficacy and will include:

- Proportion (%) of subjects achieving an IGA of clear or almost clear, as observed at Week 4, 12, 24, 36, and 52.
- In subjects who achieve 'Clear' scores for IGA, Intertriginous IGA (I-IGA) (if applicable and Modified Psoriasis Area Severity Index (mPASI)) and stop treatment to all lesions, time to restarting study drug (treatment free interval). Subjects with continual clearance will be censored at their date of last contact.
- The incidence of subjects who stop therapy during the study due to disease clearance on study. Disease clearance is defined as 'Clear' scores for IGA, I-IGA (if applicable and mPASI).
- Proportion (%) of applicable subjects with intertriginous area involvement, 'I-IGA' score of 'Clear' or 'Almost Clear' at Week 4, 12, 24, 36, and 52.
- Proportion (%) of subjects achieving a 75% reduction from Baseline of PASI (PASI-75) at Week 4, 12, 24, 36, and 52. PASI was not specifically collected but will be derived based on already reported information.
- Proportion (%) of subjects achieving a 75% reduction from Baseline of mPASI (mPASI-75) at Week 4, 12, 24, 36, and 52.
- Proportion of subjects (%) with a 2-grade improvement in IGA from Baseline as observed at Weeks 4, 12, 24, 36, 52.
- Proportion of subjects (%) with IGA Success, defined as achievement of an IGA of 'Clear' or 'Almost Clear' plus a 2-grade improvement in IGA from Baseline as observed at Weeks 4, 12, 24, 36, and 52.



Arcutis Biotherapeutics, Inc. ARQ-151-202

- Duration of IGA Success, defined as the time from the first observation of IGA Success
  to the first subsequent time a subject's disease response does not meet the criteria for
  IGA Success. The duration of IGA Success for subjects who end treatment in IGA
  Success will be censored at the last disease assessment date.
- Duration of IGA Clear or Almost Clear, defined as the time from the first observation of IGA Clear or Almost Clear to the first subsequent time a subject's disease response is not Clear or Almost Clear. The duration of IGA Clear or Almost Clear for subjects who end treatment with IGA Clear or Almost Clear will be censored at the last disease assessment date.
- Duration of PASI-50, defined as the time from the first observation of a 50% reduction from Baseline in the PASI to the first subsequent time a subject's PASI score is greater than a 50% reduction from Baseline. The duration of PASI-50 for subjects who end treatment with PASI score at least 50% less than Baseline will be censored at the last disease assessment date.
- Duration of PASI-75, defined analogously to duration of PASI-50
- Percent change from baseline in PASI score at each disease assessment
- Shift from the baseline IGA score to the last reported IGA score on study
- Frequency of disease recurrence among subjects who stop therapy due to disease clearance. Disease recurrence is defined as any instance where IGA is ≥ 2 or mPASI is greater than 0.
- Time to disease recurrence among subjects who stop therapy due to disease clearance. Time to disease recurrence is defined as the time from the last dose of ARQ-151 to the first observation of an IGA score of 2 or greater. The time to disease recurrence among subjects with clearance at the end of the study observation period will be censored at the last observed disease assessment
- The incidence of disease control among subjects who restart therapy after having stopped therapy due to disease clearance. Disease control is defined as achieving an IGA score of 0 or 1 subsequent to restarting study therapy.
- Time to disease control among subjects who restart therapy after having stopped therapy due to disease clearance. Time to disease control is the time from the restart of therapy to the first reported IGA score of 0 or 1. The time to disease control among subjects who do not achieve an IGA score of 0 or 1 by the end of the study observation period will be censored at the last observed disease assessment.



Arcutis Biotherapeutics, Inc. ARQ-151-202


#### 6. STATISTICAL AND ANALYTICAL PLANS

# 6.1 General Methodology

All statistical processing will be performed using SAS® (Version 9.4 or later) unless otherwise stated.

Descriptive statistics will be used to provide an overview of the safety and efficacy results. For categorical parameters, the number and percentage of subjects in each category will be presented. The denominator for percentage will be based on the number of subjects appropriate for the purpose of analysis. For continuous parameters, descriptive statistics will include number of subjects (n), mean, standard deviation (SD), median, minimum (min), and maximum (max).

Reported AEs, medical history terms and prior and concomitant procedures and therapies will be classified on the basis of Medical Dictionary for Regulatory Activities (MedDRA) terminology. Prior and concomitant medications will be classified on the basis of World Health Organization Drug Dictionary (WHO-DD) terminology.

### 6.1.1 Statistical Analysis

All analyses outlined herein will be performed by QST Consultations, Ltd. (QST), utilizing SAS® Version 9.4 or later. All summary tables and data listings will be prepared utilizing SAS® software.

The standard operating procedures (SOPs) of QST, will be followed in the creation and quality control of all data displays and analyses described in this SAP.

#### **6.1.2** Baseline Definition

For subjects in Cohort 1, the baseline value for safety and efficacy parameters will be defined as the last observation prior to the first dose of ARQ-151 cream in either the ARQ-151-201 study or this study. Sensitivity analyses of efficacy will be performed where the baseline value for subjects in Cohort 1 is defined as the last observation prior to the first dose of ARQ-151 0.3% cream in this study. For the purpose of these latter analyses, study procedures will not be repeated; the information from the ARQ-151-201 study Week 12 visit will be carried over to the Day 1 visit for this study.

For subjects in Cohort 2, baseline values for efficacy and safety will be defined as the last observation prior to the first dose of ARQ-151 cream 0.3% in this study. Baseline values will most commonly be from Day 1.



Arcutis Biotherapeutics, Inc. ARQ-151-202


# 6.1.3 Visit Windowing

Data will be summarized based on nominal visit indications with the exception of data captured at early termination and unscheduled visits. Data from early termination and unscheduled visits will be mapped to the most appropriate visit values based on the midpoints between scheduled visits. The analysis windows for early termination and unscheduled visits are presented in the following table.

**Analysis Windows for Efficacy and Safety Assessments** 

| Scheduled Visit | Target Study Day | Window (Days) |
|-----------------|------------------|---------------|
| Week 4 | 29 | 15 to 57 |
| Week 12 | 85 | 58 to 127 |
| Week 24 | 169 | 128 to 211 |
| Week 36 | 253 | 212 to 309 |
| Week 52 | 365 | >= 310 |

Data collected at early termination and unscheduled visits prior to study day 15 will not be analyzed, with the exception of those identified as baseline values.

For Cohort 1 subjects that were on the ARQ-151 cream 0.15% or ARQ-151 cream 0.3% arm in the Phase 2b Study (ARQ-151-201), efficacy summaries will be presented for the ARQ-151-201 visits as defined in ARQ-151-201 SAP.

For time to event analysis, no visit windowing will be done. The real study day will be used and all assessments will be eligible for analysis.

## 6.1.4 Adjustments for Covariates

No covariates are planned for this study.

#### 6.1.5 Handling of Dropouts or Missing Data

Missing data will not be imputed.

#### 6.1.6 Interim Analyses and Data Monitoring

No interim inferential analysis or data monitoring is planned for this study.



Arcutis Biotherapeutics, Inc. ARQ-151-202


#### **6.1.7** Multicenter Studies

The clinical study will be conducted under a common protocol for each investigational site with the intention of pooling the data for analysis. Every effort will be made to promote consistency in study execution at each investigational site.

#### 6.1.8 Multiple Comparisons/Multiplicity

No inferential statistical analyses are planned.

#### 6.1.9 Use of an Efficacy Subset of Subjects

No subset of subjects will be used for efficacy.

#### 6.1.10 Active-Control Studies Intended to Show Equivalence

Not applicable to this study.

#### 6.1.11 Examination of Subgroups

Summaries will be presented for the safety based on previous treatment in ARQ-151-201, and a combined ARQ-151-201 group. Additionally summaries will be presented for a complement set of subjects that did not previously participate in ARQ-151-201.

#### 6.2 Disposition of Subjects

The number of subjects included in the safety population will be summarized by previous treatment group and cohort. The number of subjects enrolled, completed, discontinued (including the reasons for discontinuation), and duration of participation (weeks) will be also be summarized. Duration of participation (weeks) is defined as (last contact date – date of first dose in ARQ-151-202 + 1) / 7.

#### **6.3** Protocol Deviations

All protocol deviations that occur will be documented and reported to Arcutis Biotherapeutics Inc.

## 6.4 Data Sets Analyzed

#### **6.4.1** Safety Population

All subjects who are enrolled and received at least one confirmed dose of ARQ-151 cream 0.15% or ARQ-151 cream 0.3% study medication in either the Phase 2b Study (ARQ-151-201) TOOL.ST.101-01.02 Statistical Analysis Plan Template




Arcutis Biotherapeutics, Inc. ARQ-151-202


or this extension study. The number of patients included in the safety population will be summarized. All analyses will be performed using the safety population.

#### 6.5 Demographic and Other Baseline Characteristics

All baseline summaries will be done on the safety population.

Sex, race, and ethnicity will be summarized by counts and percentages. Age (years) will be summarized with descriptive statistics.

IGA, I-IGA, BSA, PASI, mPASI, Height, and Weight, will be summarized at baseline with descriptive statistics.

Past/coexistent medical history information and physical examination observations and vital signs information for all subjects will be presented in a by-subject listing.

#### 6.6 Prior and Concomitant Medications

Prior and concomitant medication information for all subjects will be presented in a by-subject listing. Summary tables will be presented by World Health Organization-Anatomical Therapeutic Chemical Classification System (WHO-ATC) therapeutic category and product.

A by-subject listing of all prior and concomitant medications will be presented.

## 6.7 Analysis of Efficacy

This study is not intended to assess efficacy, but rather the IGA, I-IGA, PASI and mPASI are included to determine the need for treatment and subsequent re-treatment after treatment course in Study ARQ-151-201 or Study ARQ-151-202. Certain efficacy data and endpoints will, however, be summarized. Descriptive statistics will be used to summarize the assessment of efficacy. IGA scores will be summarized at Baseline and every scheduled visit through end of the study (Day 1 and Weeks 4, 12, 24, 36, and 52). The efficacy variable in this study is success in IGA of disease severity, defined as an IGA of 'Clear' or 'Almost Clear'. The number and percentage of patients who achieve treatment success at the scheduled study visits will be tabulated. The proportion of successes for the secondary variables of IGA, I-IGA, PASI-75 and mPASI-75 will be tabulated in a similar manner.

In subjects who achieve 'Clear' scores for IGA, I-IGA (if applicable) and mPASI (if applicable) and stop treatment to all lesions, time to restarting study drug (treatment free interval) will be calculated and analyzed. For Cohort 2 and rollover subjects previously treated with Vehicle Cream, the treatment free interval will be the number of weeks between the end of the initial



Arcutis Biotherapeutics, Inc. ARQ-151-202


treatment in study ARQ-151-202 and the start of the next treatment in study ARQ-151-202 if one should be needed or the end of the subject's participation in study ARQ-151-202. In the event that the subject's participation in the study ends without a second round of treatment, subjects will be censored at last observed disease assessment. For rollover subjects previously treated with ARQ-151 cream 0.3% or ARQ-151 cream 0.15%, the treatment free interval will be the number of days between the last treatment that began in Study ARQ-151-201 and the start of the next treatment in study ARQ-151-202 if one should be needed or the last observed disease assessment in the study ARQ-151-202. Subjects who were lost to follow up will be included using all available information. The duration of IGA success, PASI-50, PASI-75, time to disease recurrence, time to disease control will be calculated in the same manner.

The median time (number of weeks) for duration summaries will be analyzed using the Kaplan–Meier method and will be accompanied with a plot. Patients who discontinue study ARQ-151-202 without achieving the event of interest will be considered censored in the Kaplan–Meier analyses.

#### 6.8 Safety Evaluation

The following analyses will be performed; however, no formal inferential statistics will be done on safety assessments.

#### **6.8.1** Extent of Exposure

The extent of exposure to study drug in each treatment group will be summarized by total number of applications and total amount of study drug applied. Total amount of study drug will be calculated as the difference between tube weights at dispensation and return. The number and percentage of subjects who are compliant in each treatment group will be summarized. Subjects may not miss more than three consecutive days of dosing and must take at least 80% of expected doses to be considered compliant.

Subjects who were lost to follow up will be included in the total number of applications and total amount of study drug applied summaries, using their last known dose date.

#### **6.8.2** Adverse Events

All TEAEs that occur during the study will be recorded and coded based on the MedDRA dictionary, version 21.1. TEAEs are defined as AEs with an onset on or after the date of the first study drug application in this study.

TEAEs will be summarized by treatment group, the number of subjects reporting a TEAE, system organ class (SOC), preferred name, severity, relationship to study drug (causality), and

TOOL.ST.101-01.02 Statistical Analysis Plan Template



Arcutis Biotherapeutics, Inc. ARQ-151-202


seriousness. When summarizing AEs by severity and relationship, each subject will be counted once within an SOC or a preferred term by using the event with the highest severity and strongest relationship within each classification. Summaries of post active treatment emergent AEs (PATEAE) will also be presented. PATEAEs are defined as any AE that occurs after the first dose of ARQ-151 cream in either study.

Serious AEs (SAEs) will be summarized by treatment group, severity and relationship to study drug, and individual SAEs will be listed by subject. In addition, a list of subjects who prematurely discontinue from the study due to an AE, or experience an AE leading to death will be provided.

Listings will be presented for all AEs as well as for SAEs, and AEs leading to discontinuation from the study or death.

All information pertaining to AEs noted during the study will be listed by subject, detailing the verbatim description given by the Investigator, preferred term, system organ class, start date, stop date, severity, action taken regarding study drug, corrective treatment, outcome, and drug relatedness. The event onset will also be shown relative (in number of days) to date of first application. In addition, listings of SAEs and subjects who prematurely discontinue from the study due to adverse events will also be provided.

#### 6.8.3 Clinical Laboratory Evaluation

Routine blood chemistries and urinalysis will be obtained throughout the study and the results summarized by parameter at baseline and scheduled ARQ-151-202 study visits.

All clinical laboratory test results and their change from baseline will be summarized along with time point of collection.

Additionally, shifts tables will be provided describing out-of-normal range shifts for clinical laboratory results.

#### **6.8.4** Other Observations Related to Safety

## 6.8.4.1 12-Lead Electrocardiogram Measurements

Electrocardiograms (ECGs) will be tabulated at baseline and scheduled ARQ-151-202 study visits.



Arcutis Biotherapeutics, Inc. ARQ-151-202


#### 6.8.4.2 Vital Signs

Vital signs will be tabulated at baseline and scheduled ARQ-151-202 study visits. Additionally, a shift table will be used to summarize incidence of subjects who gain or lose >5% and >10% body weight over the course of the study. Any subject who gained or lost >5% body weight will be summarized in a listing with subject reported reason for weight loss (intentional, unintentional).

The incidence of shifts from baseline to last, highest, and lowest BMI category (underweight (BMI < 18.5), normal weight (18.5  $\leq$  BMI < 25), overweight (25  $\leq$  BMI < 30), obese (30  $\leq$  BMI) will be presented in shift tables.

#### 6.8.4.3 Physical Examination

Physical examination data will be presented in a by-subject listing.

#### **6.8.4.4** Local Tolerance Assessments

For the Investigator's assessment the numeric application site reaction scores will be summarized individually by using the number and percentage of subjects by visit.

#### 6.8.4.5 Patient Health Questionnaire Depression Scale

PHQ-8 data will be analyzed by a shift in state of severity using the following scoring system:

| Score | Result |
|----------|------------------------------|
| 0 to 4 | None – Minimal Depression |
| 5 to 9 | Mild Depression |
| 10 to 14 | Moderate Depression |
| 15 to 19 | Moderately Severe Depression |
| 20 to 24 | Severe Depression |

#### 6.8.4.6 Columbia-Suicide Severity Rating Scale

The C-SSRS will be analyzed per the C-SSRS Scoring and Data Analysis Guide.



Arcutis Biotherapeutics, Inc. ARQ-151-202


#### 6.8.4.7 Prior and Concomitant Medication

Prior and concomitant medication information for all subjects will be presented in a by-subject listing. Summary tables will be presented by World Health Organization-Anatomical Therapeutic Chemical Classification System (WHO-ATC) therapeutic category and product.

#### 7. DETERMINATION OF SAMPLE SIZE

A sample size of approximately 300 subjects is planned for Cohort 1 and up to approximately 100 subjects in Cohort 2 is planned for the study. This sample size will provide a sufficient population size to evaluate the long-term safety of ARQ-151 cream 0.3%.

#### 8. CHANGES IN THE PLANNED ANALYSES

The definition of baseline for Cohort 1 was changed to: the baseline value for safety and efficacy parameters (excluding laboratory and vital signs values) will be defined as the last observation prior to the first dose of ARQ-151 cream in either the ARQ-151-201 study or this study. Sensitivity analyses of IGA and PASI efficacy will be performed where the baseline value for subjects in Cohort 1 is defined as the last observation prior to the first dose of ARQ-151 0.3% cream in this study. For the purpose of these latter analyses, study procedures will not be repeated; the information from the ARQ-151-201 study Week 12 visit will be carried over to the Day 1 visit for this study.

Week 4 was added to the following secondary endpoints.

- Proportion (%) of subjects achieving an IGA of clear or almost clear
- Proportion (%) of applicable subjects with intertriginous area involvement, 'I-IGA' score of 'Clear' or 'Almost Clear'
- Proportion (%) of subjects achieving a 75% reduction from Baseline of mPASI (mPASI-75)

The following secondary endpoints were added to the analyses.

- Incidence of shifts from baseline to last, highest and lowest BMI category.
- The incidence of subjects who stop therapy during the study due to disease clearance on study. Disease clearance is defined as 'Clear' scores for IGA, I-IGA (if applicable and mPASI).



Arcutis Biotherapeutics, Inc. ARQ-151-202

- Proportion (%) of subjects achieving a 75% reduction from Baseline of PASI (PASI-75) at Week 4, 12, 24, 36, and 52. PASI was not specifically collected but will be derived based on already reported information.
- Proportion (%) of subjects achieving a 75% reduction from Baseline of mPASI (mPASI-75) at Week 4, 12, 24, 36, and 52.
- Proportion of subjects (%) with a 2-grade improvement in IGA from Baseline as observed at Weeks 4, 12, 24, 36, 52.
- Proportion of subjects (%) with IGA Success, defined as achievement of an IGA of 'Clear' or 'Almost Clear' plus a 2-grade improvement in IGA from Baseline as observed at Weeks 4, 12, 24, 36, and 52.
- Duration of IGA Success, defined as the time from the first observation of IGA Success
  to the first subsequent time a subject's disease response does not meet the criteria for
  IGA Success. The duration of IGA Success for subjects who end treatment in IGA
  Success will be censored at the last disease assessment date.
- Duration of IGA Clear or Almost Clear, defined as the time from the first observation of IGA Clear or Almost Clear to the first subsequent time a subject's disease response is not Clear or Almost Clear. The duration of IGA Clear or Almost Clear for subjects who end treatment with IGA Clear or Almost Clear will be censored at the last disease assessment date.
- Duration of PASI-50, defined as the time from the first observation of a 50% reduction from Baseline in the PASI to the first subsequent time a subject's PASI score is greater than a 50% reduction from Baseline. The duration of PASI-50 for subjects who end treatment with PASI score at least 50% less than Baseline will be censored at the last disease assessment date.
- Duration of PASI-75, defined analogously to duration of PASI-50
- Percent change from baseline in PASI score at each disease assessment
- Shift from the baseline IGA score to the last reported IGA score on study
- Frequency of disease recurrence among subjects who stop therapy due to disease clearance. Disease recurrence is defined as any instance where IGA is ≥ 2 or mPASI is greater than 0.
- Time to disease recurrence among subjects who stop therapy due to disease clearance. Time to disease recurrence is defined as the time from the last dose of ARQ-151 to the



Arcutis Biotherapeutics, Inc. ARQ-151-202


first observation of an IGA score of 2 or greater. The time to disease recurrence among subjects with clearance at the end of the study observation period will be censored at the last observed disease assessment

- The incidence of disease control among subjects who restart therapy after having stopped therapy due to disease clearance. Disease control is defined as achieving an IGA score of 0 or 1 subsequent to restarting study therapy.
- Time to disease control among subjects who restart therapy after having stopped therapy due to disease clearance. Time to disease control is the time from the restart of therapy to the first reported IGA score of 0 or 1. The time to disease control among subjects who do not achieve an IGA score of 0 or 1 by the end of the study observation period will be censored at the last observed disease assessment.

#### 9. REFERENCES

Berger, RS, Bowman JP. A reappraisal of the 21-day Cumulative Irritation Test in man. J. Toxicol Ot & Ocular Toxicol 1982:1(2);109-115.

Brion DE, Raynaud F, Plet A, Laurent P, Leduc B, and Anderson W. Deficiency of cyclic AMP-dependent protein kinases in human psoriasis. Proc. Natl. Acad. Sci. 1986; 83:5272-5276.

Hatzelmann A, Morcillo EJ, Lungarella G, Adnot S, Sanjar S, Beume R, et al. The preclinical pharmacology of roflumilast – a selective, oral phosphodiesterase 4 inhibitor in development for chronic obstructive pulmonary disease. Pulm Pharmacol Ther. 2010; 23:235–256.

Arcutis Biotherapeutics, Inc. ARQ-151-202 Version: 1

Date: 22OCT2020

# 10. INDEX OF PLANNED TABLES

| Table 14.0.1.1: Summary of Subject Enrollment and Evaluability (Enrolled Subjects: Cohort 1) |
|---|
| Table 14.0.1.2: Summary of Subject Enrollment and Evaluability (Enrolled Subjects: Cohort 2) |
| Table 14.0.1.3: Summary of Subject Enrollment and Evaluability (Enrolled Subjects)32 |
| Table 14.0.2.1: Summary of Subject Completion/Discontinuation (Safety Subjects: Cohort 1).33 |
| Table 14.0.2.2: Summary of Subject Completion/Discontinuation (Safety Subjects: Cohort 2).34 |
| Table 14.0.2.3: Summary of Subject Completion/Discontinuation (Safety Population)35 |
| Table 14.1.1.1: Summary of Subject Demographics (Safety Population: Cohort 1)36 |
| Table 14.1.1.1.2: Summary of Subject Demographics (Safety Population: Cohort 2)37 |
| Table 14.1.1.1.3: Summary of Subject Demographics (Safety Population) |
| Table 14.1.2.1.1: Primary Summary of Subject Baseline Characteristics (Safety Population: Cohort 1) |
| Table 14.1.2.1.2: Sensitivity Summary of Subject Baseline Characteristics (Safety Population: Cohort 1) |
| Table 14.1.2.2: Summary of Subject Baseline Characteristics (Safety Population: Cohort 2)45 |
| Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population) |
| Table 14.1.3.1: Summary of Concomitant Medications by ATC Level 2 Term and Standard Medication Name (Safety Population: Cohort 1) |
| Table 14.1.3.2: Summary of Concomitant Medications by ATC Level 2 Term and Standard Medication Name (Safety Population: Cohort 2) |
| Table 14.1.3.3: Summary of Concomitant Medications by ATC Level 2 Term and Standard Medication Name (Safety Population) |
| Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) |
| Table 14.2.1.1.2: Sensitivity Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) |
| Table 14.2.1.1.3: Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 2) |
| Table 14.2.1.1.4: Summary of Investigator Global Assessment (IGA) (Safety Population)77 |
| Table 14.2.1.2.1: Shift Table of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) |

Arcutis Biotherapeutics, Inc. ARQ-151-202

| Γable 14.2.1.2.2: Sensitivity Shift Table of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) | 84 |
|---|---|
| Γable 14.2.1.2.3: Shift Table of Investigator Global Assessment (IGA) (Safety Population: Cohort 2) | 85 |
| Table 14.2.1.2.4: Shift Table of Investigator Global Assessment (IGA) (Safety Population) | 86 |
| Table 14.2.2.1: Primary Summary of Intrigenous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) | 87 |
| Table 14.2.2.2: Sensitivity Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) | |
| Table 14.2.2.3: Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 2) | 96 |
| Table 14.2.2.4: Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population) | 99 |
| Table 14.2.3.1: Primary Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) | 02 |
| Γable 14.2.3.2: Sensitivity Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 1 | 09 |
| Γable 14.2.3.3: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 2) | 15 |
| Table 14.2.3.4: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population)1 | 21 |
| Table 14.2.4.1: Primary Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) | 27 |
| Γable 14.2.4.2: Sensitivity Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 1 | 33 |
| Γable 14.2.4.3: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population Cohort 2) | |
| Table 14.2.4.4: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population) | 43 |
| Γable 14.2.5.1: Summary of Duration of Treatment Free Interval and Investigator Global Assessment (IGA) Success (Safety Population: Cohort 1) | 49 |
| Figure 14.2.5.1.1: Kaplan-Meier Plot of Treatment Free Interval (Weeks) (Safety Population: Cohort 1) | 50 |
| Figure 14.2.5.1.2: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) Success (Weeks) (Safety Population: Cohort 1) | 51 |
| Γable 14.2.5.2: Summary of Duration of Treatment Free Interval and Investigator Global Assessment (IGA) Success (Safety Population: Cohort 2) | 52 |

Arcutis Biotherapeutics, Inc. ARQ-151-202

| Figure 14.2.5.2.1: Kaplan-Meier Plot of Treatment Free Interval (Weeks) (Safety Population: Cohort 2) |
|---|
| Figure 14.2.5.2.2: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) Success (Weeks) (Safety Population: Cohort 2) |
| Table 14.2.5.3: Summary of Duration of Treatment Free Interval and Investigator Global Assessment (IGA) Success (Safety Population) |
| Figure 14.2.5.3.1: Kaplan-Meier Plot of Treatment Free Interval (Weeks) (Safety Population) |
| Figure 14.2.5.3.2: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) Success (Weeks) (Safety Population) |
| Table 14.2.6.1: Summary of Disease Recurrence (Safety Population: Cohort 1)158 |
| Table 14.2.6.2: Summary of Disease Recurrence (Safety Population: Cohort 2)159 |
| Table 14.2.6.3: Summary of Disease Recurrence (Safety Population)160 |
| Table 14.2.7.1: Summary of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Safety Population: Cohort 1) |
| Figure 14.2.7.1: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Weeks) (Safety Population: Cohort 1) |
| Table 14.2.7.2: Summary of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Safety Population: Cohort 2) |
| Figure 14.2.7.2: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Weeks) (Safety Population: Cohort 2) |
| Table 14.2.7.3: Summary of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Safety Population) |
| Figure 14.2.7.3: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Weeks) (Safety Population) |
| Table 14.2.8.1.1: Primary Summary of Duration of PASI-50 (Safety Population: Cohort 1)167 |
| Figure 14.2.8.1.1: Primary Kaplan-Meier Plot of Duration of PASI-50 (Safety Population: Cohort 1) |
| Table 14.2.8.1.2: Sensitivity Summary of Duration of PASI-50 (Safety Population: Cohort 1) 169 |
| Figure 14.2.8.1.2: Sensitivity Kaplan-Meier Plot of Duration of PASI-50 (Safety Population: Cohort 1) |
| Table 14.2.8.2: Summary of Duration of PASI-50 (Safety Population: Cohort 2)171 |
| Figure 14.2.8.2: Kaplan-Meier Plot of Duration of PASI-50 (Safety Population: Cohort 2)172 |
| Table 14.2.8.3: Summary of Duration of PASI-50 (Safety Population) |
| Figure 14.2.8.3: Kaplan-Meier Plot of Duration of PASI-50 (Safety Population)174 |
| TOOL ST 101-01 02 Statistical Analysis Plan Template |

Arcutis Biotherapeutics, Inc. ARQ-151-202 Version: 1

Date: 22OCT2020

| Table 14.2.9.1: Summary of Duration of PASI-75 (Safety Population: Cohort 1) | 175 |
|---|---|
| Figure 14.2.9.1: Kaplan-Meier Plot of Duration of PASI-75 (Safety Population: Cohort 1) | 176 |
| Table 14.2.9.2: Summary of Duration of PASI-75 (Safety Population: Cohort 2) | 177 |
| Figure 14.2.9.2: Kaplan-Meier Plot of Duration of PASI-75 (Safety Population: Cohort 2) | 178 |
| Table 14.2.9.3: Summary of Duration of PASI-75 (Safety Population) | 179 |
| Figure 14.2.9.3: Kaplan-Meier Plot of Duration of PASI-75 (Safety Population) | 180 |
| Table 14.2.10.1: Summary of Time to Disease Recurrence (Safety Population: Cohort 1) | 181 |
| Figure 14.2.10.1: Kaplan-Meier Plot of Time to Disease Recurrence (Safety Population: Co 1) | |
| Table 14.2.10.2: Summary of Time to Disease Recurrence (Safety Population: Cohort 2) | 183 |
| Figure 14.2.10.2: Kaplan-Meier Plot of Time to Disease Recurrence (Safety Population: Co 2) | |
| Table 14.2.10.3: Summary of Time to Disease Recurrence (Safety Population) | 185 |
| Figure 14.2.10.3: Kaplan-Meier Plot of Time to Disease Recurrence (Safety Population) | 186 |
| Table 14.2.11.1: Summary of Disease Control (Safety Population: Cohort 1) | 187 |
| Figure 14.2.11.1: Kaplan-Meier Plot of Time to Disease Control (Safety Population: Cohort 1) | |
| Table 14.2.11.2: Summary of Disease Control (Safety Population: Cohort 2) | 189 |
| Figure 14.2.11.2: Kaplan-Meier Plot of Time to Disease Control (Safety Population: Cohort 2) | |
| Table 14.2.11.3: Summary of Disease Control (Safety Population) | |
| Figure 14.2.11.3: Kaplan-Meier Plot of Time to Disease Control (Safety Population) | |
| Table 14.3.0.1.1: Summary of Extent of Exposure (Safety Population: Cohort 1) | 193 |
| Table 14.3.0.1.2: Summary of Extent of Exposure (Safety Population: Cohort 2) | 194 |
| Table 14.3.0.1.3: Summary of Extent of Exposure (Safety Population) | 195 |
| Table 14.3.1.1.1: Summary of Local Tolerability (Safety Population: Cohort 1) | 196 |
| Table 14.3.1.1.2: Summary of Local Tolerability (Safety Population: Cohort 2) | 199 |
| Table 14.3.1.1.3: Summary of Local Tolerability (Safety Population) | 202 |
| Table 14.3.1.2.1: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population: Cohort 1) | 205 |
| Table 14.3.1.2.2: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population: Cohort 2) | 207 |

Arcutis Biotherapeutics, Inc. ARQ-151-202

| Table 14.3.1.2.3: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population) |
|---|
| Table 14.3.1.3.1: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population: Cohort 1) |
| Table 14.3.1.3.2: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population: Cohort 2) |
| Table 14.3.1.3.3: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population) |
| Table 14.3.1.4.1.1: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Inurious Behavior without Suicidal Intent Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population: Cohort 1) |
| Table 14.3.1.4.1.2: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Inurious Behavior without Suicidal Intent Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population: Cohort 1) |
| Table 14.3.1.4.1.3: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Inurious Behavior without Suicidal Intent Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population) |
| Table 14.3.1.4.2.1: Number of Patients with Suicidal-Related Treatment-Emergent Events Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population: Cohort 1) |
| Table 14.3.1.4.2.2: Number of Patients with Suicidal-Related Treatment-Emergent Events Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population: Cohort 2) |
| Table 14.3.1.4.2.3: Number of Patients with Suicidal-Related Treatment-Emergent Events Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population) |
| Table 14.3.2.1.1.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population: Cohort 1) |
| Table 14.3.2.1.1.2: Summary of Post Active Treatment-Emergent Adverse Events Characteristics (Safety Population: Cohort 1) |
| Table 14.3.2.1.2: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population: Cohort 2) |
| Table 14.3.2.1.3.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) |
| Table 14.3.2.1.3.2: Summary of Post Active Treatment-Emergent Adverse Events Characteristics (Safety Population) |

Arcutis Biotherapeutics, Inc. ARQ-151-202

| Table 14.3.2.2.1.1: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 1) |
|---|
| Table 14.3.2.2.1.2: Summary of Post Active Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 1) |
| Table 14.3.2.2.2: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 2) |
| Table 14.3.2.2.3.1: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.2.3.2: Summary of Post Active Treatment-Emergent Adverse Events System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.3.1.1: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population: Cohort 1) |
| Table 14.3.2.3.1.2: Summary of Post Active Treatment-Emergent Adverse Events by Severity (Safety Population: Cohort 1) |
| Table 14.3.2.3.2: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population: Cohort 2) |
| Table 14.3.2.3.3.1: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population) |
| Table 14.3.2.3.3.2: Summary of Post Active Treatment-Emergent Adverse Events by Severity (Safety Population) |
| Table 14.3.2.4.1.1: Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population: Cohort 1) |
| Table 14.3.2.4.1.2: Summary of Post Active Treatment-Emergent Adverse Events by Relationship (Safety Population: Cohort 1) |
| Table 14.3.2.4.2: Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population: Cohort 2) |
| Table 14.3.2.4.3.1: Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population) |
| Table 14.3.2.4.3.2: Summary of Post Active Treatment-Emergent Adverse Events by Relationship (Safety Population) |
| Table 14.3.2.5.1.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population: Cohort 1) |
| Table 14.3.2.5.1.2: Summary of Post Active Treatment-Emergent Serious Adverse Events Characteristics (Safety Population: Cohort 1) |
| Table 14.3.2.5.2: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population: Cohort 2) |

Arcutis Biotherapeutics, Inc. ARQ-151-202

| Table 14.3.2.5.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population) |
|---|
| Table 14.3.2.5.3.2: Summary of Post Active Treatment-Emergent Serious Adverse Events Characteristics (Safety Population) |
| Table 14.3.2.6.1.1: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 1) |
| Table 14.3.2.6.1.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 1)249 |
| Table 14.3.2.6.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 2) |
| Table 14.3.2.6.3.1: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.6.3.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.2.7.1.1: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population: Cohort 1) |
| Table 14.3.2.7.1.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by Severity (Safety Population: Cohort 1) |
| Table 14.3.2.7.2: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population: Cohort 2) |
| Table 14.3.2.7.3.1: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population) |
| Table 14.3.2.7.3.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by Severity (Safety Population) |
| Table 14.3.2.8.1.1: Summary of Treatment-Emergent Serious Adverse Events by Relationship (Safety Population: Cohort 1) |
| Table 14.3.2.8.1.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by Relationship (Safety Population: Cohort 1) |
| Table 14.3.2.8.2: Summary of Treatment-Emergent Serious Adverse Events by Relationship (Safety Population: Cohort 2) |
| Table 14.3.2.8.3.1: Summary of Treatment-Emergent Serious Adverse Events by Relationship (Safety Population) |
| Table 14.3.2.8.3.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by Relationship (Safety Subjects) |
| Table 14.3.3.1.1.1: Summary of Chemistry Laboratory Results (Safety Population: Cohort 1) |

Arcutis Biotherapeutics, Inc. ARQ-151-202

| Table 14.3.3.1.2.1: Summary of Hematology Laboratory Results (Safety Population: Cohort 1) | .266 |
|---|---|
| Table 14.3.3.1.3.1: Summary of Urinalysis Laboratory Results (Safety Population: Cohort 1). | .266 |
| Table 14.3.3.1.1.2: Summary of Chemistry Laboratory Results (Safety Population: Cohort 2) | .267 |
| Table 14.3.3.1.2.2: Summary of Hematology Laboratory Results (Safety Population: Cohort 2) | .270 |
| Table 14.3.3.1.3.2: Summary of Urinalysis Laboratory Results (Safety Population: Cohort 2). | .270 |
| Table 14.3.3.1.1.3: Summary of Chemistry Laboratory Results (Safety Population) | .271 |
| Table 14.3.3.1.2.3: Summary of Hematology Laboratory Results (Safety Population) | .274 |
| Table 14.3.3.1.3.3: Summary of Urinalysis Laboratory Results (Safety Population) | .274 |
| Table 14.3.3.2.1.1: Shift Summary of Chemistry Lab Results (Safety Population: Cohort 1) | .275 |
| Table 14.3.3.2.2.1: Shift Summary of Hematology Laboratory Results (Safety Population: Cohort 1) | .275 |
| Table 14.3.3.2.3.1: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population: Cohort 1) | .275 |
| Table 14.3.3.2.1.2: Shift Summary of Chemistry Lab Results (Safety Population: Cohort 2) | .276 |
| Table 14.3.3.2.2.2: Shift Summary of Hematology Laboratory Results (Safety Population: Cohort 2) | .276 |
| Table 14.3.3.2.3.2: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population: Cohort 2) | .276 |
| Table 14.3.3.2.1.3: Shift Summary of Chemistry Lab Results (Safety Population) | .277 |
| Table 14.3.3.2.2.3: Shift Summary of Hematology Laboratory Results (Safety Population) | .277 |
| Table 14.3.3.2.3.3: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population) | .277 |
| Table 14.3.4.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population: Cohort 1) | |
| Table 14.3.4.2: Summary of Electrocardiogram (ECG) Parameters (Safety Population: Cohort 2) | |
| Table 14.3.4.3: Summary of Electrocardiogram (ECG) Parameters (Safety Population) | .282 |
| Table 14.3.5.1.1: Summary of Vital Signs (Safety Population: Cohort 1) | .284 |
| Table 14.3.5.1.2: Summary of Vital Signs (Safety Population: Cohort 2) | .287 |
| Table 14.3.5.1.3: Summary of Vital Signs (Safety Population) | .290 |

Arcutis Biotherapeutics, Inc. ARQ-151-202 Version: 1

Date: 22OCT2020

| Table 14.3.5.2.1: Summary of Change in Body Weight Compared to Baseline (Safety Population: Cohort 1) |
|---|
| Table 14.3.5.2.2: Summary of Change in Body Weight Compared to Baseline (Safety Population: Cohort 2) |
| Table 14.3.5.2.3: Summary of Change in Body Weight Compared to Baseline (Safety Population) |
| Table 14.3.5.3.1: Shift Summary of Body Mass Index (BMI) Results (Safety Population: Cohort 1) |
| Table 14.3.5.3.2: Shift Summary of Body Mass Index (BMI) Results (Safety Population: Cohort 2) |
| Table 14.3.5.3.3: Shift Summary of Body Mass Index (BMI) Results (Safety Population)301 |

Table 14.0.1.1: Summary of Subject Enrollment and Evaluability (Enrolled Subjects: Cohort 1)

| | | ARQ-151-202: Roflumilast Cream 0.3% | ilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201: | A | ARQ-151-201: | |
| | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total |
| Number of Subjects Enrolled | × | ×× | × | XX |
| Number of Subjects Excluded from the | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Salety Fopulation Number of Subjects Included in the Safety Population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.0.1.2: Summary of Subject Enrollment and Evaluability (Enrolled Subjects: Cohort 2)

| Roflumilast Cream 0.3% | XX | xx ( xx.x%) | xx ( xx.x%) | |
|---|---|---|---|---|
| | Number of Subjects Enrolled | Number of Subjects Excluded from the Safety Population | Number of Subjects Included in the Safety | Population |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)


Table 14.0.1.3: Summary of Subject Enrollment and Evaluability (Enrolled Subjects)

| \(\sigma\) | Number of Subjects Enrolled Number of Subjects Excluded from the Safety Population Number of Subjects Included in the Safety | ARQ-151-201: Roflumilast Cream (N=xx) xx xx ( xx.x%) xx ( xx.x%) | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: Vehicle Cream and Cohort 2 (N=xx) xx xx xx (xx.x%) | 0.3% Total xx xx ( xx.x%) xx ( xx.x%) |
|---|---|---|---|---|
|---|---|---|---|---|

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)


Table 14.0.2.1: Summary of Subject Completion/Discontinuation (Safety Subjects: Cohort 1 )

| | ARQ-151-201: Roflumilast Cream 0.3% (N=xx) | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-201 Roflumilast Cream 0.15% Vehicle Crean (N=xx) | milast Cream 0.3% ARQ-151-201: Vehicle Cream (N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Completed Study<br>Yes<br>No | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%) xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| Reason for Discontinuation Adverse Event Lost to Follow-Up Pregnancy Protocol Deviation Withdrawal by Subject Study Terminated by Sponsor Physician Decision Lack of Efficacy Other <sup>a</sup> | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) | xx ( xx.x%) |
| Duration of Participation (Weeks) <sup>b</sup> n Mean SD Median Min. to Max. | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.X |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.1.2 for other discontinuation reasons.

<sup>b</sup> Duration of participation (weeks) is defined as (last contact date – date of first dose in ARQ-151-202 + 1) / 7 SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.0.2.2: Summary of Subject Completion/Discontinuation (Safety Subjects: Cohort 2)

| | Roflumilast Cream 0.3% $(N=xx)$ |
|---|---|
| Completed Study<br>Yes<br>No | xx ( xx.x%)<br>xx ( xx.x%) |
| Reason for Discontinuation<br>Adverse Event | xx ( xx.x%) |
| Lost to Follow-Up | |
| Pregnancy | XX ( XX.X <sup>0</sup> / <sub>0</sub> ) |
| Protocol Deviation | XX ( XX.X <sup>9</sup> / <sub>0</sub> ) |
| Withdrawal by Subject | XX ( XX.X <sup>0</sup> / <sub>0</sub> ) |
| Study Terminated by Sponsor | XX ( XX.X <sup>9</sup> / <sub>0</sub> ) |
| Physician Decision | XX ( XX.X <sup>9</sup> %) |
| Lack of Efficacy | XX ( XX.X%) |
| Other <sup>a</sup> | xx ( xx.x%) |
| Duration of Participation (Weeks) <sup>b</sup> | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | XX to XX |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.1.2 for other discontinuation reasons.

<sup>b</sup> Duration of participation (weeks) is defined as (last contact date – date of first dose + 1) / 7 SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.0.2.3: Summary of Subject Completion/Discontinuation (Safety Population)

| | ARO | ARQ-151-202: Roflumilast Cream 0.3% | 10.3% |
|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2<br>(N=xx) | Total<br>(N=xx) |
| Completed Study<br>Yes<br>No | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| Reason for Discontinuation | (%) ** ) ** | (%0 ^ ^ ) ^^ | (%^ ^^ ) ^^ |
| Lost to Follow-Up | ر<br>ر | _ ر | |
| Pregnancy | xx ( xx.x%) | <i>_</i> | xx ( xx.x%) |
| Protocol Deviation | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Withdrawal by Subject | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Study Terminated by Sponsor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Physician Decision | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lack of Efficacy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other <sup>a</sup> | XX ( XX.X%) | xx ( xx.x <sup>0</sup> %) | XX (XX.X%) |
| Duration of Participation (Weeks) <sup>b</sup> | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XXXX | XXX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.1.2 for other discontinuation reasons.
<sup>b</sup> Duration of participation (weeks) is defined as (last contact date – date of first dose in ARQ-151-202 + 1) / 7 SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.1.1.1.1: Summary of Subject Demographics (Safety Population: Cohort 1)

| | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Cream (N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Age (years) | <b>*</b> | <b>*</b> | ** | * |
| Mean | XX.XX | X.XX | XX.XX | XXX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Sex | <b>&gt;</b> | <b>&gt;</b> | <b>&gt;</b> | <b>&gt;</b> |
| 11 | ` | ` | ` | |
| Male | XX ( XX.X%) | XX ( XX.X%) | XX ( XX.X%) | XX ( XX.X%) |
| Female | xx ( xx.x%) | $XX (XX.X^{0})$ | xx ( xx.x%) | xx ( xx.x%) |
| Ethnicity | | | | |
| n | XX | XX | XX | XX |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ( xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Race | | | | |
| n | XX | XX | XX | XX |
| American Indian or Alaska Native | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ( xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ( XX.X%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ( xx.x%) |
| White | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ( xx.x%) |
| Multiple/Othera | $(\%^{\times} \times \times) \times \times$ | $(\% \times \times$ | (%x xx ) xx | (%x xx ) xx |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.4.1 for a complete list of all other races. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

# CONFIDENTIAL
Table 14.1.1.1.2: Summary of Subject Demographics (Safety Population: Cohort 2)

| Roflumilast Cream 0.3% $(N=xx)$ | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX to XX | xx.x%)<br>xx.x%) | xx.x%)<br>xx.x%) | XX.X%) XX.X%) XX.X%) XX.X%) XX.X%) XX.X%) XX.X%) |
|---|---|---|---|---|
| Roflumilast<br>(N= | × | XX () XX (X X X X X X X X X X X X X X X | x ) xx<br>x () xx | X X X X X X X X X X X X X X X X X X X |
| | Age (years) n Mean SD Median Min. to Max. | Sex<br>n<br>Male<br>Female | Ethnicity<br>n<br>Hispanic or Latino<br>Not Hispanic or Latino | Race<br>n<br>American Indian or Alaska Native<br>Asian<br>Black or African American<br>Native Hawaiian or Other Pacific Islander<br>White<br>Multiple/Other <sup>a</sup> |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.4.1 for a complete list of all other races. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.1.1.1.3: Summary of Subject Demographics (Safety Population)

| | XIII 7 | THE TOT FOR INCIDENTIAL STREET | |
|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201:<br>Vehicle Cream | |
| | Roflumilast Cream (N=xx) | and Cohort 2 $(N=xx)$ | $\begin{array}{c} \text{Total} \\ (\text{N} = xx) \end{array}$ |
| Age (years) | (333, 57) | (333, 1, 1) | (XXX XX) |
| | XX | XX | XX |
| san | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Sex | | | |
| | XX | XX | XX |
| le | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Ethnicity | | | |
| | XX | XX | xx |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | XX (XX.X%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Race | | | |
| | XX | XX | XX |
| American Indian or Alaska Native | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| White | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Multiple/Othera | (%a aa ) aa | (%0 AA ) AA | (%o^ o^ ) oo |

<sup>&</sup>lt;sup>a</sup> See Listing 16.2.4.1 for a complete list of all other races. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.1.2.1.1: Primary Summary of Subject Baseline Characteristics (Safety Population: Cohort 1)


| | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Cream (N=xx) | ARQ-151-201:<br>Vehicle Cream (N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Investigator Global Assessment n 0 - Clear 1 - Almost Clear 2 - Mild 3 - Moderate 4 - Severe | xx ( xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Intertriginous Investigator Global Assessment a n 1 - Almost Clear 2 - Mild 3 - Moderate 4 - Severe | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Body Surface Area (%) Affected n<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.X |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.1.2.1.1: Primary Summary of Subject Baseline Characteristics (Safety Population: Cohort 1)


<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

Table 14.1.2.1.1: Primary Summary of Subject Baseline Characteristics (Safety Population: Cohort 1) 

| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201: ARQ-151-201<br>Roflumilast Cream 0.15% Vehicle Crear | ARQ-151-201:<br>Vehicle Cream | Total |
|---|---|---|---|---|
| | (N=XX) | (N=xx) | (N=XX) | (x=N) |
| Height (cm) | | | | |
| | XX | XX | XX | XX |
| | X.XX | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX | XX.XX |
| | X.XX | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Weight (kg) | | | | |
| | XX | XX | XX | XX |
| | XX.X | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX | XX.XX |
| | X.XX | XX.X | XX.X | XX.X |
| lax. | xx to xx | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.1.2.1.2: Sensitivity Summary of Subject Baseline Characteristics (Safety Population: Cohort 1) 

| | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Cream (N=xx) | milast Cream 0.3% ARQ-151-201: Vehicle Cream (N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Investigator Global Assessment n 0 - Clear 1 - Almost Clear 2 - Mild 3 - Moderate 4 - Severe | XX<br>XX ( XX.X%)<br>XX ( XX.X%)<br>XX ( XX.X%)<br>XX ( XX.X%)<br>XX ( XX.X%) | xx<br>xx ( xx.x%) | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx<br>xx ( xx.x%) |
| Intertriginous Investigator Global Assessment a n 1 - Almost Clear 2 - Mild 3 - Moderate 4 - Severe | xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| Body Surface Area (%) Affected n Mean SD Median Min. to Max. | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX to XX |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

percentages. Note: Baseline is defined as the last observation prior to entry in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.1.2.1: Summary of Subject Baseline Characteristics (Safety Population: Cohort 1) 

| | ARQ-151-201: Roflumilast Cream 0.3% (N=xx) | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Crean (N=xx) | nilast Cream 0.3% ARQ-151-201: Vehicle Cream (N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Psoriasis Area Severity Index n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Modified Psoriasis Area Severity Index | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Duration of Psoriasis (Years) | | | | |
| u | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | X.XX | XX.X | XX.X | XX.X |
| Min. to Max. | XX to XX | XX to XX | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

percentages. Note: Baseline is defined as the last observation prior to entry in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.1.2.1.2: Sensitivity Summary of Subject Baseline Characteristics (Safety Population: Cohort 1)


| | ARO-151-201: | ARO-151-202: Roflumilast Cream 0.3%<br>ARO-151-201: ARO-151-201 | ilast Cream 0.3%<br>ARO-151-201: | |
|---|---|---|---|---|
| | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total |
| | (N=xx) | (N=XX) | (N=xx) | (N=xx) |
| ight (cm) | | | | |
| | XX | XX | XX | XX |
| <i>Aean</i> | XX.X | XX.X | XX.X | XX.X |
| D | XX.XX | XX.XX | XX.XX | XX.XX |
| <b>1</b> edian | XX.X | XX.X | XX.X | XX.X |
| fin. to Max. | XX to XX | xx to xx | xx to xx | xx to xx |
| Weight (kg) | | | | |
| | XX | XX | XX | XX |
| Iean | XX.X | XX.X | XX.X | XX.X |
| Ω | XX.XX | XX.XX | XX.XX | XX.XX |
| ledian | XX.X | XX.X | XX.X | XX.X |
| lin. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

percentages. Note: Baseline is defined as the last observation prior to entry in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.1.2.2: Summary of Subject Baseline Characteristics (Safety Population: Cohort 2) 

| m 0.3% | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Roflumilast Cream $0.3\%$ | | XX | $\overline{}$ | (xx.x%) | $\overline{}$ | $\overline{}$ | $\overline{}$ | | | XX | · / | $\overline{}$ | · / | xx ( xx.x%) | | XX | XX.X | XX.XX | XX.X | xx to xx |
| | Investigator Global Assessment | n | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe | Intertriginous Investigator Global | Assessment a | n | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe | Body Surface Area (%) Affected | n | Mean | SD | Median | Min. to Max. |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for percentages. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.1.2.2: Summary of Subject Baseline Characteristics (Safety Population: Cohort 2) 

| % | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | | XX | XX.X | XX.XX | XX.X | xx to xx | | XX | XX.X | XX.XX | XX.X | xx to xx | | XX | XX.X | XX.XX | XX.X | xx to xx |
| | Psoriasis Area Severity Index | n | Mean | SD | Median | Min. to Max. | Modified Psoriasis Area Sevierty Index | n | Mean | SD | Median | Min. to Max. | Duration of Psoriasis (Years) | u | Mean | SD | Median | Min. to Max. |

percentages. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

Table 14.1.2.2: Summary of Subject Baseline Characteristics (Safety Population: Cohort 2) 

| ım 0.3% | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | | XX | XX.X | XX.XX | XXX.X | xx to xx | | XX | XX.X | XX.XX | XX.X | xx to xx |
| | Height (cm) | u | Mean | SD | Median | Min. to Max. | Weight (kg) | u | Mean | SD | Median | Min. to Max. |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for percentages. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population)


| | 7 | ARO-151-202: Roflumilast Cream 0.3% | Feam 0.3% |
|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201:<br>Vehicle Cream | |
| | Roflumilast Cream $(N=xx)$ | and Cohort 2<br>(N=xx) | Total (N=xx) |
| Investigator Global Assessment | | | |
| n | XX | XX | XX |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | $xx (xx.x^{0})$ | xx ( xx.x%) | $XX (XX.X^{0})$ |
| Intertriginous Investigator Global Assessment <sup>a</sup> | | | |
| n | XX | XX | XX |
| 1 - Almost Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | XX ( XX.X%) | xx ( xx.x%) |
| Body Surface Area (%) Affected | | | |
| n | XX | XX | XX |
| Mean | XX.X | XXX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XXX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population)


| Psoriasis Area Severity Index n Mean SD Median Modified Psoriasis Area Severity Index n Median SD Median Min. to Max. | ARQ-151-201: Roflumilast Cream (N=xx) xx xx.x xx.x xx.x xx.x xx xx xx xx xx to xx xx.x xx xx | ARQ-151-201: Vehicle Cream and Cohort 2 (N=xx) xx xx.x xx to xx xx.x | Total (N=xx) xx xx.x xx.xx xx.xx xx to xx xx.xx |
|---|---|---|---|
| Psotiasis (Tears) | XX | XX | XX |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| | XXX | XXX | X.X.X |
| | V.V.V | V.VV | V.VV |
| ax. | vv to vv | vv +0 vv | VV TO VV |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population)


| Total<br>N=xx) | XX | XX.X | XX.XX | XX.X | xx to xx | | XX | XX.X | XX.XX | XX.X | xx to xx |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | XX | | | | • | | XX |
| ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: Vehicle Cream and Cohort 2 (N=xx) | XX | XX.X | XX.XX | XX.X | xx to xx | | XX | XX.X | XX.XX | XX.X | xx to xx |
| ARQ-151-201: Roflumilast Cream (N=xx) | XX | XX.X | XX.XX | XX.X | xx to xx | | XX | XX.X | XX.XX | XX.X | xx to xx |
| | (1 | | | | Лах. | ž | | | | | Лах. |
| | Height (cm)<br>n | Mean | SD | Median | Min. to N | Weight (kg) | п | Mean | $^{\mathrm{SD}}$ | Median | Min. to N |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting Clear or no intertriginous area involvement are included in denominator for

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.1.3.1: Summary of Concomitant Medications by ATC Level 2 Term and Standard Medication Name (Safety Population: Cohort 1)


| ATC Level 2 Term <sup>a</sup><br>Standard Medication Name | ARQ-151-201:<br>Roflumilast Cream $0.3\%$<br>(N=xx) | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-201 Roflumilast Cream 0.15% Vehicle Crear (N=xx) | nilast Cream 0.3% ARQ-151-201: Vehicle Cream (N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Standard Medication Name | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more concomitant medications that map to the WHO Drug Dictionary. At each level of summarization (ATC Level 2 Term or Standard Medication Name) subjects are counted once.

Note: WHO Drug Dictionary (Version xx).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.1.3.2: Summary of Concomitant Medications by ATC Level 2 Term and Standard Medication Name (Safety Population: Cohort 2)

| (Page 1 of xx) | Roflumilast Cream 0.3%<br>(N=xx) | xx ( xx.x%)<br>xx ( xx.x%) |
|---|---|---|
| | ATC Level 2 Term <sup>a</sup><br>Standard Medication Name | ATC Level 2 Term<br>Standard Medication Name |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more concomitant medications that map to the WHO Drug Dictionary. At each level of summarization (ATC Level 2 Term or Standard Medication Name) subjects are counted once.

Note: WHO Drug Dictionary (Version xx).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.1.3.3: Summary of Concomitant Medications by ATC Level 2 Term and Standard Medication Name (Safety Population)

| ATC Level 2 Term <sup>a</sup> | ARO | | |
|---|---|---|---|
| $\Delta$ TC Level 2 Term $^a$ | | ARQ-151-202: Kollumilast Cream 0.3% | 10.3% |
| A TC Leviel 2 Term $^a$ | | ARQ-151-201: | |
| ATC Level 2 Term <sup>a</sup> | ARQ-151-201: | Vehicle Cream | |
| | Roflumilast Cream | and Cohort 2 | Total |
| Standard Medication Name | (N=xx) | (N=xx) | (N=XX) |
| ATC Level 2 Term | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Standard Medication Name | xx ( xx.x%) | xx ( xx.x%) | (xx.x) xx.x% |

Note: WHO Drug Dictionary (Version xx).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more concomitant medications that map to the WHO Drug Dictionary. At each level of summarization (ATC Level 2 Term or Standard Medication Name) subjects are counted once.

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA)
(Safety Population: Cohort 1)


| Investigator Global Assessment Baseline <sup>a</sup> n 0 - Clear 1 - Almost Clear 2 - Mild | ARQ-151-201: Roflumilast Cream 0.3% (N=xx) xx xx xx (xx%) xx (xx%) xx (xx%) xx (xx%) | ARQ-151-201: | ARQ-151-201: Vehicle Cream (N=xx) xx xx xx (xx%) xx (xx%) xx (xx%) xx (xx%) | Total (N=xx) xx xx xx (xx%) xx (xx%) xx (xx%) xx (xx%) |
|---|---|---|---|---|
| 3 - Moderate<br>4 - Severe | | | | |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA)
(Safety Population: Cohort 1)


| | | | A | RQ-151-202: Roflu | ARQ-151-202: Roflumilast Cream 0.3% | | |
|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | AR<br>Roflum | ARQ-151-201: Roflumilast Cream 0.3% (N=xx) | ARG<br>Roflumila | ARQ-151-201:<br>Roflumilast Cream 0.15%<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total<br>(N=xx) |
| ARQ-151-201 Week 2<br>n | X | | XX | | NA | XX | |
| 0 - Clear | ) XX | (%XX | ) XX | (%XX | | ) xx | (%xx |
| - Almost Clear | XX ( | (%xx | ) xx | (%XX | | ) xx | (%xx |
| - Mild | XX ( | (%xx | ) xx | (%XX | | ) xx | (%xx |
| - Moderate | XX ( | (%xx | ) xx | (%XX | | ) xx | (%xx |
| 4 - Severe | xx ( | (%xx | ) xx | (%XX | | ) xx | (%XX |
| Score of Clear or Almost Clear | | | | | | | |
| Success | ) xx | (%XX | ) xx | (%XX | | ) xx | (%XX |
| Failure | xx ( | (%xx | ) xx | (%XX | | ) xx | (%XX |
| 2-Grade Improvement from Baseline<br>Success | ) XX | (%xx | ) XX | (%xx | | ) xx | (%XX |
| Failure | , xx | (%xx | xx ( | (%XX | | ) xx | (%XX |
| Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success | XX | (%xx | ×× | (%xx | | ) xx | (%xx |
| Failure | × | (%xx | ) XX | (%XX<br>(%XX) | | ) XX | (%XX) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA)
(Safety Population: Cohort 1)


| | | | ARO | -151-202: Roflu | ARO-151-202: Roflumilast Cream 0.3% | | |
|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | AlRoflum | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-1<br>Roflumilast (N= | ARQ-151-201:<br>Roflumilast Cream 0.15%<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total<br>N=xx) |
| ARQ-151-201 Week 4 | | | | | | | |
| n | XX | | XX | | NA | XX | |
| 0 - Clear | ) xx | (%xx | xx ) xx | (%xx | | ) xx | (%XX |
| 1 - Almost Clear | XX | (%xx | | (% | | ( ) xx | (%XX |
| 2 - Mild | XX | (%xx | · _ | (%xx | | ) xx | (%xx |
| 3 - Moderate | XX | (%xx | xx ) xx | (% | | ( ) xx | (%XX |
| 4 - Severe | xx ( | (%xx | , _ | (%XX | | , _ | (%xx |
| Score of Clear or Almost Clear | | | | | | | |
| Success | ) xx | (%xx | $\overline{}$ | (%) | | ) xx | (%xx |
| Failure | ) xx | (%xx | xx ) xx | (%XX | | xx ( | (%XX |
| 2-Grade Improvement from Baseline | , | ; | | : | | , | |
| Success | ) xx | (%XX | _ | (%xx | | ) xx | (%xx |
| Failure | ) xx | (%XX | xx ) xx | (%xx | | xx ( | (%XX |
| Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success Failure | ×× | xx%)<br>xx%) | xx ) xx | xx%)<br>xx%) | | ×× | xx%)<br>xx%) |
| | , | ` | , | | | , | ` |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| | | | A | RQ-151-202: Roflu | ARQ-151-202: Roflumilast Cream 0.3% | | | 1 |
|---|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | AF<br>Roflum | ARQ-151-201:<br>Roflumilast Cream $0.3\%$ | AR<br>Roflumil | ARQ-151-201:<br>Roflumilast Cream 0.15% $(N=xx)$ | ARQ-151-201:<br>Vehicle Cream $(N=xx)$ | | Total $(N=xx)$ | |
| | | (www.ti) | | (333) | (333, 71) | | (XXX LT) | 1 |
| ARQ-151-201 Week 6 | | | | | | | | |
| n | XX | | XX | | NA | XX | | |
| 0 - Clear | ) xx | (%XX | ) xx | (%XX | | ) xx | (%XX | |
| 1 - Almost Clear | ) XX | (%XX | ) xx | (%XX | | ) xx | (%XX | |
| 2 - Mild | ) XX | (%XX | ) xx | (%xx | | ) xx | (%XX | |
| 3 - Moderate | XX | (%xx | ) xx | (%xx | | XX ( | (%XX | |
| 4 - Severe | ) xx | (%xx | ) xx | (%xx | | ) xx | (%XX | |
| Score of Clear or Almost Clear | | | | | | | | |
| Success | ) xx | (%xx | ) xx | (%xx | | ) xx | (%XX | |
| Failure | ) xx | (%xx | ) xx | (%xx | | ) xx | (%xx | |
| 2-Grade Improvement from Baseline | , | ; | , | | | , | : | |
| Success | ) xx | (%xx | ) xx | (%XX | | ) xx | (%XX | |
| Failure | ) XX | (%XX | ) xx | (%xx | | ) xx | (%xx | |
| Score of Clear or Almost Clear Plus<br>2-Grade Improvement from Baseline | | | | | | | | |
| Success | ) XX | (%xx | ) xx | (%XX | | ) xx | (%xx | |
| Failure | ) XX | (%XX | ) xx | (%XX | | ) XX | (%XX | |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA)
(Safety Population: Cohort 1)


<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| ARQ | ARQ-151-201: | | | | | | |
|---|---|---|---|---|---|---|---|
| otlumila | Roflumilast Cream 0.3% (N=xx) | ARÇ<br>Roflumila<br>( | ARQ-151-201:<br>Roflumilast Cream 0.15%<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total<br>(N=xx) | |
| | | | | 41.6 | | | |
| XX | : | XX | : | NA | XX | : | |
| xx ( ) | (%xx | ) xx | (%xx | | ) xx | (%xx | |
| xx ( ) | (%xx | ) xx | (%XX | | ) xx | (%xx | |
| xx ( ) | (%XX | ) xx | (%XX | | ) xx | (%xx | |
| xx ( ) | (%XX) | ) xx | (%XX | | ) xx | (%xx | |
| xx () xx | (%XX | ) xx | (%XX | | ) xx | (%XX | |
| xx ( ) | (%XX | ) xx | (%xx | | ) xx | (%xx | |
| xx ( ) | (%X%) | ) xx | (%XX | | ) xx | (%XX | |
| xx ( | (%XX | _ | (0%XX | | ) xx | (%XX | |
| xx ( | (%xx) | ) xx | (%XX | | ) xx | (%XX | |
| | (x%) | <u> </u> | (%xx | | ) xx | (%xx | |
| _ | (%XX) | _ | XX%0) | | ) XX | (0%XX | |
| * | | (%xx | (%xx)<br>(xx) | (%xx | XX (%XX ) XX (%XX ) (XX (XX (%XX ) (XX | (%xx ) | ) xx (%x ) x |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| | | | 7 | ARQ-151-202: Roflumilast Cream 0.3% | milast Cro | eam 0.3% | | | |
|---|---|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | AR<br>Roflumi | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | Al<br>Roflum | ARQ-151-201:<br>Roflumilast Cream 0.15%<br>(N=xx) | AR | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total<br>(N=xx) | İ |
| Week 4 | | , | | , | | , | | | ı |
| n | XX | | XX | | XX | | XX | | |
| 0 - Clear | ) xx | (%XX | ) xx | (%xx | ) XX | (%XX | ) xx | (%XX | |
| 1 - Almost Clear | XX ( | (%xx | XX ( | (%xx | XX ( | (%XX | XX ( | (%xx | |
| 2 - Mild | xx ( | (%xx | ) XX | (0/XX | XX | (%xx | ) xx | (%xx | |
| 3 - Moderate | ) xx | (%xx | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | |
| 4 - Severe | ) xx | (%xx | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx | |
| Score of Clear or Almost Clear | | | | | | | | | |
| Success | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX | |
| Failure | ) xx | (%xx | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx | |
| 2-Grade Improvement from Baseline Success | XX | (%XX | ) XX | (%XX | ) XX | (%XX | ) XX | (%xx | |
| Failure | , ) XX | (%xx | ) xx | (%XX | ) XX | (0%xx | ) xx | (%xx | |
| Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success Failure | ) X X | xx%)<br>xx%) | ) xx ( | xx%6)<br>xx%0) | ) X X | xx%)<br>xx%) | ) xx | xx%)<br>xx%) | |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| Score of Clear or Almost Clear Success xx (xx%) Failure xx (xx%) | xx (%xx ) xx (%) xx (%) | xx ( xx%) xx ( xx%) xx ( xx%) | (%XX ) XX (XX ) XX (XX ) |
|---|---|---|---|

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| ARQ-151-201: Roflumilast Cream 0.3% Xx Xx Xx Xx Xx Xx Xx X | | , | ANY 151 202: INMIRITARY CLARIN 0:37/9 | 4 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
|---|---|---|---|---|---|
| XX | | 51-201:<br>Cream 0.3%<br>=xx) | ARQ-151-201: Roflumilast Cream 0.15% (N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | Total<br>(N=xx) |
| XX ( xx%) | | | | | |
| Xx ( xx%) Xx ( | | | XX | XX | XX |
| Xx ( xx%) Xx ( | ) xx | (%) | (%xx ) xx | xx ( xx%) | (%xx ) xx |
| Xx ( xx%) Xx ( | ) xx | (%) | (%xx ) xx | | |
| Xx ( xx%) Xx ( | ) xx | (%) | (%xx ) xx | | (%xx ) xx |
| Almost Clear xx (xx%) | ) xx | (%) | | (%xx ) xx | (%xx ) xx |
| xx ( xx%)<br>xx ( xx%)<br>seline<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) | ) xx | (%) | | (%XX ) XX | |
| xx ( xx%)<br>xx ( xx%)<br>seline<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) | Lear or Almost Clear | | | | |
| xx ( | ) xx | (%) | (0/XX) $(XX)$ | $\overline{}$ | (%XX ) XX |
| (%xx ) xx (%xx) xx (%xx) xx (%xx) xx | ) xx | (%) | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| xx ( | ` | | , | | |
| (%xx ) xx | ) XX | (%) | (0%XX ) XX | (0%xx ) xx | _ |
| (/0 | ) xx | (%) | (%xx () xx | (%XX ) XX | (%XX ) XX |
| /0.5.5 | | | | | |
| (%xx%)<br>(%xx ) | ) xx | (%)<br>(%) | xx ( xx%0)<br>xx ( xx%0) | xx ( xx%)<br>xx ( xx%) | (%xx ) xx<br>(0%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| Investigator Global Assessment | Roflum | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | AR<br>ARC<br>Roflumila | ARQ-151-202: Rofluminast Cream 0.5% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Cream (N=xx) | AR | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total<br>(N=xx) |
|---|---|---|---|---|---|---|---|---|
| Week 36 | × | | × | | × | | X | |
| 0 - Clear | ) XX | (%xx | ) XX | (%XX | ) xx | (%XX | ) XX | (%XX |
| 1 - Almost Clear | XX | (%XX | ) XX | (%XX | XX | (%xx | XX ( | (%xx |
| 2 - Mild | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx) |
| 3 - Moderate | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx |
| 4 - Severe | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx |
| Score of Clear or Almost Clear | | | | | | | | |
| Success | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx |
| Failure | ) XX | (%xx | ) xx | (%XX | ) XX | (%XX | ) xx | (%xx |
| 2-Grade Improvement from Baseline | , | (/0 | , | ()0 | | (/0 | , | () |
| Success<br>Failure | ×<br>X<br>X | xx /0)<br>xx %) | X<br>X<br>X | xx /0)<br>xx %) | X<br>X<br>X | xx /0)<br>xx /%) | X<br>X<br>X | (%xx<br>(%xx |
| Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success Failure | XX | xx%)<br>xx%) | ) xx | xx%)<br>xx%) | ) XX | (%xx<br>(%xx) | ) xx | xx%)<br>xx%() |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.1: Primary Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| | | | AF | ARQ-151-202: Roflumilast Cream 0.3% | milast Crea | ım 0.3% | | |
|---|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | AF<br>Roflum | ARQ-151-201: Roflumilast Cream 0.3% (N=xx) | AR(<br>Roflumila<br>( | ARQ-151-201:<br>Roflumilast Cream $0.15\%$<br>(N=xx) | ARÇ<br>Vehi<br>( | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total<br>(N=xx) |
| Week 52 | | | | | | | | |
| п | XX | | XX | | XX | | XX | |
| 0 - Clear | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX |
| 1 - Almost Clear | ) XX | (%xx | ) xx | (%xx | ) XX | (%xx | ) xx | (%XX |
| 2 - Mild | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx | ) xx | (%XX |
| 3 - Moderate | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX |
| 4 - Severe | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx |
| Score of Clear or Almost Clear | | | | | | | | |
| Success | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx |
| Failure | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx |
| 2-Grade Improvement from Baseline | ` | | ` | | , | | ` | |
| Success | ) XX | (%XX | ) xx | (%XX | )<br>X | (%XX | ) XX | (%XX |
| Failure | ) XX | (%XX | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX |
| Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline | | | | | | | | |
| Success | ) xx | (%XX | ) xx | (%XX | | (%xx | ) xx | (%XX |
| Failure | ) xx | (%XX | ) xx | (%XX | ) XX | (%xx | ) xx | (%xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.2: Sensitivity Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| | | ARQ-151-202: Roflu | milast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201: ARQ-151-201: | ARQ-151-201: | |
| | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total |
| Investigator Global Assessment | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| $Baseline^a$ | | | | |
| n | XX | XX | XX | XX |
| 0 - Clear | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| 1 - Almost Clear | (%xx ) xx | | (%xx ) xx | |
| 2 - Mild | (%xx ) xx | | | _ |
| 3 - Moderate | (%xx ) xx | (%xx () xx | (%xx ) xx | (%xx ) xx |
| 4 - Severe | (%xx ) xx | (%xx () xx | (%xx ) xx | (%xx () xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entry in ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.2: Sensitivity Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-201: ARQ-151-201: Roflumilast Cream 0.3% Roflumilast Cream 0.15% Vehicle Cream Total (N=xx) | xx | ) xx (%xx ) xx<br>) xx (%xx ) xx | xx (xx - xx%) $xx (xx - xx%)$ | xx ( xx %) | (9%xx ) xx $(9%$ xx ) xx $(9%$ xx ) xx $(9%$ xx ) xx |
|---|---|---|---|---|---|
| ARQ-151-201:<br>umilast Cream 0.3%<br>(N=xx) | $\sim$ | $\smile$ | $\smile$ | $\smile$ | |
| Investigator Global Assessment | Week 4 n 0 - Clear 1 - Almost Clear 2 - Mild | 3 - Moderate<br>4 - Severe | Score of Clear or Almost Clear<br>Success<br>Failure | 2-Grade Improvement from Baseline<br>Success<br>Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entry in ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.2: Sensitivity Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-201: Roflumilast Cream 0.15% Vehicle Cream (N=xx) (N=xx) (N=xx) | xx | xx%0) xx ( | (%xx) xx (%xx) xx (%xx) (%xx |
|---|---|---|---|
| ARQ<br>ARQ<br>Roflumilas | X X X X X X | X X X X X X X X X X X X X X X X X X X | XX ( ) XX |
| ARQ-151-201:<br>Roflumilast Cream $0.3\%$ $(N=xx)$ | xx ( xx%) | (%xx ) xx ( | (%xx ) xx |
| Investigator Global Assessment | Week 12 n 0 - Clear 1 - Almost Clear 2 - Mild 3 - Moderate 4 - Severe | Score of Clear or Almost Clear Success Failure 2-Grade Improvement from Baseline Success Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success Failure |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entry in ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)


Table 14.2.1.1.2: Sensitivity Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| | | | A ! | ARQ-151-202: Roflumilast Cream 0.3% | milast Cr | eam 0.3% | | |
|---|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | AF<br>Roflum | ARQ-151-201: Roflumilast Cream 0.3% (N=xx) | AR<br>Roflumil | ARQ-151-201:<br>Roflumilast Cream $0.15\%$ $(N=xx)$ | AR<br>Ve | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total<br>(N=xx) |
| Week 24 | | | | | | | | |
| n | XX | | XX | | XX | | XX | |
| 0 - Clear | ) XX | (%XX | ) xx | (%XX | ) xx | (%xx | ) XX | (%xx |
| 1 - Almost Clear | XX | (%xx | ) xx | (%XX | ) xx | (%xx | ) XX | (%xx |
| 2 - Mild | XX | (%XX | ) xx | (%XX | ) xx | (%xx | ) XX | (%xx |
| 3 - Moderate | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx |
| 4 - Severe | ) xx | (%xx | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx |
| Score of Clear or Almost Clear | | | | | | | | |
| Success | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx |
| Failure | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX |
| 2-Grade Improvement from Baseline | | | | | ` | | | ć |
| Success | )<br>XX | (%XX | ) xx | (0%XX | )<br>XX | (0%XX | )<br>XX | (0%XX |
| Failure | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx |
| Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline | | ć | ` | | | | ` | ć |
| Success<br>Failure | ) )<br>X X | xx%)<br>xx%) | ) )<br>X | xx%)<br>xx%) | × × | (%xx<br>(%xx | ) )<br>X X | xx%)<br>xx%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entry in ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.2: Sensitivity Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| ARQ-151-202: Roflumilast Cream 0.3% 2-151-201: ARQ-151-201: ARQ-151-201: ast Cream 0.3% Roflumilast Cream 0.15% Vehicle Cream (N=xx) N=xx) (N=xx) (N=xx) | $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) $xx$ | xx ( xx%) xx ( xx%) | ) xx (%xx ) xx ( xx ) xx ( | | ) xx (%xx ) xx | $(x^{0})$ | (%xx ) xx (%xx ) xx (%xx ) xx (%xx ) xx (%xx ) | ) xx (%xx ) xx (xx%) xx (xx%) | (%xx) xx $(%xx)$ xx $(%xx)$ xx $(%xx)$ xx $(%xx)$ |
|---|---|---|---|---|---|---|---|---|---|---|
| Jumilast | XX | X<br>X | ) XX | ××× | | ) xx | ) xx | ) XX | ) xx | ) xx |
| ARQ-151-202: Ro<br>ARQ-151-201:<br>Roflumilast Cream 0.15%<br>(N=xx) | | | | | | $\overline{}$ | _ | _ | | $\smile$ |
| ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | (%0xx ) xx<br>XX | | | (%xx ) xx (%) | | (%XX ) XX | (%XX ) XX | (%XX ) XX | (%xx ) xx | (%xx ) xx |
| F<br>Investigator Global Assessment | Week 36<br>n<br>0 - Clear | J - Almost Clear | 2 - Mild | 5 - Mouraic<br>4 - Severe | Score of Clear or Almost Clear | Success | Failure | 2-Grade Improvement from Baseline Success | Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entry in ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.2: Sensitivity Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 1) 

| Total (N=xx) | xx ( xx%) | (%xx ) xx<br>(%xx ) xx<br>(%xx ) xx<br>(%xx ) xx | (%xx ) xx (%xx ) xx |
|---|---|---|---|
| ARQ-151-201: Vehicle Cream (N=xx) | xx ( xx%) | xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) | xx ( xx%)<br>xx ( xx%) |
| ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Cream (N=xx) | xx (xx%)<br>xx (xx%)<br>xx (xx%)<br>xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (%xx ) xx<br>(%xx ) xx<br>(%xx ) xx<br>(%xx ) xx | xx (%xx ) xx<br>(%xx ) xx |
| ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | xx ( | xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) | xx ( |
| Investigator Global Assessment | Week 52 n 0 - Clear 1 - Almost Clear 2 - Mild 3 - Moderate 4 - Severe | Score of Clear or Almost Clear Success Failure 2-Grade Improvement from Baseline Success Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success Failure |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entry in ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.2.1.1.3: Summary of Investigator Global Assessment (IGA)
(Safety Population: Cohort 2)


| ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | | XX | | | | (%XX ) XX | |
|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | Baseline | n | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |

Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.3: Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 2) 

| ARQ-151-201: Roflumilast Cream 0.3% (N=xx) | | | xx ( xx/%)<br>xx ( xx/%) | _ 、 | _ | (%xx ) xx | $\overline{}$ | | (%xx ) xx | | (%XX ) XX | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | Week 4 | n<br>0 - Clear<br>1 - Alacet Clear | 1 - Annost Crear<br>2 - Mild | 3 - Moderate | 4 - Severe | Score of Clear or Almost Clear Success | Failure | 2-Grade Improvement from Baseline Success | Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline | Success | Failure |

Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)
Table 14.2.1.1.3: Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 2) 

| n 0.3% | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | | | _ 、 | (%xx<br>) | | (%xx ) | $\overline{}$ | | (%xx ) | | (%xx ) xx | |
| Ro | , | XX | × | XX<br>XX | × | XX | X | × | XX | | × | X |
| Investigator Global Assessment | Week 12 | n<br>0 - Clear | 1 - Almost Clear | z - Ivilid<br>3 - Moderate | 4 - Severe | Score of Clear or Almost Clear<br>Success | Failure | 2-Grade Improvement from Baseline Success | Failure | Score of Clear or Almost Clear Plus<br>2-Grade Improvement from Baseline | Success | Failure |

Note: No imputation of missing values.
SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.2.1.1.3: Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 2) 

| ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | xx (xx, 0, | | (%xx ) xx<br>(%xx ) xx |
|---|---|---|---|
| Investigator Global Assessment | Week 24 n 0 - Clear 1 - Almost Clear 2 - Mild 3 - Moderate 4 - Severe | Score of Clear or Almost Clear Success Failure 2-Grade Improvement from Baseline Success Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success Failure |

Note: No imputation of missing values.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.3: Summary of Investigator Global Assessment (IGA)
(Safety Population: Cohort 2)


| ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | xx%0)<br>xx%0)<br>xx%0)<br>xx%0)<br>xx%0) | xx%6) xx%6) xx%6) xx%90 | xx%)<br>xx%) |
|---|---|---|---|
| AR<br>Roflumi | ) X X X X X X X | ) | ) xx |
| Investigator Global Assessment | Week 36 n 0 - Clear 1 - Almost Clear 2 - Mild 3 - Moderate 4 - Severe | Score of Clear or Almost Clear Success Failure 2-Grade Improvement from Baseline Success Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success Failure |

Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.2.1.1.3: Summary of Investigator Global Assessment (IGA) (Safety Population: Cohort 2) 

| 3% | | | | | |
|---|---|---|---|---|---|
| ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | xx (%xx ) xx (%xx ) xx | | (%XX ) XX (%) | (%) xx ( xx%) xx ( xx%) | (%xx ) xx<br>(%xx ) xx |
| Investigator Global Assessment | Week 52 n 0 - Clear 1 - Almost Clear 2 - Mild | 3 - Moderate<br>4 - Severe | Score of Clear or Almost Clear<br>Success<br>Failure | 2-Grade Improvement from Baseline<br>Success<br>Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Success Failure |

Note: No imputation of missing values.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.4: Summary of Investigator Global Assessment (IGA) (Safety Population) 

| ARQ-151-202: Roflumilast Cream 0.3% | | | XX XX XX | ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) | ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) | (0,0) XX $(0,0)$ XX $(0,0)$ XX $(0,0)$ XX | ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) | ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) |
|---|---|---|---|---|---|---|---|---|
| | Investigator Global Assessment | Baseline <sup>a</sup> | n | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.4: Summary of Investigator Global Assessment (IGA) (Safety Population) 

| | | ARG | 2-151-202 | ARQ-151-202: Roflumilast Cream 0.3% | m 0.3% | | |
|---|---|---|---|---|---|---|---|
| Investigator Global Assessment | Al<br>Roff | ARQ-151-201:<br>Roflumilast Cream<br>(N=xx) | A V | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2<br>(N=xx) | | Total<br>(N=xx) | Ī |
| Week 4 | | | | | | | |
| n | xx | | XX | | XX | | |
| 0 - Clear | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx | |
| 1 - Almost Clear | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | |
| 2 - Mild | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | |
| 3 - Moderate | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | |
| 4 - Severe | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | |
| Score of Clear or Almost Clear | | | | | | | |
| Success | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| Failure | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx | |
| 2-Grade Improvement from Baseline | | | | | | | |
| Success | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | |
| Failure | ) xx | (%xx | ) xx | (%xx | ) xx | (%XX | |
| Score of Clear or Almost Clear Plus<br>2-Grade Improvement from Baseline | | | | | | | |
| Success | ) XX | (%XX | ) XX | (%XX | ) XX | (%XX | |
| Failure | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.4: Summary of Investigator Global Assessment (IGA) (Safety Population) 

| ARQ-151-202: Roflumilast Cream 0.3% | $ARQ-151-201: \\ ARQ-151-201: Vehicle Cream \\ Roflumilast Cream and Cohort 2 Total \\ \hline (N=xx) (N=xx) (N=xx)$ | XX XX | xx (xx%) xx (xx%) $xx (xx%) xx (xx%)$ ost Clear $xx (xx%) xx (xx%)$ $xx (xx%)$ | (xx) $(xx)$ $(xx)$ $(xx)$ $(xx)$ $(xx)$ | ) $XX$ (% $XX$ ) $XX$ (% $XX$ ) $XX$ | ) xx (%xx ) xx (%xx ) xx | Score of Clear or Almost Clear | (%XX) XX $(%XX)$ XX | ) xx (%xx ) xx (%xx ) xx ( | 2-Grade Improvement from Baseline | (% XX) XX (% XX) XX | ) xx (%xx ) xx (%xx ) xx | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline xx (xx%) xx (xx%) xx (xx%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Investigator Global Assessment | Week 12 | 0 - Clear<br>1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe | Score of Clear or Alm | Success | Failure | 2-Grade Improvement | Success | Failure | Score of Clear or Alm 2-Grade Improvement Success |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.4: Summary of Investigator Global Assessment (IGA) (Safety Population) 

| | | ARC | 2-151-202: R | ARQ-151-202: Roflumilast Cream 0.3% | n 0.3% | |
|---|---|---|---|---|---|---|
| | ARQ | ARQ-151-201: | ARQ<br>Vehi | ARQ-151-201:<br>Vehicle Cream | | |
| Investigator Global Assessment | Roflun (1 | Roflumilast Cream (N=xx) | and | and Cohort 2 (N=xx) | | Total<br>(N=xx) |
| Week 24 | | | | | | |
| n | XX | | XX | | XX | |
| 0 - Clear | $\overline{}$ | (%XX | $\overline{}$ | (%XX | ) xx | (%XX |
| 1 - Almost Clear | ( ) XX | (%XX | $\overline{}$ | (%xx | ) xx | (%xx |
| 2 - Mild | $\overline{}$ | (%xx | ) xx | (%xx | ) xx | (%XX |
| 3 - Moderate | ( ) XX | (%XX | $\overline{}$ | (%xx | ) xx | (%xx |
| 4 - Severe | xx ( | (%xx | $\overline{}$ | (%xx | ) xx | (%xx |
| Score of Clear or Almost Clear | | | | | | |
| Success | $\overline{}$ | (%xx | $\overline{}$ | (%xx | ) xx | (%XX |
| Failure | xx ( | (%XX | ) xx | (%xx | ) xx | (%XX |
| 2-Grade Improvement from Baseline | | | | | | |
| Success | $\overline{}$ | (%XX | | (%xx | ) xx | (%XX |
| Failure | xx ( | (%xx | ) xx | (%xx | ) xx | (%XX |
| Score of Clear or Almost Clear Plus<br>2-Grade Improvement from Baseline | | | | | | |
| Success | | (%xx | ) XX | (%XX | ) XX | (%XX |
| Failure | xx ( | (%xx | | (%xx | ) xx | (%xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.1.4: Summary of Investigator Global Assessment (IGA)
(Safety Population)


| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201: Vehicle Cream Roflumilast Cream and Cohort 2 Total (N=xx) (N=xx) | XX XX | xx (xx%) xx (xx%) xx (xx%) xx (xx%) ost Clear $xx (xx%) xx (xx%) xx (xx%)$ | (xx)(xx)(xx) $(xx)(xx)(xx)$ $(xx)(xx)(xx)$ | ) XX $(\%XX)$ XX $(\%XX)$ XX | ) xx (%xx ) xx (%xx ) xx | Score of Clear or Almost Clear | (%XX) XX $(%XX)$ XX | ) xx (%) xx ( xx%) xx ( (xx ) xx ( xx%) xx ( xx ) xx ( x | 2-Grade Improvement from Baseline | (% XX) XX (% XX) XX | ) xx (%xx ) xx (%xx ) xx (%xx ) xx | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline Xx (xx%) xx (xx%) xx (xx%) xx (xx%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Investigator Global Assessment | Week 36 | 0 - Clear<br>1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe | Score of Clear or Almo | Success | Failure | 2-Grade Improvement | Success | Failure | Score of Clear or Almostrate Improvement Success |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.1.4: Summary of Investigator Global Assessment (IGA) (Safety Population) 

| | 10ta1<br>(N=xx) | X | $\overline{}$ | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx | | (%xx ) xx | (%xx ) xx | | (%xx ) xx | (%XX ) XX | | (%XX) XX | ر |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: Vehicle Cream | and Conort 2<br>(N=xx) | XX | (%XX ) XX | (%XX ) XX | (%xx ) xx | (%xx ) xx | (%xx ) xx | | (%xx) xx | (%xx ) xx | | (%xx ) xx | (%xx ) xx | | (%xx ) xx | ر |
| | Nollumiasi Cream | × | $\overline{}$ | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx | | (%xx ) xx | (%xx ) xx | | (%xx ) xx | (%XX ) XX | | (%XX) XX $(%XX)$ XX | ر |
| | Investigator Global Assessment | Week 52<br>n | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe | Score of Clear or Almost Clear | Success | Failure | 2-Grade Improvement from Baseline | Success | Failure | Score of Clear or Almost Clear Plus 2-Grade Improvement from Baseline | Success | ranure |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.1.2.1: Shift Table of Investigator Global Assessment (IGA) (Safety Population: Cohort 1)

| ARQ-151-201:<br>Roflumilast Cream 0.3% (N=xx) | | | Last Reported IGA | | |
|---|---|---|---|---|---|
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| 1 - Almost Clear | xx (xx.x%) | $XX (XX.X^{0})$ | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx (xx.x%) |
| 2 - Mild | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx ( xx.x%) | $xx (xx.x^{0})$ | xx (xx.x%) |
| 3 - Moderate | xx (xx.x%) | (xx) ( $xx$ | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx (xx.x) |
| 4 - Severe | (xx.x) xx.x | (XX, XX, X) | XX (XX.X) | (xx.x) (xx.x) | xx (xx.x) |
| ARQ-151-201:<br>Rofiumilast Crosm 0 15% (N=vv) | | | I act Renorted IGA | | |
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - Almost Clear | (xx.x) xx | (xx.x) xx.x | ( XX.X%) | (xx.x) xx | xx (xx.x) |
| 2 - Mild | (xx.x) xx.x% | (XX.X) XX | (%X.XX ) XX | (xx.x) xx | (xx.x) |
| 3 - Moderate | $xx (xx.x^{0})$ | xx (xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) |
| 4 - Severe | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx ( xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) |
| ARQ-151-201: | | | | | |
| Vehicle Cream (N=xx) | | | Last Reported IGA | | |
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx ( xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) |
| 1 - Almost Clear | $xx (xx.x^{0})$ | xx (xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) |
| 2 - Mild | xx (xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | $xx (xx.x^{0})$ | xx (xx.x) |
| 3 - Moderate | xx (xx.x%) | xx (xx.x) | xx ( xx.x%) | xx (xx.x) | xx (xx.x%) |
| 4 - Severe | xx (xx.x%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x%) |
| Total (N=xx) | | | Last Reported IGA | | |
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx ( xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) |
| 1 - Almost Clear | xx (xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | xx (xx.x) | xx (xx.x%) |
| 2 - Mild | $xx (xx.x^{0})$ | (xx) ( $xx$ | xx ( xx.x%) | $xx (xx.x^{0})$ | xx (xx.x%) |
| 3 - Moderate | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.2.2: Sensitivity Shift Table of Investigator Global Assessment (IGA) (Safety Population: Cohort 1)

| ARQ-151-201:<br>Roflumilast Cream 0.3% (N=xx) | | | Last Reported IGA | | |
|---|---|---|---|---|---|
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x) | $xx (xx.x^{0})$ |
| 1 - Almost Clear | $xx (xx.x^{0})$ | xx (xx.x%) | xx (xx.x) | $xx (xx.x^{0})$ | xx (xx.x) |
| 2 - Mild | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx (xx.x%) | $xx (xx.x^{0})$ | xx (xx.x) |
| 3 - Moderate | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx (xx.x) | $xx (xx.x^{0})$ | xx (xx.x) |
| 4 - Severe | $XX (XX.X^{0})$ | (XX.XX) | (XX.XX) | (xx.x) (xx.x) | xx (xx.x) |
| ARQ-151-201: | | | | | |
| Roflumilast Cream 0.15% (N=xx) | | | Last Reported IGA | | |
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | $xx (xx.x^{0})$ | xx ( xx.x%) | xx ( xx.x%) | (xx.x) xx $(xx.x)$ | $XX (XX.X^{0})$ |
| 1 - Almost Clear | xx (xx.x%) | (xx.x) xx.x | xx ( xx.x%) | (xx.x) xx $(xx.x)$ | xx ( xx.x%) |
| 2 - Mild | (XX.X) XX | (xx) ( $xx$ ) | (xx.x) | (xx.x) xx | ( xx.x%) |
| 3 - Moderate | (xx.x) xx.x% | xx ( xx.x%) | xx ( xx.x%) | (xx.x) xx $(xx.x)$ | (xx.x) ( $xx.x$ %) |
| 4 - Severe | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx ( xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) |
| ARQ-151-201: | | | | | |
| Vehicle Cream (N=xx) | | | Last Reported IGA | | |
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | $xx (xx.x^{0})$ | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | (xx.x) ( $xx.x$ %) |
| 1 - Almost Clear | xx (xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | $xx (xx.x^{0})$ | xx (xx.x) |
| 2 - Mild | xx (xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | xx (xx.x) | xx (xx.x%) |
| 3 - Moderate | xx (xx.x%) | $xx (xx.x^{0})$ | xx (xx.x%) | $xx (xx.x^{0})$ | xx (xx.x%) |
| 4 - Severe | xx (xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | xx (xx.x) | xx (xx.x%) |
| Total (N=xx) | | | Last Reported IGA | | |
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | $xx (xx.x^{0})$ | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ |
| 1 - Almost Clear | xx (xx.x%) | $xx (xx.x^{0})$ | xx (xx.x) | $xx (xx.x^{0})$ | xx (xx.x%) |
| 2 - Mild | xx (xx.x%) | $xx (xx.x^{0})$ | xx (xx.x%) | $xx (xx.x^{0})$ | xx (xx.x%) |
| 3 - Moderate | xx (xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| 4 - Severe | $xx (xx.x^{0})$ | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Baseline is defined as the last observation prior to entry in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.1.2.3: Shift Table of Investigator Global Assessment (IGA) (Safety Population: Cohort 2)

| <b>Soflumilast Cream 0.3% (N=xx)</b> | | | Last Reported IGA | JA | |
|---|---|---|---|---|---|
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | | 4 - Severe |
| 0 - Clear | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | $(xx.x^{0/0})$ | $xx (xx.x^{0})$ |
| 1 - Almost Clear | xx ( xx.x%) | (xx.x) xx | XX ( XX.X%) | | xx ( xx.x%) |
| 2 - Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | | xx ( xx.x%) |
| 3 - Moderate | $xx (xx.x^{0})$ | xx ( xx.x%) | xx ( xx.x%) | | xx ( xx.x%) |
| 4 - Severe | xx (xx.x%) | xx ( xx.x%) | (xx.x) (xx.x) | | xx (xx.x%) |

Table 14.2.1.2.4: Shift Table of Investigator Global Assessment (IGA) (Safety Population)

| ARQ-151-201:<br>Roflumilast Cream (N=xx) | | | Last Reported IGA | | |
|---|---|---|---|---|---|
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | xx (xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | (xx.x) ( $xx.x$ ) | $XX (XX.X^{0})$ |
| 1 - Almost Clear | $xx (xx.x^{0})$ | xx (xx.x) | $XX (XX.X^{0})$ | (xx.x) ( $xx.x$ ) | $XX (XX.X^{0})$ |
| 2 - Mild | (xx.x) xx | (xx.x) | $XX (XX.X^{0})$ | (0.000) XX $(0.000)$ | XX (XX.X) |
| 3 - Moderate | $xx (xx.x^{0})$ | (xx.x) | $xx (xx.x^{0})$ | (0.000) XX $(0.000)$ | xx ( xx.x%) |
| 4 - Severe | (xx.x) xx | (xx.x) xx. | (XX, XX, X) | (0.000) XX | (xx.x) |
| ARQ-151-201: Vehicle Cream | | | | | , |
| and Cohort 2 (N=xx) | | | Last Reported IGA | | |
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) | $XX (XX.X^{0})$ |
| 1 - Almost Clear | xx (xx.x%) | xx (xx.x%) | $xx (xx.x^{0})$ | (xx.x) ( $xx.x$ ) | xx (xx.x%) |
| 2 - Mild | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx (xx.x) | $xx (xx.x^{0})$ |
| 3 - Moderate | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx (xx.x) | $xx (xx.x^{0})$ |
| 4 - Severe | $xx (xx.x^{0})$ | xx (xx.x) | $xx (xx.x^{0})$ | (xx.x) ( $xx.x$ ) | xx (xx.x%) |
| Total $(N=xx)$ | | | Last Reported IGA | | |
| Baseline IGA | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe |
| 0 - Clear | xx (xx.x%) | xx (xx.x%) | $xx (xx.x^{0})$ | xx (xx.x) | xx (xx.x%) |
| 1 - Almost Clear | $xx (xx.x^{0})$ | xx (xx.x) | $xx (xx.x^{0})$ | (xx.x) ( $xx.x$ ) | $xx (xx.x^{0})$ |
| 2 - Mild | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx (xx.x) | xx ( xx.x%) | $xx (xx.x^{0})$ |
| 3 - Moderate | xx (xx.x%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | $xx (xx.x^{0})$ |
| 4 - Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (%x.xx) xx | xx (xx.x%) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.2.1: Primary Summary of Intrigenous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| | | | ARO-151-202: Roflumilast Cream 0.3% | umilast Cream 0.3% | |
|---|---|---|---|---|---|
| Intertriginous Investigator Global<br>Assessment | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | 1-201:<br>Sream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15%<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | Total (N=xx) |
| $Baseline^a$ | | | | | |
| 1 - Almost Clear | (%xx ) xx | (0) | $\overline{}$ | (%xx ) xx | (%xx ( xx%) |
| 2 - Mild | $\sqrt{xx}$ ) $xx$ | (0) | $\overline{}$ | (%xx ) xx | (%xx ) xx |
| 3 - Moderate | (%xx ) xx | (0) | (%xx ( xx%) | (%xx ) xx | (%xx ) xx |
| 4 - Severe | %xx ) xx | (0) | | (%xx ) xx | (0/xx) $(xx/0)$ |
| ARQ-151-201 Week 2 | | | | | |
| n | XX | | XX | NA | XX |
| 0 - Clear | (%xx ) xx | (0) | $\overline{}$ | | (%xx ) xx |
| 1 - Almost Clear | %xx ) xx | (0) | (%xx ( )xx | | (%xx ) xx |
| 2 - Mild | %xx ) xx | (0) | $\overline{}$ | | (%xx ) xx |
| 3 - Moderate | (%xx ) xx | (0) | $\overline{}$ | | (%xx ) xx |
| 4 - Severe | (%xx ) xx | (0) | (%XX ) XX | | (%xx ) xx |
| Score of Clear or Almost Clear | | | | | |
| Success | (%xx ) xx | (0) | | | (%xx ) xx |
| Failure | (%xx ) xx | (9) | (0/2xx) $(xx)$ | | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.2.1: Primary Summary of Intrigenous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| | | ARO-151-202: Roflumilast Cream 0.3% | unilast Cream 0.3% | |
|---|---|---|---|---|
| Intertriginous Investigator Global<br>Assessment | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | A<br>Roflum | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | Total (N=xx) |
| ARQ-151-201 Week 4 | ; | ; | × 1. | ; |
| | | , | NA | , |
| 0 - Clear | ٠ | | | |
| 1 - Almost Clear | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| 2 - Mild | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| 3 - Moderate | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| 4 - Severe | (%xx ) xx | (%XX ) XX | | (%XX ) XX |
| Score of Clear or Almost Clear | | | | |
| Success | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| Failure | (%XX ) XX | (%XX ) XX | | (%xx ) xx |
| ARQ-151-201 Week 6 | | | | |
| n | XX | XX | NA | XX |
| 0 - Clear | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| 1 - Almost Clear | (%xx ) xx | $\overline{}$ | | (%xx ) xx |
| 2 - Mild | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| 3 - Moderate | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| 4 - Severe | (%xx ) xx | (%XX ) XX | | (%XX ) XX |
| Score of Clear or Almost Clear | | | | |
| Success | (%XX ) XX | (%XX ) XX | | _ |
| Failure | (0%XX ) XX | $\overline{}$ | | (%XX ) XX |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.2.1: Primary Summary of Intrigenous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| | | ARO-151-202: Roffi | ARO-151-202: Roflumilast Cream 0 3% | | |
|---|---|---|---|---|---|
| Intertriginous Investigator Global<br>Assessment | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | A<br>Roflum | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total<br>(N=xx) |
| ARQ-151-201 Week 8 | | | <b>4</b> | | |
| n<br>0 | , | , | NA | XX | (/0 |
| u - Clear | ٠ ر | _ \ | | XX<br>XX | XX%) |
| 1 - Almost Clear | (%XX ) XX | (%XX ) XX | | ) xx | (0%XX |
| 2 - Mild | (%xx ) xx | (%xx ) xx | | ) xx | (%XX |
| 3 - Moderate | (%xx ) xx | xx ( xx%) | | ) xx | (%XX |
| 4 - Severe | (%xx ) xx | (%xx ) xx | | ) xx | (%XX |
| Score of Clear or Almost Clear | | | | | |
| Success | (0%XX ) XX | (%xx ) xx | | ) xx | (%XX |
| Failure | (%xx ) xx | (%XX ) XX | | ) xx | (%XX |
| ARQ-151-201 Week 12 | | | | | |
| n | XX | XX | NA | XX | |
| 0 - Clear | (%xx ) xx | xx ( xx%) | | ) xx | (%XX |
| 1 - Almost Clear | (%xx ) xx | (%xx ( xx%) | | ) xx | (%XX |
| 2 - Mild | (%xx ) xx | (%xx ( xx%) | | ) xx | (%XX |
| 3 - Moderate | (%xx ) xx | (%xx ( xx%) | | ) xx | (%XX |
| 4 - Severe | (%xx ) xx | (%XX) $XX$ | | ) xx | (%XX |
| Score of Clear or Almost Clear | | | | | |
| Success | (0%XX ) XX | (%xx ) xx | | ) xx | (%XX |
| Failure | (%xx ) xx | (%XX ) XX | | ) xx | (%XX |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.2.1: Primary Summary of Intrigenous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| Intertriginous Investigator Global<br>Assessment | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | .01:<br>am 0.3% | AF<br>Roflumi | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Cream (N=xx) | umilast C<br>Al<br>Ve | Cream 0.3% ARQ-151-201: Vehicle Cream (N=xx) | | Total<br>(N=xx) |
|---|---|---|---|---|---|---|---|---|
| Week 4 | × | | XX | | × | | X | |
| 0 - Clear | (%xx ) xx | | ) xx | (0/XX | )<br>XX | (%XX | ) XX | (%xx |
| 1 - Almost Clear | (%xx ) xx | | ) xx | (%XX | , )<br>XX | (%xx | ) xx | (%xx |
| 2 - Mild | | | ) xx | (%XX | XX | (%xx | ) xx | (%xx |
| 3 - Moderate | (%xx ) xx | | ) xx | (%XX | XX | (%XX | ) xx | (%XX |
| 4 - Severe | (%xx ) xx | | ) xx | (%xx | ) xx | (%xx | ) xx | (%XX |
| Score of Clear or Almost Clear | | | | | | | | |
| Success | (%xx ) xx | | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx |
| Failure | (%xx ) xx | | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX |
| Week 12 | | | | | | | | |
| n | XX | | XX | | XX | | XX | |
| 0 - Clear | (%xx ) xx | | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx |
| 1 - Almost Clear | (%xx ) xx | | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx |
| 2 - Mild | (%xx ) xx | | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx |
| 3 - Moderate | (%xx ) xx | | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx |
| 4 - Severe | (%xx ) xx | | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX |
| Score of Clear or Almost Clear | | | | | | | | |
| Success | (%xx ) xx | | ) xx | (0%XX | ) xx | (%XX | ) xx | (%xx |
| Failure | (%xx ) xx | | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.2.1: Primary Summary of Intrigenous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| Intertriginous Investigator Global | ARQ-151-201:<br>Roflumilast Cream 0.3% $(N=xx)$ | AR<br>Offumi | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Crean (N=xx) | milast Cl<br>AF<br>Ve | Cream 0.3% ARQ-151-201: Vehicle Cream | | Total<br>(N=xx) | ĺ |
|---|---|---|---|---|---|---|---|---|
| 11011000001 | (VV VI) | | (WV AT) | | (VV ) I | | (vv ) | İ |
| Week 24 | × | XX | | XX | | XX | | |
| n - Clear | (%XX ) XX | )<br>XX | (%XX | X<br>X | (%xx | XX<br>XX | (%xx | |
| 1 - Almost Clear | (%xx) xx | ( ) xx | (%XX | ×× | (%xx | XX | (%xx | |
| 2 - Mild | (%xx ) xx | ) xx | (%XX | xx ( | (%XX | XX ( | (%xx | |
| 3 - Moderate | (%xx ) xx | ) xx | (%XX | xx ( | (%xx | XX ( | (%xx | |
| 4 - Severe | (%xx ) xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx | |
| Score of Clear or Almost Clear | | | | | | | | |
| Success | (%xx) xx | ) xx | (%XX | ) XX | (%xx | ) xx | (%xx | |
| Failure | (%xx ) xx | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx | |
| Week 36 | | | | | | | | |
| n | XX | XX | | XX | | XX | | |
| 0 - Clear | (%xx ) xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx | |
| 1 - Almost Clear | (%xx ) xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| 2 - Mild | (%xx ) xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| 3 - Moderate | (%xx ) xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| 4 - Severe | (%xx ) xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx | |
| Score of Clear or Almost Clear | | | | | | | | |
| Success | (%xx ) xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx | |
| Failure | (%xx ) xx | ) xx | (%XX | ) XX | (%xx | ) xx | (%XX | |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.2.1: Primary Summary of Intrigenous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| | | ARQ-151-202: Roflumilast Cream 0.3% | milast Cream 0.3% | |
|---|---|---|---|---|
| Intertriginous Investigator Global | ARQ-151-201:<br>Roflumilast Cream 0.3% | A<br>Roflun | ARQ-151-201:<br>Vehicle Cream | Total |
| Assessment | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 52 | | | | |
| n | XX | XX | XX | XX |
| 0 - Clear | (%xx ) xx | _ | _ | |
| 1 - Almost Clear | (%xx ) xx | _ | _ | |
| 2 - Mild | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| 3 - Moderate | (%xx ) xx | | _ | |
| 4 - Severe | (%xx ) xx | | (%xx ) xx | |
| Score of Clear or Almost Clear | | | | |
| Success | (%xx ) xx | (%xx () xx | (%XX ) XX | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast Cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.2.2: Sensitivity Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| | | ARQ-151-202: Rofl | ARQ-151-202: Roflumilast Cream 0.3% | |
|---|---|---|---|---|
| Intertriginous Investigator Global<br>Assessment | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-201: Roflumilast Cream 0.15% (N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | Total<br>(N=xx) |
| $Baseline^a$ | | | | |
| n | XX | XX | XX | XX |
| 1 - Almost Clear | (%xx ) xx | $\overline{}$ | (%xx ) xx | $\overline{}$ |
| 2 - Mild | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx (xx%)) xx |
| 3 - Moderate | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| 4 - Severe | (%xx ) xx | · | (%xx ) xx | · |
| Week 4 | | | | |
| u | XX | XX | XX | XX |
| 0 - Clear | (%xx ) xx | (%xx ) xx | (%XX ) XX | $\overline{}$ |
| 1 - Almost Clear | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| 2 - Mild | (%xx ) xx | (%xx ) xx | (%xx ) xx | |
| 3 - Moderate | (%xx ) xx | (%xx ) xx | (%xx ) xx | $\overline{}$ |
| 4 - Severe | (0/2) XX | (%XX ) XX | (%xx ) xx | (%XX ) XX |
| Score of Clear or Almost Clear Success | (%xx ) xx | (%xx ) xx | (%XX ) XX | (%xx ) xx |
| Failure | (%XX ) XX | (0)XX ) XX | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.2.2: Sensitivity Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| | | | A | ARQ-151-202: Roflumilast Cream 0.3% | milast Cı | ream 0.3% | | | 1 |
|---|---|---|---|---|---|---|---|---|---|
| Intertriginous Investigator Global | ARQ<br>Roflumila | ARQ-151-201:<br>Roflumilast Cream 0.3% | AR<br>Roflumi | ARQ-151-201:<br>Roflumilast Cream 0.15% | AF<br>Ve | ARQ-151-201:<br>Vehicle Cream | | Total | |
| Assessment Week 12 | | (N=xx) | | (N=xx) | | (N=xx) | | (N=xx) | ĺ |
| п | XX | | XX | | XX | | XX | | |
| 0 - Clear | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| 1 - Almost Clear | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | |
| 2 - Mild | _ | (%xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX | |
| 3 - Moderate | _ | (%xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx | |
| 4 - Severe | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| Score of Clear or Almost Clear | | | | | | | | | |
| Success | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx | |
| Failure | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| Week 24 | | | | | | | | | |
| n | XX | | XX | | XX | | XX | | |
| 0 - Clear | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | |
| 1 - Almost Clear | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | |
| 2 - Mild | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | |
| 3 - Moderate | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | |
| 4 - Severe | ) xx | (%XX | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx | |
| Score of Clear or Almost Clear | | | | | | | | | |
| Success | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| Failure | ) XX | (%xx | ) xx | (%XX | ) XX | (%xx | ) xx | (%xx | |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages.

Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.2.2: Sensitivity Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| Intertriginous Investigator Global<br>Assessment | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 % Roflumilast Cream 0.15% Vehicle Crean (N=xx) | umilast Cream 0.3% ARQ-151-201: Vehicle Cream (N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Week 36 n 0 - Clear 1 - Almost Clear | (%xx ) xx<br>(%xx ) xx<br>(xx) xx | xx (%xx ) xx (%) xx (xx ) xx | $\sim$ | xx (%xx ) xx (%) xx (%) |
| 2 - Mild<br>3 - Moderate<br>4 - Severe | (%xx ) xx<br>(xx ) xx<br>(xx ) xx | xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) | xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) | xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) |
| Score of Clear or Almost Clear<br>Success<br>Failure | (%xx ) xx<br>(xx ) xx | xx ( xx%) xx ( xx%) | (%xx ) xx<br>(%xx ) xx | (%xx ) xx (xx%) xx |
| Week 52<br>n<br>0 - Clear | (%xx ) xx | xx<br>xx ( xx%) | (%xx ) xx | xx xx (%) |
| <ul><li>1 - Almost Clear</li><li>2 - Mild</li><li>3 - Moderate</li><li>4 - Severe</li></ul> | xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) | | xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%) | xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( xx%)<br>xx ( x%%) |
| Score of Clear or Almost Clear<br>Success<br>Failure | (%xx ) xx<br>(xx ) xx | xx () xx%) xx () x | (%xx ) xx (xx%) xx (xx%) | xx ( xx%) xx ( xx%) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages.

Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.2.3: Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 2)


| Intertriginous Investigator Global<br>Assessment | Roflumilast Cream 0.3%<br>(N=xx) |
|---|---|
| $\mathrm{Baseline}^{\mathrm{a}}$ | |
| n | XX |
| 0 - Clear | |
| 1 - Almost Clear | (%xx ) xx |
| 2 - Mild | |
| 3 - Moderate | |
| 4 - Severe | (%xx ) xx |
| Week 4 | |
| u | XX |
| 0 - Clear | (%XX ) XX |
| 1 - Almost Clear | |
| 2 - Mild | |
| 3 - Moderate | |
| 4 - Severe | (%xx ) xx |
| Score of Clear or Almost Clear Success Failure | xx ( xx%) xx ( xx%) |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.2.3: Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 2) 

| Intertriginous Investigator Global<br>Assessment | Roflumilast Cream 0.3%<br>(N=xx) | ·• |
|---|---|---|
| Week 12 | | |
| n | | |
| 0 - Clear | $\overline{}$ | |
| 1 - Almost Clear | _ | |
| 2 - Mild | | |
| 3 - Moderate | (%xx ) xx | |
| 4 - Severe | (%xx ) xx | |
| Score of Clear or Almost Clear | | |
| Success | | |
| Failure | (%XX ) XX | |
| West 24 | | |
| ************************************** | | |
| n | | |
| 0 - Clear | $\overline{}$ | |
| 1 - Almost Clear | $\overline{}$ | |
| 2 - Mild | | |
| 3 - Moderate | | |
| 4 - Severe | (%xx ) xx | |
| Come of Close on Almost Close | | |
| Score of Clear of Almost Clear | , | |
| Success | (%xx ) xx | |
| Failure | $\overline{}$ | |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.2.2.3: Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% (N=xx) | | xx ( xxx,0) xx (xx,0) xx ( | | (%xx ) xx (%xx) xx (%xx) | XX | | _ ر | xx ( xx%)<br>xx ( xx%) | (%XX ) XX |
|---|---|---|---|---|---|---|---|---|---|
| Intertriginous Investigator Global<br>Assessment | Week 36 | 1 - Almost Clear 2 - Mild | 3 - Productate<br>4 - Severe | Score of Clear or Almost Clear Success Failure | Week 52<br>n | 0 - Clear | 2 - Mild | 3 - Moderate<br>4 - Severe | Score of Clear or Almost Clear Success |

<sup>&</sup>lt;sup>a</sup> Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.2.4: Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population) 

| | | ARC | )-151-202: Rc | ARQ-151-202: Roflumilast Cream 0.3% | n 0.3% | | 1 |
|---|---|---|---|---|---|---|---|
| | AF | ARO-151-201: | ARQ-Vehicl | ARQ-151-201:<br>Vehicle Cream | | | i. |
| Intertriginous Investigator Global | Rofl | Roflumilast Cream | and C | and Cohort 2 | | Total | |
| Assessment Baseline <sup>a</sup> | | (N=xx) | S | (N=xx) | | (N=xx) | |
| n | XX | | XX | | XX | | |
| 1 - Almost Clear | ) xx | (%XX | | (%x | ) xx | (%xx | |
| 2 - Mild | ) xx | (%XX | | (%x | ) xx | (%XX | |
| 3 - Moderate | ) xx | (%XX | x ) xx | (%xx | ) xx | (%XX | |
| 4 - Severe | ) xx | (%xx | | (%x | ) xx | (%xx | |
| Week 4 | | | | | | | |
| u | XX | | XX | | XX | | |
| 0 - Clear | ) xx | (%XX | $\overline{}$ | (%x | ) xx | (%XX | |
| 1 - Almost Clear | ) xx | (%XX | x ) xx | (%xx | ) xx | (%XX | |
| 2 - Mild | ) xx | (%XX | $\overline{}$ | (%x | ) xx | (%XX | |
| 3 - Moderate | ) xx | (%XX | $\overline{}$ | (%x | ) xx | (%xx | |
| 4 - Severe | ) xx | (%XX | _ | (%x | ) xx | (0%XX | |
| Score of Clear or Almost Clear | | | | | | | |
| Success | ) xx | (%XX | | (%x | ) xx | (%XX | |
| Failure | ) xx | (%XX | x ) xx | (%xx | ) xx | (%XX | |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.2.4: Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population: Cohort 1) 

| | | ARC | ARQ-151-202: Roflumilast Cream 0.3% | last Cream 0.3% | |
|---|---|---|---|---|---|
| Intertriginous Investigator Global | AF<br>Roff | ARQ-151-201:<br>Roflumilast Cream | ARQ-151-201: Vehicle Cream and Cohort 2 | 01:<br>am<br>2 | Total |
| Assessment<br>Week 12 | | (IN-XX) | (XX-NI) | | (IN-XX) |
| n | XX | | XX | XX | |
| 0 - Clear | ) xx | (%XX | $\overline{}$ | XX | (%xx ) |
| 1 - Almost Clear | ) xx | (%XX | (%xx ) xx | XX | (%xx ) |
| 2 - Mild | ) xx | (%XX | $\overline{}$ | XX | (%xx ) |
| 3 - Moderate | ) xx | (%XX | $\overline{}$ | XX | (%xx ) |
| 4 - Severe | ) xx | (%xx | $\overline{}$ | XX | (%xx ) |
| Score of Clear or Almost Clear | | \/\0 | | | ( o |
| Success | ) XX | (0/XX | _ | XX | (0%XX ) |
| Failure | ) xx | (%XX | (%xx ) xx | XX | (%xx ) |
| Week 24 | | | | | |
| n | XX | | XX | XX | |
| 0 - Clear | ) xx | (%XX | $\overline{}$ | XX | (%xx ) |
| 1 - Almost Clear | ) xx | (0%XX | (%xx ) xx | XX | (%xx ) |
| 2 - Mild | ) xx | (%XX | $\overline{}$ | XX | (%xx ) |
| 3 - Moderate | ) xx | (%XX | (%xx ) xx | XX | (%xx ) |
| 4 - Severe | ) xx | (%xx | $\overline{}$ | XX | (%xx ) |
| Score of Clear or Almost Clear | | | | | |
| Success | ) xx | (%XX | (%xx ) xx | XX | (%xx ) |
| Failure | ) xx | (%xx | (%xx ) xx | XX | (%xx ) |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.2.4: Summary of Intertriginous Investigator Global Assessment (I-IGA) (Safety Population) 

| | | ARO | -151-202: Rof | ARQ-151-202: Roflumilast Cream 0.3% | .3% | |
|---|---|---|---|---|---|---|
| | ARO. | ARO-151-201: | ARQ-151-201:<br>Vehicle Cream | 1-201:<br>Cream | | |
| Intertriginous Investigator Global | Roflum | Roflumilast Cream | and Cohort 2 | hort 2 | | Total |
| Week 36 | | (VV-) | | ) | | (YV-VI) |
| n | XX | | XX | | XX | |
| 0 - Clear | x ) xx | (%x | (%xx ) xx | (0) | ) xx | (%xx |
| 1 - Almost Clear | x ) xx | (%xx | (%xx ) xx | (0) | ) xx | (%xx |
| 2 - Mild | x ) xx | (%x | $xx$ ( $xx^{0}$ | (0) | ) xx | (%XX |
| 3 - Moderate | x ) xx | (%x | $\mathbf{x}\mathbf{x}$ ) $\mathbf{x}\mathbf{x}$ | (0) | ) xx | (%xx |
| 4 - Severe | x ) xx | x%) | (%xx ) xx | (%) | ) xx | (%xx |
| Score of Clear or Almost Clear | | | | | | |
| Success | x ) xx | (%xx | (%xx ) xx | (0) | ) xx | (%xx |
| Failure | x ) xx | (%x | ) xx | (%) | ) xx | (%XX |
| Week 52 | | | | | | |
| n | XX | | XX | | XX | |
| 0 - Clear | x ) xx | (%x | (%xx ) xx | (0) | ) xx | (%xx |
| 1 - Almost Clear | x ) xx | (%x | $xx$ ( $xx^{0}$ | (0) | ) xx | (%xx |
| 2 - Mild | x ) xx | (%XX | (%xx ) xx | (0) | ) xx | (%XX |
| 3 - Moderate | x ) xx | (%x | (%xx ) xx | (0) | ) xx | (%xx |
| 4 - Severe | x ) xx | (%x | (%xx ) xx | (0) | ) xx | (%xx |
| Score of Clear or Almost Clear | | | | | | |
| Success | $\overline{}$ | (%XX | $\overline{}$ | (0) | ) xx | (%xx |
| Failure | x ) xx | (%x | (%xx ) xx | (%) | ) xx | (%XX |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Collected for subjects with intertriginous involvement. Subjects reporting no intertriginous area involvement are included in denominator for percentages. Note: Collected post-baseline for subjects with a severity of at least mild. No imputation of missing values. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.2.3.1: Primary Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201: ARQ-151-201: | Roflumilast Cream 0.3% Roflumilast Cream 0.15% Vehicle Cream Total | $(N=xx) \qquad (N=xx) \qquad (N=xx)$ | | XX XX XX XX XX XX | XX XX XX XX | XX.XX XX.XX XX.XX | XX XX XX XX | vy ct vy vy vy ct vy vy vy ct vy |
|---|---|---|---|---|---|---|---|---|---|
| | ARQ-151-201: | Roflumilast Cream 0.3% | rea and Severity Index | Baseline <sup>a</sup> | | Mean | | | Min to May |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.2.3.1: Primary Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| | Total | (N=xx) | | XX | XX | XX.X | XX | xx to xx | | XX.X | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%XX ) XX | (%xx ) xx | | (%XX ) XX | (%XX ) XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ilast Cream 0.3% | ARQ-151-201:<br>Vehicle Cream | (N=xx) | | NA | | | | | | | | | | | | | | | | | | | | |
| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | (N=xx) | | XX | XX | XX.X | xx | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%xx ) xx | (%xx ) xx | | (%xx ) xx | (%XX ) XX |
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | (N=xx) | | XX | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%xx ) xx | (%XX ) XX | | (%xx ) xx | (%xx ) xx |
| | | Psoriasis Area and Severity Index | ARQ-151-201 Week 2 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>PASI-50</u> | Success | Failure | <u>PASI-75</u> | Success | Failure |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

Table 14.2.3.1: Primary Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| | ABO-151-201: | ARO-151-202: INSTRUMENTAL CLEGITI 0:370<br>ARO-151-201: ARO-151-20 | ARO-151-201 | |
|---|---|---|---|---|
| | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total |
| Psoriasis Area and Severity Index | (N=XX) | (N=xx) | (N=xx) | (N=xx) |
| 101 201 WCCN 1 | XX | XX | NA | XX |
| Mean | XX | XX | | XX |
| 0 | XX.X | XX.X | | XX.X |
| edian | XX | XX | | XX |
| in. to Max. | xx to xx | xx to xx | | xx to xx |
| nange from Baseline | | | | |
| Mean | XX | XX | | XX.X |
| SD | XX.X | XX.X | | XX.X |
| Median | XX | XX | | XX |
| Min. to Max | xx to xx | xx to xx | | xx to xx |
| rcent Change from Baseline | | | | |
| Mean | XX | XX | | XX |
| SD | XX.X | XX.X | | XX.X |
| Median | XX | XX | | XX |
| Min. to Max. | xx to xx | xx to xx | | xx to xx |
| <u>PASI-50</u> | | | | |
| Success | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | | (%XX ) XX |
| PASI-75 | | | | |
| Success | (%xx ) xx | (%xx ) xx | | (%XX ) XX |
| Failure | (%xx ) xx | (%xx ) xx | | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

Table 14.2.3.1: Primary Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| Profitatis ARQ-151-201: ARQ-152-201: AR | | | ARQ-151-202: Roflumilast Cream 0.3% | ilast Cream 0.3% | |
|---|---|---|---|---|---|
| N | | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| Baseline xx xx x xx x xx x xx x xx xx x | Psoriasis Area and Severity Index | (N=XX) | (N=xx) | (N=xx) | (N=xx) |
| xx | n n | XX | XX | NA | X |
| xx | Mean | XX | XX | | XX |
| xx | SD | XX.X | XX.X | | XX.X |
| xx | Median | XX | XX | | XX |
| xx | Min. to Max. | xx to xx | xx to xx | | xx to xx |
| xxx xxx xxx xx | Change from Baseline | | | | |
| xx | Mean | XX | XX | | XX.X |
| xx xx bxx xx | SD | XX.X | XXX.X | | XX.X |
| xx | Median | XX | XX | | XX |
| xx | Min. to Max | xx to xx | xx to xx | | xx to xx |
| xx, | Percent Change from Baseline | | | | |
| xx. xx. xx x | Mean | XX | XX | | XX |
| xx xx< | SD | XX.X | XX.X | | XX.X |
| Max. xx to xx xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xx%) xx (xxx%) xx (xxx%) xx (xxx%) xx (xxx%) xx (xxx%) xx (xxx%) xx (xxxX) xx (xxxX) xx (xxxX) xx (xxxX) xx (xxxX) xx (xxxX) xx (xxxX) xx (xxxX) xx (xxxX) </td <td>Median</td> <td>XX</td> <td>XX</td> <td></td> <td>XX</td> | Median | XX | XX | | XX |
| ) xx (%xx ) xx (%xx ) xx (xx ) | Min. to Max. | xx to xx | xx to xx | | xx to xx |
| XX ( XX ) XX ( XX%) XX ( XX ) XX ( X | <u>PASI-50</u> | | | | |
| ) xx ( 0,0 xx ) | Success | $\overline{}$ | | | |
| ) xx ( $\%$ xx ( $\%$ xx ) xx ( $\%$ xx ( $\%$ xx ( $\%$ xx ) xx ( $\%$ xx ( $\%$ xx ( $\%$ xx ) xx ( $\%$ xx ( $\%$ xx ( $\%$ xx ) xx ( $\%$ x ( $\%$ xx ( $\%$ x ( | Failure | $\overline{}$ | $\overline{}$ | | $\overline{}$ |
| ) $xx ( xx / xx ) xx ( xx / xx ) xx$ | PASI-75 | | | | |
| ) XX $(\%XX)$ XX $(\%XX)$ XX | Success | $\overline{}$ | | | $\overline{}$ |
| | Failure | | | | $\overline{}$ |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

Table 14.2.3.1: Primary Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| | A BO 151 301 | ARQ-131-202; Rollumiast Cream 0.5% | Mast Cleam 0.370 | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-131-201:<br>Vehicle Cream | Total |
| Psoriasis Area and Severity Index<br>ARO-151-201 Week 8 | (X=X) | (N=XX) | (N=xx) | (N=xx) |
| | XX | xx | NA | XX |
| | XX | XX | | XX |
| | XX.X | XX.X | | XX.X |
| | XX | XX | | XX |
| Max. | xx to xx | xx to xx | | xx to xx |
| Change from Baseline | | | | |
| | XX | XX | | XX.X |
| | XX.X | XX.X | | XX.X |
| TI TI | XX | XX | | XX |
| o Max | xx to xx | xx to xx | | xx to xx |
| Percent Change from Baseline | | | | |
| | XX | XX | | XX |
| | XX.X | XX.X | | XX.X |
| п | XX | XX | | XX |
| Min. to Max. | xx to xx | xx to xx | | xx to xx |
| | (%xx ) xx | (%xx ) xx | | (%xx) xx |
| 3 0 | <i>_</i> | | | _ ر |
| PASI-75 | | | | |
| SS | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| Failure | (%XX ) XX | (%xx ) xx | | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

Table 14.2.3.1: Primary Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| Psoriasis Area and Severity Index | ARQ-151-201:<br>Roflumilast Cream $0.3\%$<br>(N=xx) | ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Cream (N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| ARQ-151-201 Week 12 | | | | |
| | XX | XX | NA | XX |
| | XX | XX | | XX |
| | XXX.X | XXX.X | | XXX.X |
| | XX | XX | | XX |
| ×. | xx to xx | xx to xx | | xx to xx |
| m Baseline | | | | |
| | XX | XX | | XX.X |
| | XX.X | XX.X | | XX.X |
| | XX | XX | | XX |
| Лах | xx to xx | xx to xx | | xx to xx |
| Percent Change from Baseline | | | | |
| | XX | XX | | XX |
| | XX.X | XX.X | | XX.X |
| | XX | XX | | XX |
| Max. | xx to xx | xx to xx | | xx to xx |
| <u>PASI-50</u> | | | | |
| | (%xx ) xx | (%xx ) xx | | (%xx) xx |
| | (%xx ) xx | (%xx ) xx | | (%xx) xx |
| | (0/xx) xx | (%xx ) xx | | (%xx) xx |
| | (%XX ) XX | (%xx ) xx | | (%xx) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

Table 14.2.3.1: Primary Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| Psoriasis Area and Severity Index Week 4 Nean Mean Median Min. to Max. SD Min. to Max. Median Min. to Max. SD Min. to Max. SD Min. to Max. Median Min. to Max. Min. to Max. Min. to Max. Min. to Max. Median Min. to Max. Min. to Max. Min. to Max. Median Median Min. to Max. Median Median Min. to Max. Median Min. to Max. Median Median Min. to Max. Median Median Min. to Max. Median Min. to Max. Median Median Min. to Max. Median Med | 201: ARQ-151-201: am $0.3\%$ Roflumilast Cream $0.15\%$ | ARO-151-201 | |
|---|---|---|---|
| <b>'</b> | | Vehicle Cream | Total |
| XX | | (N=xx) | (N=XX) |
| XX | | | |
| XX | XX | XX | XX |
| X X X X | XX | XX | XX |
| × | X XX.X | XX.X | XX.X |
| | XX | XX | XX |
| XX XX XX | xx xx xx to xx | xx to xx | xx to xx |
| XX | | | |
| XX | XX | XX | XX.X |
| XX | X XX.X | XX.X | XX.X |
| XX XX XX | XX | XX | XX |
| XX | XX XX XX to XX | xx to xx | xx to xx |
| XX XX XX | | | |
| XX XX | XX | XX | XX |
| xx to xx | XX.X | XX.X | XX.X |
| ) XX | XX | XX | XX |
| ) XX | xx xx xx to xx | xx to xx | xx to xx |
| ) XX | | | |
| ) ^^ | (%) xx (%) (%) | (%xx ) xx | (%xx) xx |
| ) vv | (%) xx (%xx) (%) | (%xx ) xx | (%xx ) xx |
| <u>PASI-75</u> | | | |
| Success xx (xx%) | ) XX | (%xx ) xx | (%xx ) xx |
| Failure xx (xx%) | (%) xx (0%) | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

Note to the programmer: Repeat this page for Week 12, 24, 36 and 52.

TOOL.AN.10-01.01 Statistical Analysis Plan Template
Table 14.2.3.2: Sensitivity Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| VV VV VV |
|----------|
|----------|

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

Table 14.2.3.2: Sensitivity Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| | ARQ-151-201:<br>Roflumilast Cream 0 3% | ARQ-151-201:<br>Roflumilast Cream 0 15% | ARQ-151-201:<br>Vehicle Cream | Total |
|---|---|---|---|---|
| Psoriasis Area and Severity Index | (N=XX) | (N=xx) | (N=xx) | (N=xx) |
| Week 4 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | XX | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| <u>PASI-50</u> | | | | |
| Success | (%xx () xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%XX ) XX |
| <u>PASI-75</u> | | | | |
| Success | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.3.2: Sensitivity Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| | A RO_151_201 | ARO-151-201: | A RO-151-201 | |
|---|---|---|---|---|
| | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total |
| Psoriasis Area and Severity Index<br>Week 12 | (N=XX) | (N=xx) | (N=xx) | (N=xx) |
| u | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | XX | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| <u>PASI-50</u> | | | | |
| Success | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%XX) XX |
| Failure | (%xx ) xx | (%xx ) xx | xx ( xx%) | (%XX ) XX |
| PASI-75 | | | | |
| Success | (%xx ) xx | (0%XX ) XX | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (0%XX ) XX | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.3.2: Sensitivity Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| | | ARQ-151-202: Roflumilast Cream 0.3% | ilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | |
| | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total |
| <b>Psoriasis Area and Severity Index</b> | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 24 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| <u>PASI-50</u> | | | | |
| Success | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| <u>PASI-75</u> | | | | |
| Success | (%XX ) XX | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.3.2: Sensitivity Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| | | ARQ-151-202: Roflumilast Cream 0.3% | ilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | |
| | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total |
| <b>Psoriasis Area and Severity Index</b> | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Week 36 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| <u>PASI-50</u> | | | | |
| Success | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| <u>PASI-75</u> | | | | |
| Success | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.3.2: Sensitivity Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 1) 

| ARQ-151-201: .3% Roflumilast Cream 0.15% | | | ARO-151-202: Roflumilast Cream 0.3% | nilast Cream 0.3% | |
|---|---|---|---|---|---|
| N | | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | Total |
| xx | soriasis Area and Severity Index | KOHUMMIASI CIEAM 0.3% $(N=xx)$ | Komumiasi Cream 0.13% $(N=xx)$ | v enicie Cream<br>(N=xx) | N=XX |
| xx | Week 52 | | | | |
| xx | n | XX | XX | XX | XX |
| xx xx xx xx xx | Mean | XX | XX | XX | XX |
| xx | SD | XX.X | XX.X | XX.X | XX.X |
| xx | Median | XX | XX | XX | XX |
| xx | Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| xx. | Change from Baseline | | | | |
| xx.x xx.x xx xx to xx xx xx xx.x xx.x xx.x xx.x xx xx xx xx xx xx to xx xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) | Mean | XX | XX | XX | XX |
| xx | SD | XX.X | XX.X | XX.X | XX.X |
| xx xx bxx xx | Median | XX | XX | xx | XX |
| xx | Min. to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| xx, | Percent Change from Baseline | | | | |
| xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. xx. <td>Mean</td> <td>XX</td> <td>XX</td> <td>XX</td> <td>XX</td> | Mean | XX | XX | XX | XX |
| xx xx< | SD | XX.X | XX.X | XX.X | XX.X |
| dax. xx to xx xx to xx xx to xx xx xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) xx ( xx%) | Median | XX | XX | XX | XX |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| ) xx (%xx ) xx (%xx ) xx (%xx ) xx (xx | <u>PASI-50</u> | | | | |
| ) xx (%xx ) xx (%xx ) xx (%xx ) xx (%xx ) xx ( %xx ) xx | Success | $\overline{}$ | | | $\overline{}$ |
| ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) $xx$ (% $xx$ ) $xx$ | Failure | | | | |
| ) xx ( %xx ) xx ( xx%) xx | PASI-75 | | | | |
| ) XX $(0.00000000000000000000000000000000000$ | Success | $\overline{}$ | | | $\overline{}$ |
| | Failure | $\overline{}$ | $\overline{}$ | $\overline{}$ | $\overline{}$ |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.3.3: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 2) 

| n 0.3% | | | | | |
|---|---|---|---|---|---|
| Roflumilast Cream $0.3\%$ $(N=xx)$ | XX | XX | XXX.X | XX | xx to xx |
| Psoriasis Area and Severity Index<br>Baseline | u | Mean | SD | Median | Min. to Max. |

Table 14.2.3.3: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% | (xx=N) | XX | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%XX ) XX | (%XX ) XX | | (%XX ) XX | (%XX ) XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Psoriasis Area and Severity Index<br>Week 4 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>PASI-50</u> | Success | Failure | PASI-75 | Success | Failure |

Table 14.2.3.3: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% $(N=xx)$ | ×× | ···· XX | XX.X | XX | xx to xx | | XX | XX.X | XX | XX to XX | | XX | XX.X | XX | XX to XX | | (%XX ) XX | (%XX ( ) XX | | (%XX ) XX | (%XX ) XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Psoriasis Area and Severity Index | Week 12<br>n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>PASI-50</u> | Success | Failure | PASI-75 | Success | Failure |

Table 14.2.3.3: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% | (x=N) | | XX | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%XX ) XX | (%XX ) XX | | (%XX ) XX | xx ( xx%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Psoriasis Area and Severity Index | Week 24 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>PASI-50</u> | Success | Failure | PASI-75 | Success | Failure |

Table 14.2.3.3: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% | (xx=N) | XX | XX | XX.X | XX | XX to XX | | XX | XXX.X | XX | XX to XX | | XX | XX.X | XX | XX to XX | | (%XX ( XX%) | (%XX ) XX | | (%XX ) XX | (%XX ) XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Psoriasis Area and Severity Index<br>Week 36 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>PASI-50</u> | Success | Failure | <u>PASI-75</u> | Success | Failure |

Table 14.2.3.3: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% (N=xx) | XX | XX | XX.X | XX | XX to XX | | XX | XX.X | XX | XX to XX | | XX | XX.X | XX | XX to XX | | (%XX ) XX | (%XX ) XX | | (%XX ) XX | (%xx ) xx |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Psoriasis Area and Severity Index<br>Week 52 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>PASI-50</u> | Success | Failure | <u>PASI-75</u> | Success | Failure |

Table 14.2.3.4: Summary of Psoriasis Area and Severity Index (PASI)
(Safety Population)


| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201: Vehicle Cream | _ | $(N=xx) \qquad (N=xx)$ | | XX XX XX | XX XX XX | XX.XX XX.XX | XX XX XX | xx to xx |
|---|---|---|---|---|---|---|---|---|---|
| | | | Psoriasis Area and Severity Index | Baseline <sup>a</sup> | n | Mean | SD | Median | Min. to Max. |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.3.4: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population) 

| ARO-151-202: Roflumilast Cream 0.3% | ARQ-151-201: | ARQ-151-201: Vehicle Cream | Roflumilast Cream and Cohort 2 Total | $\frac{(N=xx)}{(N=xx)} \qquad \frac{(N=xx)}{(N=xx)}$ | | XX XX XX | XX XX XX | XX.X XX.X XX.X | XX XX XX | XX to XX | | XX XX.X | XX.X XX.X | XX XX XX | XX to XX | ne | XX XX XX | XX.X XX.X XX.X | XX XX XX | XX to XX | | (%XX) XX $(%XX)$ XX $(%XX)$ XX | ) $xx (0.0000000000000000000000000000000000$ | | (%xx ) xx (%xx ) xx (%xx ) xx |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Psoriasis Area and Severity Index | Week 4 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>PASI-50</u> | Success | Failure | PASI-75 | Success |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

Table 14.2.3.4: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population) 

| ARO-151-202: Roflumilast Cream 0.3% | ARQ-151-201: | ARQ-151-201: Vehicle Cream | Roflumilast Cream and Cohort 2 Total | $(N=xx) \qquad (N=xx) \qquad (N=xx) \qquad (N=xx)$ | | xx xx xx | XX XX XX | XX.X XX.X | XX XX XX | XX to XX | | XX XX.X | XX.X XX.X | XX XX XX | XX to XX XX to XX XX to XX | Saseline | XX XX XX | XX.X XX.X | XX XX XX | XX to XX | | (%XX) $(XX)$ $(XX)$ $(XX)$ $(XX)$ $(XX)$ | ) $XX$ ( $\%X$ ) $XX$ ( $\%X$ ) $XX$ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Psoriasis Area and Severity Index | Week 12 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | PASI-50 | Success | Failure | PASI-75 | Character |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.3.4: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population) 

| Week 24 n Mean SD Median Min. to Max. Change from Baseline Median Min. to Max Percent Change from Baseline Mean SD Median Min. to Max Percent Change from Baseline Mean SD Mean Min. to Max SD Median Min. to Max. | Roflumilast Cream (N=xx) xx xx xxx xxx xx | Vehicle Cream and Cohort 2 (N=xx) xx | Total (N=xx) xx |
|---|---|---|---|
| ASI-50<br>Success<br>Failure<br>ASI-75<br>Success<br>Failure | (%xx ) xx<br>(%xx ) xx<br>(%xx ) xx<br>(%xx ) xx | (%xx ) xx<br>(xx ) xx<br>(xx ) xx<br>(xx ) xx | (%XX ) XX<br>(%XX ) XX<br>(%XX ) XX |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

Table 14.2.3.4: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population) 

| ARQ-151-2 | ARQ-151-201: Vehicle Cream<br>Roflumilast Cream and Cohort 2 | (XX=X) | XX XX XX | XX XX XX | XX.X XX.X | XX XX XX | . xx to xx | l Baseline | XX XX XX | XXX.X XX.XX | XX XX XX | ax xx to xx xx to xx xx to xx xx to xx | nge from Baseline | XX XX XX | XXX.X XX.XX | XX XX XX | ax. xx to xx xx to xx xx to xx xx to xx | | ) XX $(\%XX)$ XX $(\%XX)$ XX | ) xx | | | ) XX (0%XX ) XX | nd Severity Index I Baseline ax ax age from Baseline ax. | ARQ-151-201: Roflumilast Cream (N=xx) | ARQ-151-201: Vehicle Cream and Cohort 2 (N=xx) xx | L L X X X X X X X X X X X X X X X X X X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | oriasis Area and Severity Index<br>Week 36 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | PASI-50 | Success | Failure | PASI-75 | Success | :<br>: | Psoriasis Area and Severity Index Week 36 n Mean SD Median Min. to Max. Change from Baseline Mean SD Median Min. to Max Percent Change from Baseline Mean SD Median Min. to Max Percent Change from Baseline Min. to Max Percent Change from Baseline Min. to Max Percent Change from Baseline Min. to Max Percent Change from Baseline Min. to Max. Parlure Success Failure PASI-75 Success Failure Failure Failure Failure | | | ARQ-151-201: Roflumilast Cream |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

Table 14.2.3.4: Summary of Psoriasis Area and Severity Index (PASI) (Safety Population) 

| ARO-151-202: Roflumilast Cream 0.3% | ARQ-151-201: | Roflumilast Cream and Cohort 2 Total | V Index $V$ | | xx xx xx | XX XX XX | XX.X XX.X | XX XX XX | XX to XX XX XX to XX | | XX XX XX | XX.X XX.X | XX XX XX | XX to XX XX XX to XX XX to XX | seline | XX XX XX | XX.X XX.X | XX XX XX | XX to XX XX XX to XX XX to XX | | (% XX) $(XX)$ $(XX)$ $(XX)$ $(XX)$ $(XX)$ | ) XX $(\%XX)$ XX $(\%XX)$ XX | | (%aa ) aa | ) $\nabla v = (\rho/\nabla v) \nabla v = (\rho/\nabla v) \nabla v$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Psoriasis Area and Severity Index | Week 52 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>PASI-50</u> | Success | Failure | PASI-75 | Success | |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

Note: No imputation of missing values. PASI-50 is defined as a 50% reduction from baseline of PASI. PASI-75 is defined as a 75% reduction from Baseline of PASI.

PASI.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.1: Primary Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
|---|---|---|---|---|
| Modified Psoriasis and Severity Index | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Baseline <sup>a</sup> | | | | |
| n | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| ARQ-151-201 Week 2 | | | | |
| n | XX | XX | NA | XX |
| Mean | XX | XX | | XX |
| SD | XX.XX | XX.XX | | XX.XX |
| Median | XX | XX | | XX |
| Min. to Max. | xx to xx | xx to xx | | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | | XX |
| SD | XX.XX | XX.XX | | XX.XX |
| Median | XX | XX | | XX |
| Min. to Max | xx to xx | xx to xx | | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | | XX |
| SD | XX.XX | XX.XX | | XX.XX |
| Median | XX | XX | | XX |
| Min. to Max.<br>mPASI-75 | xx to xx | xx to xx | | xx to xx |
| Success | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| Failure | (/0*** / *** | (/0**** ) **** | | (/0 |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.4.1: Primary Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| | | | , | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| Modified Psoriasis and Severity Index<br>ARQ-151-201 Week 4 | (xx=N) | (xx=N) | (N=XX) | (N=XX) |
| n | XX | XX | NA | XX |
| Mean | XX | XX | | XX |
| SD | XX.X | XX.X | | XX.X |
| Median | XX | XX | | XX |
| Min. to Max. | xx to xx | xx to xx | | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | | XX.X |
| SD | XX.X | XX.X | | XX.X |
| Median | XX | XX | | XX |
| Min. to Max | xx to xx | xx to xx | | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | | XX |
| SD | XX.X | XX.X | | XX.X |
| Median | XX | XX | | XX |
| Min. to Max. | xx to xx | xx to xx | | xx to xx |
| S 2000017 | | | | |
| Success | (0%XX ) XX | (0%XX ) XX | | (%XX ) XX |
| Failure | (%xx ) xx | (%XX ) XX | | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.1: Primary Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| eam 0.3% | ARQ-151-201:<br>Vehicle Cream Total | | NA | XX | XX.X | XX | xx to xx | | XX.X | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | (%xx ) xx | $(\%^{\alpha})$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201: AR<br>Roflumilast Cream 0.15% Ve | | XX | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | (%xx ) xx | (70222) 222 |
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | (N=XX) | XX | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | (%xx) xx | (70'22') '22' |
| | | <b>Modified Psoriasis and Severity Index</b><br>ARQ-151-201 Week 6 | u | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max.<br>mPASI-75 | Success | D.:11::00 |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.1: Primary Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.4.1: Primary Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | Total |
|---|---|---|---|---|
| Modified Psoriasis and Severity Index<br>ARQ-151-201 Week 12 | Notinitiasi Creatii 0.3 % (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| u | XX | XX | NA | XX |
| Mean | XX | XX | | XX |
| SD | XX.X | XX.X | | XX.X |
| Median | XX | XX | | XX |
| Min. to Max. | xx to xx | xx to xx | | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | | XX.X |
| SD | XX.X | XX.X | | XXXX |
| Median | XX | XX | | XX |
| Min. to Max | xx to xx | xx to xx | | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | | XX |
| SD | XX.X | XX.X | | XX.X |
| Median | XX | XX | | XX |
| Min. to Max.<br>mPASI-75 | xx to xx | xx to xx | | xx to xx |
| Success | (%xx ) xx | (%xx ) xx | | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | | (%xx) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.1: Primary Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| | ARQ-151-201: | ARQ-151-202: Rotlumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Doctumilast Cream 0.15% Valigle Cream | ARQ-151-201:<br>Vehicle Creem | Total |
|---|---|---|---|---|
| Modified Psoriasis and Severity Index<br>Week 4 | NOTION (N=XX) | (N=xx) | (N=xx) | 10tat<br>(N=xx) |
| | XX | XX | XX | XX |
| | XX | XX | XX | XX |
| | XX.X | XX.X | XX.X | XX.X |
| | XX | XX | XX | XX |
| Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| from Baseline | | | | |
| | XX | XX | XX | XX.X |
| | XX.X | XX.X | XX.X | XX.X |
| an | XX | XX | XX | XX |
| to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | | |
| | XX | XX | XX | XX |
| | XX.X | XX.X | XX.X | XX.X |
| an | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Success | (%xx ) xx | (%xx ) xx | (%XX ) XX | (%XX ) XX |
| Failure | (%XX) XX | (%xx ) xx | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note to the programmer: Repeat this page for Week 12, 24, 36 and 52.

Table 14.2.4.2: Sensitivity Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
|---|---|---|---|---|
| Modified Psoriasis and Severity Index Baseline <sup>a</sup> | (N=XX) | (N=xx) | (N=xx) | (XX=N) |
| n | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Week 4 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX | XX | XX | XX |
| Min. to Max.<br>mP ASI-75 | xx to xx | xx to xx | xx to xx | xx to xx |
| Success | (%XX ) XX | (%XX ) XX | (%XX ) XX | (%xx ) xx |
| Failure | (%xx ) xx | (%XX ) XX | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.4.2: Sensitivity Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| | ARQ-151-201: | ARQ-151-202: Roflumilast Cream 0.3%<br>ARQ-151-201: ARQ-151-20 | nilast Cream 0.3%<br>ARQ-151-201: | |
|---|---|---|---|---|
| Modified Psoriasis and Severity Index<br>Week 12 | Roflumilast Cream 0.3%<br>(N=xx) | Roflumilast Cream 0.15% (N=xx) | Vehicle Cream (N=xx) | $\begin{array}{c} \text{Total} \\ \text{(N=xx)} \end{array}$ |
| | XX | XX | XX | XX |
| | XX | XX | xx | XX |
| | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| | xx to xx | xx to xx | xx to xx | xx to xx |
| | XX | XX | XX | XX.X |
| | XX.X | XX.X | XX.X | XX.X |
| | XX | XX | xx | XX |
| | xx to xx | xx to xx | xx to xx | xx to xx |
| line | | | | |
| | XX | XX | XX | XX |
| | XX.X | XX.X | XX.X | XX.X |
| | XX | XX | XX | XX |
| | xx to xx | xx to xx | xx to xx | xx to xx |
| | (%xx ) xx | (%xx ) xx | (%XX ) XX | (%XX ) XX |
| | (%xx ) xx | (%xx ) xx | (%XX ) XX | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.2: Sensitivity Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| | | ARQ-151-202: Roflumilast Cream 0.3% | nilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| Modified Psoriasis and Severity Index<br>Week 24 | (N=xx) | (N=xx) | (N=XX) | (N=XX) |
| n | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max.<br>mPASI-75 | xx to xx | xx to xx | xx to xx | xx to xx |
| Success | (%xx ) xx | (%xx ) xx | (0/xx) $xx$ | (%xx ) xx |
| Failure | (%XX ) XX | (%XX ) XX | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.2: Sensitivity Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| | | ARQ-151-202: Roflumilast Cream 0.3% | ilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| <b>Modified Psoriasis and Severity Index</b><br>Week 36 | (x=N) | (N=xx) | (xx=N) | (X=X) |
| n | XX | XX | XX | XX |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | | |
| Mean | XX | XX | XX | XX |
| SD | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX |
| Min. to Max.<br>mPASI-75 | xx to xx | xx to xx | xx to xx | xx to xx |
| Success | (%xx ) xx | (%xx ) xx | (%xx ) xx | (0/2) XX |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx | (0/xx) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.2: Sensitivity Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 1) 

| Cream 0.3% ARQ-151-201: Valida Craam | | XX | XX | XX.X XX.X | XX | xx to xx xx to xx | | XX | XX.X XX.X | XX | xx to xx xx to xx | | XX | XX.X | XX | xx to xx xx xx to xx | | (%xx) xx $(%xx)$ | (%XX) XX $(%XX)$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-201: ARQ-151-20 | | XX | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | ) xx (0%xx ) xx | xx (%xx ) xx |
| ARQ-151-201: | Notiumas Cream 0.5 % (N=xx) | XX | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%xx ) xx | (%xx ) xx |
| | Modified Psoriasis and Severity Index<br>Week 52 | п | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | mPASI-75 | Success | Failure |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.3: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 2) 

| % | | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | XX | XX | XX.X | XX | xx to xx | | XX | XX | XX.X | XX | xx to xx | | XX | XXX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%xx ) xx | (%xx ) xx |
| Modified Psoriasis and Severity Index<br>Baseline | n | Mean | SD | Median | Min. to Max. | Week 4 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | mPASI-75 | Success | Failure |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.3: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% (N=xx) | XX | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%XX ) XX | xx ( xx%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Modified Psoriasis and Severity Index<br>Week 12 | п | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | mPASI-75 | Success | Failure |

Table 14.2.4.3: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% (N=xx) | XX | XX | XXX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XXX.X | XX | xx to xx | | XX ( xX%) | (%XX ) XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Modified Psoriasis and Severity Index</b><br>Week 24 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | <u>mPASI-75</u> | Success | Failure |

Table 14.2.4.3: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% | (N=xx) | | XX | XX | XX.X | XX | XX to XX | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%XX ) XX | xx ( xx%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Modified Psoriasis and Severity Index | Week 30 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | mPASI-75 | Success | Failure |

Table 14.2.4.3: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population: Cohort 2)

| (Saiot) 1 oparation: Conort 2) |
|--------------------------------|

| Roflumilast Cream 0.3% | (N=xx) | XX | XX | XXX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | XX | XX.X | XX | xx to xx | | (%XX ) XX | xx ( xx%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Modified Psoriasis and Severity Index<br>Week 52 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | Mean | SD | Median | Min. to Max | Percent Change from Baseline | Mean | SD | Median | Min. to Max. | mPASI-75 | Success | Failure |

Table 14.2.4.4: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population) 

| .3% | | | Total | (N=xx) | | XX | XX | XX.XX | XX | xx to xx |
|---|---|---|---|---|---|---|---|---|---|---|
| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201: | Vehicle Cream | and Cohort 2 | (N=xx) | | XX | XX | XX.XX | XX | xx to xx |
| ARQ-15 | | ARQ-151-201: | Roflumilast Cream | (N=xx) | | XX | XX | XX.XX | XX | xx to xx |
| | | | | Modified Psoriasis and Severity Index | Baseline <sup>a</sup> | n | Mean | SD | Median | Min. to Max. |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.4.4: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population) 

| Modified Psoriasis and Severity Index Week 4 n Mean SD Median Min. to Max. Change from Baseline Mean SD Median Min. to Max Percent Change from Baseline Mean SD Median Min. to Max Percent Change from Baseline Mean SD Median SD Median SD Success |
|---|
|---|

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template
Table 14.2.4.4: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population) 

| | ARQ-1 | ARQ-151-202: Roflumilast Cream 0.3% | 0.3% |
|---|---|---|---|
| | | ARQ-151-201: | |
| | ARQ-151-201: | Vehicle Cream | |
| | AR Roflumilast Cream | and Cohort 2 | Total |
| Modified Psoriasis and Severity Index | (N=xx) | (N=xx) | (N=xx) |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX | XX | XX |
| SD | XX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX | XX | XX.X |
| SD | XX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX | XX | XX |
| SD | XX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| mPASI-75 | | | |
| Success | (%XX ) XX | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%XX ) XX | (%XX ) XX |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.4: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population) 

| | ARQ-151-201: | ARQ-151-201:<br>Vehicle Cream | |
|---|---|---|---|
| | Roflumilast Cream | and Cohort 2 | Total |
| Modified Psoriasis and Severity Index | (x=x) | (N=xx) | (N=XX) |
| Week 24 | | | |
| n | XX | XX | XX |
| Mean | XX | xx | XX |
| SD | XX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX | XX | XX |
| SD | XX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX | XX | XX |
| SD | XXX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| mPASI-75 | | | |
| Success | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.4: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population) 

| | ARO | ARQ-151-202: Roflumilast Cream 0.3% | 10.3% |
|---|---|---|---|
| | | ARQ-151-201: | |
| | ARQ-151-201: | Vehicle Cream | |
| | Roflumilast Cream | and Cohort 2 | Total |
| Modified Psoriasis and Severity Index | (N=xx) | (N=xx) | (N=xx) |
| Week 36 | | | |
| n | XX | XX | XX |
| Mean | XX | XX | XX |
| SD | XX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| Mean | XX | XX | XX |
| SD | XX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max | xx to xx | xx to xx | xx to xx |
| Percent Change from Baseline | | | |
| Mean | XX | XX | XX |
| SD | XX.X | XX.X | XX.X |
| Median | XX | XX | XX |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| mPASI-75 | | | |
| Success | (%XX () XX | (%xx ) xx | (%xx ) xx |
| Failure | (%xx ) xx | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.4.4: Summary of Modified Psoriasis and Severity Index (mPASI) (Safety Population) 

| | | ARQ-151-202: Roflumilast Cream 0.3%<br>ARQ-151-201: | n 0.3% |
|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream | Vehicle Cream and Cohort 2 | Total |
| Modified Psoriasis and Severity Index | (N=xx) | (N=xx) | (N=xx) |
| | XX | XX | XX |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX | XX | XX |
| | xx to xx | xx to xx | xx to xx |
| Mean | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX | XX | XX |
| | xx to xx | xx to xx | xx to xx |
| seline | | | |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX | XX | XX |
| | xx to xx | xx to xx | xx to xx |
| | (%xx ) xx | (%xx ) xx | (%xx) xx |
| | (%xx ) xx | (%xx ) xx | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. Note: No imputation of missing values. mPASI-75 is defined as a 75% reduction from baseline of mPASI. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.5.1: Summary of Duration of Treatment Free Interval and Investigator Global Assessment (IGA) Success (Safety Population: Cohort 1)

| | | | A | ARQ-151-202: Roflumilast Cream 0.3% | milast C | ream 0.3% | | | I |
|---|---|---|---|---|---|---|---|---|---|
| | AI<br>Roflum | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | AF<br>Roflumi | ARQ-151-201:<br>Roflumilast Cream 0.15%<br>(N=xx) | AF<br>Ve | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | | Total (N=xx) | |
| Number of Subjects who Achieved Disease<br>Clearance and Stopped Treatment | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx | |
| Treatment Free Interval (Weeks) n | | XX | | X | | XX | | XX | |
| Resumed Treatment<br>Censored | ) )<br>X X | (%xx<br>(%xx)<br>(xx) | ) XX XX | xx<br>xx%)<br>xx%) | ) XX X | (%XX<br>(%XX)<br>(%XX | XX XX | (%xx<br>(%xx) | |
| Number of Subjects With IGA Success | ) xx | (%XX | ) xx | (%XX | ) XX | (%xx | ) xx | (%xx | |
| Duration of IGA Success (Weeks) n Median <sup>a</sup> Disease Recurrence Censored | ) XX | xx xx (%) (%xx xx/%) | ) xx | xx<br>xx%)<br>xxx<br>xx,0%) | ) XX ( | xx<br>xx,<br>(%)<br>xx,<br>xx,<br>xx,<br>xx, | ) xx | xx<br>xx (%xx<br>xx x | |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Disease clearance is defined as Clear scores for IGA, I-IGA (if applicable) and mPASI (if applicable).

IGA success defined as achievement of an IGA of Clear or Almost Clear plus a 2-grade improvement in IGA. Duration of IGA success is defined as the time from first observation of IGA success to the first subsequent time a subject's disease response does not meet the criteria for IGA success. Subjects Treatment free interval is defined as time to re-starting study drug for subjects who achieved disease clearance and stopped treatment to all lesions. Subjects not re-starting study drug before ending participation in the study were censored at the day of the last observed disease assessment. with a continued success at end of participation in the study were censored at the day of the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Figure 14.2.5.1.1: Kaplan-Meier Plot of Treatment Free Interval (Weeks) (Safety Population: Cohort 1)



Note: Treatment free interval is defined as time to re-starting study drug for subjects who achieved Clear scores for IGA, I-IGA (if applicable) and mPASI (if applicable), and stopped treatment to all lesions. Subjects not re-starting study drug before ending participation in the study were censored at the day of the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Figure 14.2.5.1.2: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) Success (Weeks) (Safety Population: Cohort 1)



Note: IGA success defined as achievement of an IGA of Clear or Almost Clear plus a 2-grade improvement in IGA. Duration of IGA success is defined as the time from first observation of IGA success to the first subsequent time a subject's disease response does not meet the criteria for IGA success. Subjects with a continued success at end of participation in the study were censored at the day of the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.5.2: Summary of Duration of Treatment Free Interval and Investigator Global Assessment (IGA) Success (Safety Population: Cohort 2)

| 0.3% | | | | | |
|---|---|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | (%XX ) XX | xx<br>xx (%xx ) xx | | X | (%xx ) xx (%xx ) xx |
| | Number of Subjects who Achieved Disease<br>Clearance and Stopped Treatment | Treatment Free Interval (Weeks) n Median <sup>a</sup> Resumed Treatment | Censored Number of Subjects With IGA Success | Duration of IGA Success (Weeks) | Median* Disease Recurrence Censored |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Disease clearance is defined as Clear scores for IGA, I-IGA (if applicable) and mPASI (if applicable).

IGA success defined as achievement of an IGA of Clear or Almost Clear plus a 2-grade improvement in IGA. Duration of IGA success is defined as the time from first observation of IGA success to the first subsequent time a subject's disease response does not meet the criteria for IGA success. Subjects Treatment free interval is defined as time to re-starting study drug for subjects who achieved disease clearance and stopped treatment to all lesions. Subjects not re-starting study drug before ending participation in the study were censored at the day of the last observed disease assessment. with a continued success at end of participation in the study were censored at the day of the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Note: Treatment free interval is defined as time to re-starting study drug for subjects who achieved Clear scores for IGA, I-IGA (if applicable) and mPASI (if applicable), and stopped treatment to all lesions. Subjects not re-starting study drug before ending participation in the study were censored at the day of

the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template




Note: IGA success defined as achievement of an IGA of Clear or Almost Clear plus a 2-grade improvement in IGA. Duration of IGA success is defined as the time from first observation of IGA success to the first subsequent time a subject's disease response does not meet the criteria for IGA success. Subjects with a continued success at end of participation in the study were censored at the day of the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.5.3: Summary of Duration of Treatment Free Interval and Investigator Global Assessment (IGA) Success (Safety Population)

| | | ARQ. | .151-202:<br>AR | ARQ-151-202: Roflumilast Cream 0.3%<br>ARQ-151-201: | 0.3% | |
|---|---|---|---|---|---|---|
| | AR(<br>Roflur | ARQ-151-201:<br>Roflumilast Cream<br>(N=xx) | Vel<br>an | Vehicle Cream and Cohort 2 (N=xx) | | Total<br>(N=xx) |
| Number of Subjects who Achieved Disease<br>Clearance and Stopped Treatment | (%xx ) xx | (%XX | ) xx | (%xx) | ) xx | (%xx ) xx |
| Treatment Free Interval (Weeks) | | XX | | XX | | XX |
| Median <sup>a</sup><br>Resumed Treatment | ) XX | XX<br>(%XX) | XX | XX<br>(%XX | ) XX | XX<br>(%XX) |
| Censored | ) xx | (0/ <sub>0</sub> XX | XX ( | (%xx | XX | (0/ <sub>0</sub> XX |
| Number of Subjects With IGA Success | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx |
| Duration of IGA Success (Weeks) | | × | | × | | × |
| $\mathrm{Median}^{a}$ | | XX | | XX | | XX |
| Disease Recurrence | ) xx | (%xx | ) xx | (%XX | ) xx | (%XX |
| Censored | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Disease clearance is defined as Clear scores for IGA, I-IGA (if applicable) and mPASI (if applicable).

Treatment free interval is defined as time to re-starting study drug for subjects who achieved disease clearance and stopped treatment to all lesions. Subjects not re-starting study drug before ending participation in the study were censored at the day of the last observed disease assessment.

IGA success defined as achievement of an IGA of Clear or Almost Clear plus a 2-grade improvement in IGA. Duration of IGA success is defined as the time from first observation of IGA success to the first subsequent time a subject's disease response does not meet the criteria for IGA success. Subjects with a continued success at end of participation in the study were censored at the day of the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Note: Treatment free interval is defined as time to re-starting study drug for subjects who achieved Clear scores for IGA, I-IGA (if applicable) and mPASI (if applicable), and stopped treatment to all lesions. Subjects not re-starting study drug before ending participation in the study were censored at the day of the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Figure 14.2.5.3.2: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) Success (Weeks) (Safety Population)



Note: IGA success defined as achievement of an IGA of Clear or Almost Clear plus a 2-grade improvement in IGA. Duration of IGA success is defined as the time from first observation of IGA success to the first subsequent time a subject's disease response does not meet the criteria for IGA success. Subjects with a continued success at end of participation in the study were censored at the day of the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.6.1: Summary of Disease Recurrence (Safety Population: Cohort 1)

| | Roflum | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | AI<br>ARG<br>Roflumila | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Cream (N=xx) | nilast Cr<br>AR<br>Vel | Cream 0.3% ARQ-151-201: Vehicle Cream (N=xx) | | Total<br>(N=xx) |
|---|---|---|---|---|---|---|---|---|
| Total Number of Instances of Disease<br>Recurrence Following Clearance | | | | | | | | |
| n | XX | | xx | | XX | | xx | |
| 0 | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx |
| _ | ) xx | (%XX | ) xx | (%XX | ) xx | (%XX | ) xx | (%xx |
| 2 | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx |
| 8 | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx |
| ++ | XX ( | (%xx | ) xx | (%xx | XX | (%xx | XX ( | (%xx |
| Number of Instances of Disease Recurrence<br>Following Clearance Through Week 24a | | | | | | | | |
| n | XX | | XX | | XX | | XX | |
| П | \<br>\<br>\<br>\<br>\ | (%) | )<br>X X | (%)^^^ | \<br>\<br>\<br>\ | (%)^^ | ) | (%)^^ |
| o | \ | (70 XX<br>(70 XX | v ; | xx (0) | \<br>\<br>\<br>\ | (70 XX | v ; | (70/0% |
| <b>-</b> ( | XX<br>XX | XX.70) | ) xx | XX70) | y<br>XX | (0/XX<br>(0/) | yx<br>XX | (0/XX) |
| 2 | )<br>XX | (%XX | ) xx | (0/XX | ) XX | (%XX | ) xx | (%XX |
| 33 | ) xx | (%XX | ) xx | (%XX | )<br>X | (%xx | ) xx | (%xx |
| 4+ | ) xx | (%XX | ) xx | (%XX | ) XX | (%xx | ) xx | (%xx |
| Number of Instances of Disease Recurrence<br>Following Clearance Through Week 52a | | | | | | | | |
| n | XX | | XX | | XX | | XX | |
| 0 | ) XX | (%xx | ) xx | (0%XX | ) xx | (%xx | ) xx | (%XX |
| - | XX ( | (%XX | ) XX | (%xx | XX | (%xx | XX ( | (%xx |
| 2 | xx ( | (%xx | ) xx | (%xx | ) xx | (%xx | ) xx | (%xx |
| 3 | ) xx | (%XX | ) xx | (%xx | ) xx | (%XX | ) xx | (%xx |
| ++ | ) xx | (%XX | ) xx | (0%XX | ) xx | (%xx | ) xx | (%XX |

<sup>&</sup>lt;sup>a</sup> Percentages calculated out of total number of subjects who participated in study through the respective visit. Note: Disease clearance defined as an IGA of Clear and mPASI of 0. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.6.2: Summary of Disease Recurrence (Safety Population: Cohort 2)

| ARQ-151-201:<br>Roflumilast Cream 0.3% $(N=xx)$ | | XX | (%XX ) XX | (%xx ) xx | (%XX ) XX | (%XX ) XX | (%xx ) xx | | XX | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ( xx%) | (%xx ) xx | | XX | (%xx ) xx | (%xx ) xx | (%XX ) XX | (%xx ( xx%) | (%xx ) xx |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Total Number of Instances of Disease<br>Recurrence Following Clearance | n | 0 | 1 | 2 | 3 | ++ | Number of Instances of Disease Recurrence<br>Following Clearance Through Week 24a | n | 0 | 1 | 2 | 3 | ++ | Number of Instances of Disease Recurrence<br>Following Clearance Through Week 52a | n | 0 | 1 | 2 | 3 | 4+ |

<sup>&</sup>lt;sup>a</sup> Percentages calculated out of total number of subjects who participated in study through the respective visit. Note: Disease clearance defined as an IGA of Clear and mPASI of 0. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.6.3: Summary of Disease Recurrence (Safety Population)

| | | ARO | ARO-151-202: Roflumilast Cream 0.3% | t Cream 0.3% | |
|---|---|---|---|---|---|
| | ARQ<br>Roflun | ARQ-151-201:<br>Roflumilast Cream | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2 | | Total |
| | D | (X=XX) | (N=xx) | | (N=xx) |
| Total Number of Instances of Disease<br>Recurrence Following Clearance | | | | | |
| n | XX | | XX | XX | |
| 0 | ( ) xx | (%XX | (%xx) xx | ) xx | (%XX |
| | ) xx | (%xx | (%xx ) xx | ) xx | (%XX |
| 2 | ( ) xx | (%xx | (%xx) xx | ) xx | (%XX |
| | ( ) xx | (%xx | (%xx) xx | ) xx | (%XX |
| 4+ | ) xx | (%xx | (%XX ) XX | ) xx | (%XX |
| Number of Instances of Disease Recurrence<br>Following Clearance Through Week 24 <sup>a</sup> | | | | | |
| )<br>u | XX | | XX | XX | |
| 0 | ) xx | (%xx | (%xx) xx | ) xx | (%XX |
| | $\overline{}$ | (%XX | (%xx ) xx | ) xx | (%XX |
| 2 | ) xx | (%XX | (0/xx) $(xx)$ | ) xx | (%XX |
| | xx ( | (%XX | (%xx ) xx | ) xx | (%XX |
| 4+ | ) xx | (%xx | (%xx ) xx | ) xx | (%XX |
| Number of Instances of Disease Recurrence<br>Following Clearance Through Week 24 <sup>a</sup> | | | | | |
| n | XX | | XX | XX | |
| 0 | ) xx | (%XX | (%xx ) xx | ) xx | (%XX |
| | xx ( | (%XX | (%xx ) xx | ) xx | (%XX |
| 2 | xx ( | (%XX | (%xx ) xx | ) xx | (%XX |
| 33 | ) xx | (%XX | (%xx ) xx | ) xx | (%XX |
| 4+ | ) xx | (%XX | (%xx ) xx | ) xx | (%XX |

<sup>&</sup>lt;sup>a</sup> Percentages calculated out of total number of subjects who participated in study through the respective visit. Note: Disease clearance defined as an IGA of Clear and mPASI of 0. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.7.1: Summary of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Safety Population: Cohort 1)

| Duration of IGA of Clear or Almost Clear (Weeks) | 201:<br>cam 0.3% ] | ARQ-151-201: ARQ-151-201 Roflumilast Cream 0.15% Vehicle Cream (N=xx) (N=xx) (N=xx) | ARQ-151-201: Vehicle Cream (N=xx) xx | Total (N=xx) xx |
|---|---|---|---|---|
| | xx (%xx ) xx | xx (%xx ) xx x x x x x x x x x x x x x x x x | XX (%XX ) XX (%0,0) Ax | (%XX ) XX |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Duration of IGA of Clear or Almost Clear is defined as the time from the first observation of IGA Clear or Almost Clear to the first subsequent time a subject's IGA is not Clear or Almost Clear. The duration of IGA Clear or Almost Clear for subjects who end treatment with IGA Clear or Almost Clear will be censored at the last IGA date.

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Figure 14.2.7.1: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Weeks) (Safety Population: Cohort 1)



subject's IGA is not Clear or Almost Clear. The duration of IGA Clear or Almost Clear for subjects who end treatment with IGA Clear or Almost Clear Note: Duration of IGA of Clear or Almost Clear is defined as the time from the first observation of IGA Clear or Almost Clear to the first subsequent time a

will be censored at the last IGA date.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.7.2: Summary of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Safety Population: Cohort 2)

| Roflumilast Cream 0.3% (N=xx) | | XX | XX | (%XX ) XX | (%xx ) xx |
|---|---|---|---|---|---|
| | Duration of IGA of Clear or Almost Clear (Weeks) | n | $Median^a$ | Disease Recurrence | Censored |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Duration of IGA of Clear or Almost Clear is defined as the time from the first observation of IGA Clear or Almost Clear to the first subsequent time a subject's IGA is not Clear or Almost Clear. The duration of IGA Clear or Almost Clear for subjects who end treatment with IGA Clear or Almost Clear.

will be censored at the last IGA date.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Figure 14.2.7.2: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Weeks) (Safety Population: Cohort 2)



Note: Duration of IGA of Clear or Almost Clear is defined as the time from the first observation of IGA Clear or Almost Clear to the first subsequent time a subject's IGA is not Clear or Almost Clear or Almost Clear or Almost Clear for subject's IGA is not Clear or Almost Clear or Almo will be censored at the last IGA date.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.7.3: Summary of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Safety Population)

| ilast Cream 0.3% | | $\begin{array}{ccc} 1 & 1 & 1 & 1 \\ 1 & 1 & 1 & 1 \\ 1 & 1 &$ | | | XX | XX | (%xx ) xx | (%xx ) xx |
|---|---|---|---|---|---|---|---|---|
| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201:<br>Vehicle Cream | m and conort 2 $(N=xx)$ | | | XX | XX | (%xx ) xx | (%xx ) xx |
| | ARQ-151-201: | Konumhast Creat (N=xx) | | | XX | XX | (%xx ) xx | (%xx ) xx |
| | | | Duration of IGA of Clear or Almost Clear | (Weeks) | n | $Median^a$ | Disease Recurrence | Censored |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

will be censored at the last IGA date.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

subject's IGA is not Clear or Almost Clear. The duration of IGA Clear or Almost Clear for subjects who end treatment with IGA Clear or Almost Clear Note: Duration of IGA of Clear or Almost Clear is defined as the time from the first observation of IGA Clear or Almost Clear to the first subsequent time a

Figure 14.2.7.3: Kaplan-Meier Plot of Duration of Investigator Global Assessment (IGA) of Clear or Almost Clear (Weeks) (Safety Population)



subject's IGA is not Clear or Almost Clear. The duration of IGA Clear or Almost Clear for subjects who end treatment with IGA Clear or Almost Clear Note: Duration of IGA of Clear or Almost Clear is defined as the time from the first observation of IGA Clear or Almost Clear to the first subsequent time a will be censored at the last IGA date.
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.8.1.1: Primary Summary of Duration of PASI-50 (Safety Population: Cohort 1)

| | | ARQ-151-202: Roflumilast Cream 0.3% | milast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| | (x = N) | (N=xx) | (X=X) | (X=X) |
| Duration of PASI-50 (Weeks) | | | | |
| n | XX | XX | XX | XX |
| $Median^a$ | XX | XX | XX | XX |
| Disease Recurrence | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Censored | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%XX ) XX |

Median determined using the Kaplan-Meier method.

Note: Duration of PASI-50 is defined as the time from the first observation of a 50% reduction from baseline in the Psoriasis Area and Severity Index (PASI) to the first subsequent time a subjects's PASI score is greater than a 50% reduction from baseline. The duration of PASI-50 for subjects who end treatment with PASI score at least 50% less than baseline will be censored at the last disease assessment date.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Figure 14.2.8.1.1: Primary Kaplan-Meier Plot of Duration of PASI-50 (Safety Population: Cohort 1)



to the first subsequent time a subjects's PASI score is greater than a 50% reduction from baseline. The duration of PASI-50 for subjects who end treatment Note: Duration of PASI-50 is defined as the time from the first observation of a 50% reduction from baseline in the Psoriasis Area and Severity Index (PASI) with PASI score at least 50% less than baseline will be censored at the last disease assessment date.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.8.1.2: Sensitivity Summary of Duration of PASI-50 (Safety Population: Cohort 1)

| | | ARQ-151-202: Roflumilast Cream 0.3% | milast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | F |
| | Kollumliast Cream 0.3% $(N=xx)$ | Kollumlast Cream 0.13% (N=xx) | (N=xx) | 10001 $(N=xx)$ |
| Duration of PASI-50 (Weeks) | | | | |
| n | XX | XX | XX | XX |
| $Median^a$ | XX | XX | XX | XX |
| Disease Recurrence | (0%XX ) XX | (%xx ) xx | (%xx ) xx | (%XX ) XX |
| Censored | (%xx ) xx | (%xx ) xx | (0/xx) $(xx)$ | (%xx ) xx |

Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Duration of PASI-50 is defined as the time from the first observation of a 50% reduction from baseline in the Psoriasis Area and Severity Index (PASI) to the first subsequent time a subjects's PASI score is greater than a 50% reduction from baseline. The duration of PASI-50 for subjects who end treatment with PASI score at least 50% less than baseline will be censored at the last disease assessment date.



to the first subsequent time a subjects's PASI score is greater than a 50% reduction from baseline. The duration of PASI-50 for subjects who end treatment Note: Duration of PASI-50 is defined as the time from the first observation of a 50% reduction from baseline in the Psoriasis Area and Severity Index (PASI) with PASI score at least 50% less than baseline will be censored at the last disease assessment date. Baseline is defined as the last observation prior to entrance into the ARQ-151-202 study.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)


Table 14.2.8.2: Summary of Duration of PASI-50 (Safety Population: Cohort 2)

| Roflumilast Cream $0.3\%$ $(N=xx)$ | | XX | XX | xx ( xx%) | xx ( xx%) |
|---|---|---|---|---|---|
| | Duration of PASI-50 (Weeks) | n | $Median^a$ | Disease Recurrence | Censored |

to the first subsequent time a subjects's PASI score is greater than a 50% reduction from baseline. The duration of PASI-50 for subjects who end treatment <sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Duration of PASI-50 is defined as the time from the first observation of a 50% reduction from baseline in the Psoriasis Area and Severity Index (PASI) with PASI score at least 50% less than baseline will be censored at the last disease assessment date. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



to the first subsequent time a subjects's PASI score is greater than a 50% reduction from baseline. The duration of PASI-50 for subjects who end treatment Note: Duration of PASI-50 is defined as the time from the first observation of a 50% reduction from baseline in the Psoriasis Area and Severity Index (PASI) with PASI score at least 50% less than baseline will be censored at the last disease assessment date. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.8.3: Summary of Duration of PASI-50 (Safety Population)

| 0.3% | Total<br>(N=xx) | (%xx ) xx<br>(%xx ) xx<br>xx x x |
|---|---|---|
| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2<br>(N=xx) | xx (%xx ) xx (xx) xx (xx) xx (xx) xx |
| ARO | ARQ-151-201:<br>Roflumilast Cream<br>(N=xx) | (%xx ) xx<br>(%xx ) xx |
| | | Duration of PASI-50 (Weeks) n Median <sup>a</sup> Disease Recurrence Censored |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

to the first subsequent time a subjects's PASI score is greater than a 50% reduction from baseline. The duration of PASI-50 for subjects who end treatment Note: Duration of PASI-50 is defined as the time from the first observation of a 50% reduction from baseline in the Psoriasis Area and Severity Index (PASI) with PASI score at least 50% less than baseline will be censored at the last disease assessment date.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Figure 14.2.8.3: Kaplan-Meier Plot of Duration of PASI-50 (Safety Population)



to the first subsequent time a subjects's PASI score is greater than a 50% reduction from baseline. The duration of PASI-50 for subjects who end treatment Note: Duration of PASI-50 is defined as the time from the first observation of a 50% reduction from baseline in the Psoriasis Area and Severity Index (PASI) with PASI score at least 50% less than baseline will be censored at the last disease assessment date.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.9.1: Summary of Duration of PASI-75 (Safety Population: Cohort 1)

| | | ARQ-151-202: Roflumilast Cream 0.3% | milast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| | (N=XX) | (X=N) | (N=XX) | (XX=N) |
| Duration of PASI-75 (Weeks) | | | | |
| n | XX | XX | xx | XX |
| Median <sup>a</sup> | XX | XX | XX | XX |
| Disease Recurrence | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Censored | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |

to the first subsequent time a subjects's PASI score is greater than a 75% reduction from baseline. The duration of PASI-75 for subjects who end treatment with PASI score at least 75% less than baseline will be censored at the last disease assessment date.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME) <sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Duration of PASI-75 is defined as the time from the first observation of a 75% reduction from baseline in the Psoriasis Area and Severity Index (PASI)

Figure 14.2.9.1: Kaplan-Meier Plot of Duration of PASI-75 (Safety Population: Cohort 1)



to the first subsequent time a subjects's PASI score is greater than a 75% reduction from baseline. The duration of PASI-75 for subjects who end treatment Note: Duration of PASI-75 is defined as the time from the first observation of a 75% reduction from baseline in the Psoriasis Area and Severity Index (PASI) with PASI score at least 75% less than baseline will be censored at the last disease assessment date. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.9.2: Summary of Duration of PASI-75 (Safety Population: Cohort 2)

| 10.3% | | | | | |
|---|---|---|---|---|---|
| Roflumilast Cream $0.3\%$ | | XX | XX | ( <sub>0</sub> / <sub>0</sub> xx ) xx | (%xx ) xx |
| | Duration of PASI-75 (Weeks) | n | $Median^a$ | Disease Recurrence | Censored |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Duration of PASI-75 is defined as the time from the first observation of a 75% reduction from baseline in the Psoriasis Area and Severity Index (PASI) to the first subsequent time a subjects's PASI score is greater than a 75% reduction from baseline. The duration of PASI-75 for subjects who end treatment with PASI score at least 75% less than baseline will be censored at the last disease assessment date.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Note: Duration of PASI-75 is defined as the time from the first observation of a 75% reduction from baseline in the Psoriasis Area and Severity Index (PASI) to the first subsequent time a subjects's PASI score is greater than a 75% reduction from baseline. The duration of PASI-75 for subjects who end treatment with PASI score at least 75% less than baseline will be censored at the last disease assessment date. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.9.3: Summary of Duration of PASI-75 (Safety Population)

| ARQ-151-202: Roflumilast Cream 0.3%<br>ARQ-151-201: | ARQ-151-201: Vehicle Cream Roflumilast Cream and Cohort 2 Total (N=xx) (N=xx) | | XX XX XX | XX XX XX | (%xx) xx $(%xx)$ xx $(%xx)$ xx $(%xx)$ | (%xx) xx $(%xx)$ xx $(%xx)$ xx $(%xx)$ |
|---|---|---|---|---|---|---|
| | ARQ-1<br>Roflumil<br>(N= | Duration of PASI-75 (Weeks) | n | $Median^a$ | Disease Recurrence xx (xx) | Censored xx ( xx |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

to the first subsequent time a subjects's PASI score is greater than a 75% reduction from baseline. The duration of PASI-75 for subjects who end treatment Note: Duration of PASI-75 is defined as the time from the first observation of a 75% reduction from baseline in the Psoriasis Area and Severity Index (PASI) with PASI score at least 75% less than baseline will be censored at the last disease assessment date.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Figure 14.2.9.3: Kaplan-Meier Plot of Duration of PASI-75 (Safety Population)



Note: Duration of PASI-75 is defined as the time from the first observation of a 75% reduction from baseline in the Psoriasis Area and Severity Index (PASI) to the first subsequent time a subjects's PASI score is greater than a 75% reduction from baseline. The duration of PASI-75 for subjects who end treatment with PASI score at least 75% less than baseline will be censored at the last disease assessment date.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.10.1: Summary of Time to Disease Recurrence (Safety Population: Cohort 1)

| | | ARQ-151-202: Roflumilast Cream 0.3% | milast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | |
| | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Total |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Time to Disease Recurrence (Weeks) | | | | |
| n | XX | XX | XX | XX |
| Median <sup>a</sup> | XX | XX | XX | XX |
| Disease Recurrence | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Censored | (%xx ) xx | (%xx ) xx | (%XX ) XX | (%xx ) xx |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

first observation of an IGA score of 2 or greater. The time to disease recurrence among subjects with clearance at the end of the study observation period will be censored at the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME) Note: Restricted to subjects who stop therapy due to disease clearance. Time to disease recurrence is defined as the time from the last dose of ARQ-151 to the

Figure 14.2.10.1: Kaplan-Meier Plot of Time to Disease Recurrence (Safety Population: Cohort 1)



first observation of an IGA score of 2 or greater. The time to disease recurrence among subjects with clearance at the end of the study observation period Note: Restricted to subjects who stop therapy due to disease clearance. Time to disease recurrence is defined as the time from the last dose of ARQ-151 to the will be censored at the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.10.2: Summary of Time to Disease Recurrence (Safety Population: Cohort 2)

| Roflumilast Cream 0.3% (N=xx) | | XX | XX | (%XX ) XX | (%XX ) XX |
|---|---|---|---|---|---|
| | Duration of PASI-75 (Weeks) | n | $Median^a$ | Disease Recurrence | Censored |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

Note: Restricted to subjects who stop therapy due to disease clearance. Time to disease recurrence is defined as the time from the last dose of ARQ-151 to the first observation of an IGA score of 2 or greater. The time to disease recurrence among subjects with clearance at the end of the study observation period will be censored at the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



Note: Restricted to subjects who stop therapy due to disease clearance. Time to disease recurrence is defined as the time from the last dose of ARQ-151 to the first observation of an IGA score of 2 or greater. The time to disease recurrence among subjects with clearance at the end of the study observation period will be censored at the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.2.10.3: Summary of Time to Disease Recurrence (Safety Population)

| am 0.3% | | | Total | (N=xx) | | XX | XX | (%xx ) xx | ( <sub>0</sub> / <sub>0</sub> XX ) XX |
|---|---|---|---|---|---|---|---|---|---|
| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201: | Vehicle Cream | and Cohort 2 | (N=xx) | | XX | XX | (%xx ) xx | (%xx ) xx |
| AR | | ARQ-151-201: | Roflumilast Cream | (N=xx) | | XX | XX | (%xx ) xx | (%XX ) XX |
| | | | | | Duration of PASI-75 (Weeks) | n | Median <sup>a</sup> | Disease Recurrence | Censored |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

first observation of an IGA score of 2 or greater. The time to disease recurrence among subjects with clearance at the end of the study observation period Note: Restricted to subjects who stop therapy due to disease clearance. Time to disease recurrence is defined as the time from the last dose of ARQ-151 to the

will be censored at the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



first observation of an IGA score of 2 or greater. The time to disease recurrence among subjects with clearance at the end of the study observation period Note: Restricted to subjects who stop therapy due to disease clearance. Time to disease recurrence is defined as the time from the last dose of ARQ-151 to the will be censored at the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.11.1: Summary of Disease Control (Safety Population: Cohort 1)

| | | ARQ-151-202: Koflumilast Cream 0.3% | ımılast Cream 0.5% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roffinnilast Cream 0.3% | ARQ-151-201: Roffinmilast Cream 0 15% | ARQ-151-201: Vehicle Gream | Total |
| | (N=XX) | (N=xx) | (N=xx) | (N=xx) |
| ime to Disease Control (Weeks) | | | | |
| и | XX | XX | XX | XX |
| Median <sup>a</sup> | XX | XX | XX | XX |
| Disease Control | (%xx ) xx | (%xx ) xx | (%xx ) xx | (%xx ) xx |
| Censored | (%xx ) xx | (%xx ) xx | (%XX ) XX | (%XX ) XX |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

therapy to the first reported IGA score of Clear or Almost Clear. The time to disease control among subjects who do not achieve an IGA score of Clear or Almost Clear by the end of the study observation period will be censored at the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME) Note: Restricted to subjects who restart therapy after having stopped therapy due to disease clearance. Time to disease control is the time from the restart of

Figure 14.2.11.1: Kaplan-Meier Plot of Time to Disease Control (Safety Population: Cohort 1)



therapy to the first reported IGA score of 0 or 1. The time to disease control among subjects who do not achieve an IGA score of 0 or 1 by the end of the Note: Restricted to subjects who restart therapy after having stopped therapy due to disease clearance. Time to disease control is the time from the restart of study observation period will be censored at the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.2.11.2: Summary of Disease Control (Safety Population: Cohort 2)

| Roflumilast Cream 0.3% (N=xx) | | XX | XX | (%XX ) XX | xx ( xx%) |
|---|---|---|---|---|---|
| | Time to Disease Control (Weeks) | n | Median <sup>a</sup> | Disease Control | Censored |


Median determined using the Kaplan-Meier method.

Note: Restricted to subjects who restart therapy after having stopped therapy due to disease clearance. Time to disease control is the time from the restart of therapy to the first reported IGA score of 0 or 1. The time to disease control among subjects who do not achieve an IGA score of 0 or 1 by the end of the study observation period will be censored at the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)



therapy to the first reported IGA score of 0 or 1. The time to disease control among subjects who do not achieve an IGA score of 0 or 1 by the end of the Note: Restricted to subjects who restart therapy after having stopped therapy due to disease clearance. Time to disease control is the time from the restart of study observation period will be censored at the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.2.11.3: Summary of Disease Control (Safety Population)

| | Total (N=xx) | | XX | XX | (%XX | (%XX |
|---|---|---|---|---|---|---|
| ARQ-151-202: Roflumilast Cream 0.3%<br>ARQ-151-201:<br>Vehicle Cream | and Cohort 2 (N=xx) | | XX | XX | ) xx (%xx ) xx | ) xx (%xx ) xx |
| ARO-151-201: | Roflumilast Cream (N=xx) | | XX | XX | (%xx ) xx | (%xx ) xx |
| | | Time to Disease Control (Weeks) | n | $Median^a$ | Disease Control | Censored |

<sup>&</sup>lt;sup>a</sup> Median determined using the Kaplan-Meier method.

therapy to the first reported IGA score of 0 or 1. The time to disease control among subjects who do not achieve an IGA score of 0 or 1 by the end of the Note: Restricted to subjects who restart therapy after having stopped therapy due to disease clearance. Time to disease control is the time from the restart of study observation period will be censored at the last observed disease assessment. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)



therapy to the first reported IGA score of 0 or 1. The time to disease control among subjects who do not achieve an IGA score of 0 or 1 by the end of the Note: Restricted to subjects who restart therapy after having stopped therapy due to disease clearance. Time to disease control is the time from the restart of study observation period will be censored at the last observed disease assessment.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.3.0.1.1: Summary of Extent of Exposure (Safety Population: Cohort 1)

<sup>&</sup>lt;sup>a</sup> A subject was considered compliant with the dosing regimen if the subject did not miss more than 3 consecutive days dosing and applied >= 80% of expected

doses while participating in the study.

Note: Lost to Follow-Up subjects were included using all available information. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.0.1.2: Summary of Extent of Exposure (Safety Population: Cohort 2)

| Roflumilast Cream $0.3\%$ (N=xx) | | XX | XX.X | XX.XX | XX.X | xx to xx | | XX | XX.X | XX.XX | XX.X | xx to xx | (%XX ) XX | xx ( xx%) xx | (%XX ) XX | xx ( xx%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Number of Applications | Z | Mean | SD | Median | Min. to Max. | Amount of Drug Used (g) | )<br>Z | Mean | SD | Median | Min. to Max. | Completed $>= 80\%$ of Expected Doses | Completed < 80% of Expected Doses | Compliant <sup>a</sup> | Not Compliant |

<sup>&</sup>lt;sup>a</sup> A subject was considered compliant with the dosing regimen if the subject did not miss more than 3 consecutive days dosing and applied >= 80% of expected doses while participating in the study.

Note: Lost to Follow-Up subjects were included using all available information.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.0.1.3: Summary of Extent of Exposure (Safety Population)

| • | ARQ-1 | ARQ-151-202: Roflumilast Cream 0.3% | 0.3% |
|---|---|---|---|
| | | ARQ-151-201: | |
| | ARQ-151-201:<br>Roflumilast Cream | Vehicle Cream | Total |
| | (N=xx) | | (N=xx) |
| Number of Applications | | | |
| N | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Amount of Drug Used (g) | | | |
| | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Completed >= 80% of Expected Doses | ( )XX ( )XX | (%xx ) xx | (%XX ) XX |
| Completed < 80% of Expected Doses | (%XX ) XX | (%XX ) XX | (%xx ) xx |
| Compliant <sup>a</sup> | (%XX) XX | (%XX ) XX | (%XX ) XX |
| Not Compliant | (%XX ) XX | (%xx ) xx | (%XX ) XX |

<sup>&</sup>lt;sup>a</sup> A subject was considered compliant with the dosing regimen if the subject did not miss more than 3 consecutive days dosing and applied >= 80% of expected

doses while participating in the study.

Note: Lost to Follow-Up subjects were included using all available information. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.1: Summary of Local Tolerability (Safety Population: Cohort 1) 

| | A<br>Roflur | ARQ-151-201: ARQ-151-201: Roflumilast Cream 0.3% Roflumilast Cream 0.15% | ARQ-151-201<br>Roflumilast Cream ( | Q-151-201: ARQ-151-201: st Cream 0.15% Vehicle Cream | ARQ-<br>Vehic | ARQ-151-201:<br>Vehicle Cream | | Total |
|---|---|---|---|---|---|---|---|---|
| Investigator Local Tolerability Dermal Response | | (N=XX) | =\( \) | (N=xx) | | (N=xx) | | (N=xx) |
| Baseline | | | | | | | | |
| n | XX | | XX | | XX | | XX | |
| 0 - no evidence of irritation | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | (%X.XX | ) xx | xx.x% |
| 1 - minimal erythema, barely perceptible | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | xx.x%) | ) xx | xx.x% |
| 2 - definite erythema, readily visible; minimal | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | xx.xx%) | ) xx | xx.x% |
| edema or minimal popular response | | | | | | | | |
| 3 - erythema and papules | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | (%X.XX | ) xx | xx.x% |
| 4 - definite edema | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | xx.x%) | ) xx | xx.x% |
| 5 - erythema, edema and papules | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | (%X.XX | ) xx | xx.x% |
| 6 - vesicular eruption | ) xx | (%X.XX | xx ( xx.x%) | (%) | XX (XX. | XX.X%) | ) xx | xx.x% |
| 7 - strong reaction spreading beyond application | XX ( | (%x.xx | xx ( xx.x%) | (%) | xx ( xx. | (%x.xx | ) xx | (%x.xx |
| site | | | | | | | | |
| Week 4 | | | | | | | | |
| n | XX | | XX | | XX | | XX | |
| 0 - no evidence of irritation | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | (%X.XX | ) xx | xx.x% |
| 1 - minimal erythema, barely perceptible | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | xx.x%) | ) xx | xx.x% |
| 2 - definite erythema, readily visible; minimal | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | (%X.XX | ) xx | xx.x% |
| edema or minimal popular response | | | | | | | | |
| 3 - erythema and papules | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | (%X.XX | ) xx | xx.x% |
| 4 - definite edema | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | xx.x%) | ) xx | xx.x% |
| 5 - erythema, edema and papules | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | xx.x%) | ) xx | xx.x% |
| 6 - vesicular eruption | ) xx | (%X.XX | xx ( xx.x%) | (%) | xx ( xx. | xx.x%) | ) xx | xx.x% |
| 7 - strong reaction spreading beyond application | ) XX | (%X.XX | xx ( xx.x%) | (%) | xx (xx. | XX.X%) | ) XX | xx.x% |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.1.1.1: Summary of Local Tolerability (Safety Population: Cohort 1) 

| | | ARO-151-202: Ro | ARO-151-202: Roflumilast Cream 0.3% | | |
|---|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3 | ARQ-151-201: ARQ-151-201: Roflumilast Cream 0.3% Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | | Total |
| Investigator Local Tolerability Dermal Response | (N=xx) | (N=XX) | (N=xx) | | (N=xx) |
| Week 12 | | | | | |
| n | XX | XX | XX | XX | |
| 0 - no evidence of irritation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| 1 - minimal erythema, barely perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| 2 - definite erythema, readily visible; minimal | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x) | ) xx | xx.x%) |
| edema or minimal popular response | | | | | |
| 3 - erythema and papules | xx (xx.x) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| 4 - definite edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| 5 - erythema, edema and papules | xx (xx.x) | xx ( xx.x%) | (%X.XX ) XX | ) xx | xx.x%) |
| 6 - vesicular eruption | xx (xx.x) | xx ( xx.x%) | (%X.XX ) XX | ) xx | xx.x%) |
| 7 - strong reaction spreading beyond application | (%X.XX ) XX | xx ( xx.x%) | (xx.x) xx.x% | ) xx | xx.x%) |
| site | | | | | |
| Week 24 | | | | | |
| n | XX | XX | XX | XX | |
| 0 - no evidence of irritation | xx (xx.x) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| 1 - minimal erythema, barely perceptible | xx (xx.x) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x% |
| 2 - definite erythema, readily visible; minimal | xx (xx.x) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| edema or minimal popular response | | | | | |
| 3 - erythema and papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| 4 - definite edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| 5 - erythema, edema and papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x%) |
| 6 - vesicular eruption | xx (xx.x) | xx ( xx.x%) | xx ( xx.x%) | ) xx | XX.X%) |
| 7 - strong reaction spreading beyond application | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | ) xx | XX.X%) |
| site | | | | | |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.1.1.1: Summary of Local Tolerability (Safety Population: Cohort 1) 

| | | | ARO-151-202: Roflumilast Cream 0.3% | flumilas | t Cream 0.3% | | |
|---|---|---|---|---|---|---|---|
| | ARQ-151-201: ARQ-151-201: Roflumilast Cream 0.13% Roflumilast Cream 0.15% | A<br>3% Roflumi | ARQ-151-201:<br>milast Cream 0.15% | AF<br>Ve | ARQ-151-201:<br>Vehicle Cream | | Total |
| Investigator Local Tolerability Dermal Response | (N=xx) | | (N=xx) | | (N=xx) | | (N=xx) |
| Week 36 | | | | | | | |
| n | XX | XX | | XX | | XX | |
| 0 - no evidence of irritation | $xx (xx.x^{0})$ | ) xx | XX.X%) | ) xx | XX.X%) | ) xx | xx.x%) |
| 1 - minimal erythema, barely perceptible | $xx (xx.x^{0})$ | ) xx | XX.X%) | ) xx | XX.X%) | ) xx | xx.x%) |
| 2 - definite erythema, readily visible; minimal | $xx (xx.x^{0})$ | ) xx | xx.x%) | ) xx | (%X.XX | ) xx | xx.x%) |
| edema or minimal popular response | | | | | | | |
| 3 - erythema and papules | (xx.x) xx.x | ) xx | XX.X%) | ) xx | xx.x%) | ) xx | xx.x%) |
| 4 - definite edema | $xx (xx.x^{0})$ | ) xx | XX.X%) | ) xx | xx.x%) | ) xx | xx.x%) |
| 5 - erythema, edema and papules | xx (xx.x) xx | ) xx | xx.x%) | ) xx | (%X.XX | ) xx | xx.x%) |
| 6 - vesicular eruption | xx ( xx.x%) | ) xx | XX.X%) | ) xx | XX.X%) | ) XX | xx.x%) |
| 7 - strong reaction spreading beyond application | (xx.x) xx $(xx.x)$ | ) xx | (%X.XX | ) xx | (%x.xx | xx ( | (%X.XX |
| site | | | | | | | |
| Week 52 | | | | | | | |
| n | XX | XX | | XX | | XX | |
| 0 - no evidence of irritation | $xx (xx.x^{0})$ | ) xx | XX.X%) | ) xx | XX.X%) | ) xx | xx.x%) |
| 1 - minimal erythema, barely perceptible | xx (xx.x) xx | ) xx | xx.x%) | ) xx | xx.x%) | ) xx | xx.x%) |
| 2 - definite erythema, readily visible; minimal | $xx (xx.x^{0})$ | ) xx | xx.x% | ) xx | xx.x%) | ) xx | xx.x%) |
| edema or minimal popular response | | | | | | | |
| 3 - erythema and papules | $xx (xx.x^{0})$ | ) xx | XX.X% | ) xx | (%X.XX | ) xx | xx.x%) |
| 4 - definite edema | $xx (xx.x^{0})$ | ) xx | xx.x% | ) xx | xx.xx%) | ) xx | xx.x%) |
| 5 - erythema, edema and papules | xx (xx.x) xx | ) xx | xx.x% | ) xx | xx.x%) | ) xx | xx.x%) |
| 6 - vesicular eruption | xx (xx.x) xx | ) xx | XX.X%) | ) xx | xx.x%) | ) xx | XX.X%) |
| 7 - strong reaction spreading beyond application | xx ( xx.x%) | ) xx | xx.x%) | ) xx | (%x.xx | ) xx | (%X.XX |
| site | | | | | | | |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.1.1.2: Summary of Local Tolerability (Safety Population: Cohort 2) 

| Baseline In oe vidence of irritation - strong reaction spreadible beyond application - no evidence of irritation - the finite edema - the finite each and papules - the finite each |
|---|
|---|

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.3.1.1.2: Summary of Local Tolerability (Safety Population: Cohort 2) 

| Investigator Local Tolerability Dermal Response | Roflumilast Cream 0.3% (N=xx) |
|---|---|
| Week 12 | |
| n<br>n = na avidance af imitation | XX |
| 1 - minimal erythema, barely perceptible | _ ر |
| 2 - definite erythema, readily visible; minimal | |
| 3 - erythema and papules | (%X:XX ) XX |
| 4 - definite edema | |
| 5 - erythema, edema and papules | <i>_</i> |
| 6 - vesicular eruption | xx ( xx.x%) |
| 7 - strong reaction spreading beyond application | xx ( xx.x%) |
| 2116 | |
| Week 24 | |
| u | XX |
| 0 - no evidence of irritation | xx ( xx.x%) |
| 1 - minimal erythema, barely perceptible | xx ( xx.x%) |
| 2 - definite erythema, readily visible; minimal | xx ( xx.x%) |
| edema or minimal popular response | |
| 3 - erythema and papules | xx ( xx.x%) |
| 4 - definite edema | xx ( xx.x%) |
| 5 - erythema, edema and papules | xx ( xx.x%) |
| 6 - vesicular eruption | xx ( xx.x%) |
| 7 - strong reaction spreading beyond application | xx ( xx.x%) |
| Site | |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.2: Summary of Local Tolerability (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% (N=xx) | | XX | $XX (XX, X^{0})$ | XX ( XX.X%) | ) xx | | _ \ | XX (XX.X''0) | $XX (XX, X^{0/0})$ | XX (XX.X%) | ) xx | | | XX | XX ( XX.X%) | XX ( XX.X%) | ) xx | | XX ( XX.X%) | XX ( XX.X%) | XX ( XX.X <sup>0</sup> / <sub>0</sub> ) | XX ( XX.X%) | ) xx |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Investigator Local Tolerability Dermal Response | Week 36 | n | 0 - no evidence of irritation | 1 - minimal erythema, barely perceptible | 2 - definite erythema, readily visible; minimal | edema or minimal popular response | 3 - erythema and papules | 4 - definite edema | 5 - erythema, edema and papules | 6 - vesicular eruption | 7 - strong reaction spreading beyond application | site | Week 52 | n | 0 - no evidence of irritation | 1 - minimal erythema, barely perceptible | 2 - definite erythema, readily visible; minimal | edema or minimal popular response | 3 - erythema and papules | 4 - definite edema | 5 - erythema, edema and papules | 6 - vesicular eruption | 7 - strong reaction spreading beyond application |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.3: Summary of Local Tolerability (Safety Population)


| | ARO | ARQ-151-202: Kollumilast Cream 0.5% | ım 0.3% |
|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream | ARQ-151-201:<br>Vehicle Cream | Total |
| Investigator Local Tolerability Dermal Response<br>Baseline | (N=xx) | (xx=N) | (XX=N) |
| n | XX | XX | XX |
| 0 - no evidence of irritation | xx ( xx.x%) | $XX (XX.X^{0})$ | $xx (xx.x^{0})$ |
| 1 - minimal erythema, barely perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - definite erythema, readily visible; minimal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 - erythema and namiles | (%x xx ) xx | (%x xx ) xx | (%x:xx ) xx |
| 4 - definite edema | _ | _ | <i>-</i> |
| 5 - erythema, edema and namiles | <i>-</i> | <i>-</i> | <i>-</i> |
| 6 - vesicular eruption | <i>-</i> | <i>-</i> | <i>-</i> |
| 7 - strong reaction spreading beyond application | <i>_</i> | <i>_</i> | <i></i> |
| site | | | |
| Week 4 | | | |
| n | XX | XX | XX |
| 0 - no evidence of irritation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 - minimal erythema, barely perceptible | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 - definite erythema, readily visible; minimal | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0/0})$ |
| edema or minimal popular response | | | |
| 3 - erythema and papules | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| 4 - definite edema | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 5 - erythema, edema and papules | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6 - vesicular eruption | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 7 - strong reaction spreading beyond application | XX ( XX.X%) | xx ( xx.x%) | (xx.x) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.3: Summary of Local Tolerability (Safety Population) 

| | ARO- | ARO-151-202: Roflumilast Cream 0.3% | eam 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201:<br>Vehicle Cream | | |
| Investigator Local Tolorability Dermal Resnonse | Roflumilast Cream | and Cohort 2 $(N=xx)$ | | Total (N=xx) |
| Week 12 | (VV LT) | (WY AT) | | (www.tr) |
| n | XX | XX | XX | |
| 0 - no evidence of irritation | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | xx.x% |
| 1 - minimal erythema, barely perceptible | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | xx.x% |
| 2 - definite erythema, readily visible; minimal | xx ( xx.x%) | $xx (xx.x^{0})$ | ) xx | xx.x%) |
| edema or minimal popular response | | | | |
| 3 - erythema and papules | xx ( xx.x%) | $xx (xx.x^{0})$ | ) xx | xx.x% |
| 4 - definite edema | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | xx.x%) |
| 5 - erythema, edema and papules | xx ( xx.x%) | (xx.x) | ) xx | xx.x% |
| 6 - vesicular eruption | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | xx.x%) |
| 7 - strong reaction spreading beyond application | xx ( xx.x%) | (x, x, x, x) | ) xx | xx.x%) |
| site | | | | |
| Week 24 | | | | |
| n | XX | XX | XX | |
| 0 - no evidence of irritation | xx ( xx.x%) | xx ( xx.x%) | ) xx | (%x.xx |
| 1 - minimal erythema, barely perceptible | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x% |
| 2 - definite erythema, readily visible; minimal | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | xx.x%) |
| edema or minimal popular response | | | | |
| 3 - erythema and papules | xx ( xx.x%) | xx ( xx.x%) | ) xx | xx.x% |
| 4 - definite edema | xx ( xx.x%) | $XX (XX.X^{0})$ | ) xx | xx.x%) |
| 5 - erythema, edema and papules | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | xx.x%) |
| 6 - vesicular eruption | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | xx.x%) |
| 7 - strong reaction spreading beyond application | xx ( xx.x%) | $xx (xx.x^{0})$ | ) xx | xx.x%) |
| site | | | | |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME\(DATE\,TIME\)

Table 14.3.1.1.3: Summary of Local Tolerability (Safety Population) 

| | | | ARQ-151-201: | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream | -201:<br>t Cream | Vehicle Cream and Cohort 2 | Total |
| Investigator Local Tolerability Dermal Response | (X = X) | (X | (N=xx) | (N=XX) |
| Week 36 | | | | |
| n | XX | | XX | XX |
| 0 - no evidence of irritation | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 1 - minimal erythema, barely perceptible | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 2 - definite erythema, readily visible; minimal | ( xx.x ) xx | | ( xx.xx ) xx | xx ( xx.x%) |
| edema or minimal popular response | | | | |
| 3 - erythema and papules | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 4 - definite edema | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 5 - erythema, edema and papules | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 6 - vesicular eruption | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 7 - strong reaction spreading beyond application | XX ( XX.X%) | _ | xx ( xx.x%) | xx ( xx.x%) |
| site | | | | |
| Week 52 | | | | |
| n | XX | | XX | XX |
| 0 - no evidence of irritation | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 1 - minimal erythema, barely perceptible | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 2 - definite erythema, readily visible; minimal | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| edema or minimal popular response | | | | |
| 3 - erythema and papules | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 4 - definite edema | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 5 - erythema, edema and papules | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 6 - vesicular eruption | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) |
| 7 - strong reaction spreading beyond application | (%x:xx) xx | | (%x:xx ) xx | (%X.XX) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.1.2.1: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population: Cohort 1) 

| | | ARO-151-202: Rc | ARO-151-202: Roflumilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | |
| | Roflumilast Cream 0. | Roflumilast Cream 0.3% Roflumilast Cream 0.15% | Vehicle Cream | Total |
| Patient Health Questionnaire Depression Scale | (N=xx) | (N=xx) | (N=xx) | (N=XX) |
| Baseline | | | | |
| n | XX | XX | XX | XX |
| None - Minimal Depression (0 to 4) | (xx.x) xx.x | xx ( xx.x%) | xx ( xx.x%) | $(xx.x^{0/2})$ |
| Mild Depression (5 to 9) | (xx.x) ( $xx.x$ ) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | (xx.x) (xx.x) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Moderately Severe Depression (15 to 19) | (xx.x) ( $xx.x$ ) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | (0%x.xx ) xx | xx ( xx.x%) |
| Week 4 | | | | |
| n | XX | XX | XX | XX |
| None - Minimal Depression (0 to 4) | (xx.x) (xx.x) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Mild Depression (5 to 9) | (xx.x) (xx.x) | xx (xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | (xx.x) ( $xx.x$ ) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Moderately Severe Depression (15 to 19) | (xx.x) ( $xx.x$ ) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | XX ( XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | | | |
| n | XX | XX | XX | XX |
| None - Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | $xx (xx.x^{0})$ | xx (xx.x) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | $xx (xx.x^{0})$ | xx (xx.x) | xx ( xx.x%) |
| Moderately Severe Depression (15 to 19) | (xx.x) (xx.x) | xx (xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | (0%x.xx (xx) | xx ( xx.x%) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME\(DATE\,TIME\)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.1.2.1: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population: Cohort 1) 

| | | ARO-151-202: RG | ARO-151-202; Roflumilast Cream 0.3% | | |
|---|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201: ARQ-151-201:<br>Roflumilast Cream 0.3% Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | | Total |
| Patient Health Questionnaire Depression Scale | (N=xx) | (N=XX) | (N=xx) | | (N=xx) |
| Week 24 | | | | | |
| n<br>Mone Minimal Democration (0 to 4) | , | , | XX xx / xx | XX | (%)0 |
| Mild Denression (5 to 9) | (0/V.X.) XX X $(0/V.X.)$ XX | (%x xx ) xx<br>(xx xx ) xx | $(0/2)^{-1}$ | YY | (%x xx x%) |
| Moderate Depression (10 to 14) | _ | <i>_</i> | _ | XX | (%X:XX |
| Moderately Severe Depression (15 to 19) | <i>-</i> | <i>_</i> | <i>_</i> | ) xx | (%X.XX |
| Severe Depression (20 to 24) | xx ( xx.x%) | XX ( XX.X%) | xx ( xx.x%) | ) xx | xx.x%) |
| Week 36 | | | | | |
| n | XX | XX | XX | XX | |
| None - Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | ) xx | xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | ) xx | xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | ) xx | xx.x%) |
| Moderately Severe Depression (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | ) xx | xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) | ) xx | xx.x%) |
| Week 52 | | | | | |
| n | XX | XX | XX | XX | |
| None - Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | (%X.XX |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | ) xx | xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | ) xx | xx.x%) |
| Moderately Severe Depression (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | ) xx | xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | (x, x, x, x) | ) xx | xx.x%) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.3.1.2.2: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population: Cohort 2) 

| $\overline{5}$ |
|----------------|
| $_{\rm jo}$ |
| _ |
| e. |
| age |
| Ξ. |

| Roflumilast Cream 0.3% $(N=xx)$ | xx (xx.x%) | xx<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
|---|---|---|---|
| Patient Health Questionnaire Depression Scale | Baseline n None - Minimal Depression ( 0 to 4) Mild Depression (5 to 9) Moderate Depression (10 to 14) Moderately Severe Depression (15 to 19) Severe Depression (20 to 24) | Week 4 n None - Minimal Depression ( 0 to 4) Mild Depression (5 to 9) Moderate Depression (10 to 14) Moderately Severe Depression (15 to 19) Severe Depression (20 to 24) | Week 12 n None - Minimal Depression ( 0 to 4) Mild Depression (5 to 9) Moderate Depression (10 to 14) Moderately Severe Depression (15 to 19) Severe Depression (20 to 24) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.2.2: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population: Cohort 2) 

| $\widehat{z}$ |
|---------------|
| ot |
| $\sim$ |
| age |
| ್ಷ |

| .3% | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | | XX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | | XX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | | XX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Patient Health Questionnaire Depression Scale | Week 24 | n | None - Minimal Depression (0 to 4) | Mild Depression (5 to 9) | Moderate Depression (10 to 14) | Moderately Severe Depression (15 to 19) | Severe Depression (20 to 24) | Week 36 | n | None - Minimal Depression (0 to 4) | Mild Depression (5 to 9) | Moderate Depression (10 to 14) | Moderately Severe Depression (15 to 19) | Severe Depression (20 to 24) | Week 52 | n | None - Minimal Depression (0 to 4) | Mild Depression (5 to 9) | Moderate Depression (10 to 14) | Moderately Severe Depression (15 to 19) | Severe Depression (20 to 24) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.2.3: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population)


| | ARC | ARO-151-202: Roflumilast Cream 0.3% | am 0.3% |
|---|---|---|---|
| Patient Health Questionnaire Depression Scale | ARQ-151-201:<br>Roflumilast Cream<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2<br>(N=xx) | Total (N=xx) |
| Baseline<br>n | XX | XX | XX |
| None - Minimal Depression (0 to 4) | $XX (XX.X^{0})$ | $xx (xx.x^{0})$ | $XX (XX.X^{0})$ |
| Mild Depression (5 to 9) | $(xx.x^{0})$ | (xx.x) xx $(xx.x)$ | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe Depression (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| Week 4 | | | |
| n | XX | XX | XX |
| None - Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe Depression (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 | | | |
| n | xx | XX | XX |
| None - Minimal Depression (0 to 4) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild Depression (5 to 9) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Depression (10 to 14) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderately Severe Depression (15 to 19) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Depression (20 to 24) | xx ( xx.x%) | (0.000) XX $(0.000)$ XX | $XX (XX.X^{0})$ |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME\(DATE\,TIME\)

Table 14.3.1.2.3: Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) (Safety Population)


| | | ARO-1 | 51-202: Roff | ARQ-151-202: Roflumilast Cream 0.3% | .3% | | |
|---|---|---|---|---|---|---|---|
| Patient Health Questionnaire Depression Scale | AI<br>Rofi | ARQ-151-201:<br>Roflumilast Cream<br>(N=xx) | ARQ-1<br>Vehicle<br>and Co | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2<br>(N=xx) | | Total<br>(N=xx) | ı |
| Week 24<br>n | X | | XX | | × | | |
| None - Minimal Depression (0 to 4) | $\overline{}$ | xx.x%) | $\overline{}$ | | $\overline{}$ | XX.X% | |
| Mild Depression (5 to 9) | ) xx | xx.x%) | <u> </u> | | <u> </u> | xx.x%) | |
| Moderate Depression (10 to 14)<br>Moderate V Severe Depression (15 to 19) | ) XX | XX.X%)<br>xx x%) | (%x.xx) xx | | XX | XX.X%) | |
| Severe Depression (20 to 24) | | XX.X%) | | | | (%x.xx | |
| Week 36 | | | | | | | |
| n | XX | | XX | | XX | | |
| None - Minimal Depression (0 to 4) | ) xx | xx.x%) | xx ( xx.x%) | | ) xx | xx.x%) | |
| Mild Depression (5 to 9) | ) xx | xx.x%) | xx ( xx.x%) | | ) xx | xx.x%) | |
| Moderate Depression (10 to 14) | ) xx | xx.xx%) | xx ( xx.x%) | | ) xx | xx.x%) | |
| Moderately Severe Depression (15 to 19) | ) xx | xx.x%) | xx ( xx.x%) | | ) xx | xx.x%) | |
| Severe Depression (20 to 24) | ) xx | xx.x%) | xx ( xx.x%) | | ) xx | (%X.XX | |
| Week 52 | | | | | | | |
| п | XX | | XX | | xx | | |
| None - Minimal Depression (0 to 4) | ) xx | xx.x%) | xx ( xx.x%) | | ) xx | xx.x%) | |
| Mild Depression (5 to 9) | ) xx | xx.x%) | (%x.xx ) xx | | ) xx | xx.x%) | |
| Moderate Depression (10 to 14) | ) xx | xx.x%) | (%x.xx ) xx | | ) xx | xx.x%) | |
| Moderately Severe Depression (15 to 19) | ) xx | xx.x%) | (%x.xx) xx | | ) xx | (%X.XX | |
| Severe Depression (20 to 24) | ) xx | xx.x%) | xx ( xx.x%) | (%) | ) xx | xx.x%) | |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME\(DATE\,TIME\)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.3.1.3.1: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population: Cohort 1)

(Page 1 of 8)

PHQ-8 for (ARQ-151-201: Roflumilast Cream 0.3%)

| | | | | | | Week 4 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Baseline | | None | | Mild | | Moderate | Moderate | Moderately Severe | | Severe |
| None | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | xx ) xx | (%X.XX | ) xx | (%X.XX |
| Mild | XX | (%x.xx) | X | (%x.xx) | XX | (%x.xx) | xx ) xx | (%x.xx | xx ( | (%X.XX |
| Moderate | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | xx ) xx | (%x.xx | XX | (%X.XX |
| Moderately Severe | XX | (%x.xx ) | X | (%x.xx) | XX | ( xx.xx ) | xx ) xx | (%x.xx | xx | (%x.xx |
| Severe | XX | (%x.xx) | X | (%x.xx) | X | ( xx.xx ) | xx ) xx | (%X.XX | ) xx | (%X.XX |
| | | | | | | Week 12 | | | | |
| Baseline | | None | | Mild | | Moderate | Moderate | Moderately Severe | | Severe |
| None | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | xx ) xx | (%x.xx | ) xx | (%X.XX |
| Mild | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | xx ) xx | (%x.xx | xx ( | (%x.xx |
| Moderate | XX | (%x.xx) | XX | (%x.xx ) | XX | ( xx.xx %) | xx ) xx | xx.x%) | ) xx | (%x.xx |
| Moderately Severe | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx) | xx ) xx | (%x.xx | ) xx | (%x.xx |
| Severe | XX | ( xx.xx ) | X | ( xx.xx ) | X | ( xx.x%) | xx ) xx | (%x.xx | ) xx | (%X.XX |
| | | | | | | Week 24 | | | | |
| <u>Baseline</u> | | None | | Mild | | Moderate | Moderate | Moderately Severe | | Severe |
| None | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx) | xx ) xx | (%X.XX | ) xx | (%X.XX |
| Mild | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx) | xx ) xx | (%x.xx | ) xx | (%x.xx |
| Moderate | XX | (%x.xx) | XX | (%x.xx) | XX | ( xx.xx %) | xx ) xx | xx.x%) | ) xx | xx.x%) |
| Moderately Severe | XX | (%x.xx ) | XX | (%x.xx ) | XX | (%x.xx) | xx ) xx | (%x.xx | ) xx | (%x.xx |
| Severe | XX | (%x:xx ) | XX | (%x.xx ) | XX | (%x.xx) | xx ) xx | (%X.XX | ) xx | (%X.XX |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study.

SOURCE: USERNAME\SPONSOR\PROJECTYJOBNAME (DATE,TIME)

Table 14.3.1.3.1: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population: Cohort 1)

(Page 2 of 8)

Week 36

PHQ-8 for (ARQ-151-201: Roflumilast Cream 0.3%)

| <u>Baseline</u> | None | Mild | Moderate | Moderately Severe | <b>O</b> I | Severe |
|---|---|---|---|---|---|---|
| None | xx ( xx.x%) | ( xx.x%) xx | xx ( xx.x%) | ( XX.X%) XX | ) xx | (%x.xx |
| Mild | xx ( xx.x%) | ( xx.x%) | xx ( xx.x%) | ( xx.x%) | ) xx | (%x.xx |
| Moderate | xx ( xx.x%) | ( xx.x%) xx | xx ( xx.x%) | ( XX.X%) XX | ) xx | %x.xx |
| Moderately Severe | xx ( xx.x%) | ( xx.x%) xx | xx ( xx.x%) | ( xx.x%) | )<br>XX | %x.xx |
| Severe | xx ( xx.x%) | ( xx.x%) xx | ( xx.x%) | xx ( xx.x%) | XX | xx.xx(%) |
| | | | Week 52 | | | |
| <u>Baseline</u> | None | Mild | Moderate | Moderately Severe | 6)1 | Severe |
| None | xx ( xx.x%) | (xx.x) xx | ( xx.xx ) xx | $(xx.x^{0})$ | ) xx | xx.xx |
| Mild | xx ( xx.x%) | (xx.x) xx | xx ( xx.x%) | (xx.x) (xx.x%) | ) xx | (%x.xx) |
| Moderate | xx ( xx.x%) | (%x.xx) xx | ( xx.x ) xx | xx ( xx.x%) | )<br>XX | xx.x% |
| Moderately Severe | xx ( xx.x%) | ( xx.x%) | xx ( xx.x%) | ( xx.x%) | ) xx | xx.x% |
| Severe | xx ( xx.x%) | (xx.x) xx | ( xx.x ) xx | (XX.XX) | ) xx | %x.xx |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note to Programmer - Repeat for each treatment group (ARQ-151-201: Roflumilast Cream 0.15%; ARQ-151-201: Vehicle Cream; Total)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.1.3.2: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population: Cohort 2)


| PHQ-8 for (Roflumilast Cream 0.3%) | | | | | | Week 4 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Bacalina | | None | | M:13 | | Moderate | Moderately Severe | | Correre | |
| None | XX | (%x xx ) | XX | (%x xx ) | XX | ( xx x%) | $xx = (xx x^{0/6})$ | ×× | | |
| Mild | X | (%X:XX) | X | (%X:XX) | X | (%X::XX<br>) | | X | (%x:xx) | |
| Moderate | X | ( xx.xx ) | × | ( xx.x%) | × | ( xx.xx ) | <i>-</i> | X | (%x.xx) | |
| Moderately Severe | XX | (%x.xx ) | XX | (%x.xx ) | X | (%x.xx) | $(xx.x^{0})$ | XX | (%x.xx) | |
| Severe | XX | ( xx.xx ) | XX | (%x.xx) | X | ( xx.xx ) | xx ( xx.x%) | X | (%x.xx) | |
| | | | | | | Week 12 | | | | |
| Baseline | | None | | Mild | | Moderate | Moderately Severe | 431 | Severe | |
| None | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | (xx.x) xx | XX | (%x.xx ) | |
| Mild | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | ( xx.x%) | XX | (%x.xx ) | |
| Moderate | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | (xx.x) xx | XX | (%x.xx) | |
| Moderately Severe | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | ( xx.x%) | XX | (%x.xx) | |
| Severe | XX | ( xx.x%) | XX | ( xx.x%) | X | (%x.xx ) | $xx (xx.x^{0})$ | XX | (%x.xx) | |
| | | | | | | Week 24 | | | | |
| Baseline | | None | | Mild | | Moderate | Moderately Severe | 431 | Severe | ] |
| None | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | ( xx.x%) | XX | (%x.xx ) | |
| Mild | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | xx (xx.x%) | XX | (%x.xx ) | |
| Moderate | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx) | xx (xx.x) | XX | (%x.xx ) | |
| Moderately Severe | X | (%x.xx ) | XX | (%x.xx ) | X | (%x.xx) | xx (xx.x%) | XX | (%x.xx ) | |
| Severe | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | ( xx.xy ) xx | XX | (%x.xx ) | |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14); Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.3.2: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population: Cohort 2)


| | | | | | Week 36 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Baseline | None | | Mild | | Moderate | Moc | Moderately Severe | lc) | Severe | |
| None | ( xx.x%) | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | |
| Mild | ( xx.x%) | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | |
| Moderate | ( xx.x%) | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx | XX | (%x.xx) | |
| Moderately Severe | ( xx.x ) xx | XX | (%x.xx ) | XX | ( xx.xx ) | XX | (%x.xx) | XX | (%x.xx) | |
| Severe | xx ( xx.x%) | XX | ( xx.xx ) | XX | ( xx.xx ) | XX | (0%x.xx | XX | (%x.xx) | |
| | | | | | Week 52 | | | | | |
| Baseline | None | | Mild | | Moderate | Moc | Moderately Severe | (DI | Severe | ĺ |
| None | xx ( xx.x%) | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | |
| Mild | xx ( xx.x%) | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | |
| Moderate | xx ( xx.x%) | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | |
| Moderately Severe | ( xx.x%) | XX | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) | |
| Severe | xx ( xx.x%) | XX | (%x.xx) | XX | ( xx.xx ) | XX | (%x.xx) | XX | (%x.xx) | |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14); Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note to Programmer - Do not repeat for any other treatements.

Table 14.3.1.3.3: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population)


| ream) |
|------------|
| CC |
| oflumilas |
| ~ |
| RQ-151-201 |
| -151- |
| ARC |
| 8 for ( |
| PHQ. |

| | | | | | Week 4 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| aseline | None | | Mild | | Moderate | Mo | Moderately Severe | <u>ere</u> | | Severe |
| None | xx ( xx.x. <sup>9</sup> %) | xx (0 | (%x.xx) | XX | (%x.xx) | XX | ( xx.xx ) | XX | $\overline{}$ | (%X.XX |
| Mild | xx (xx.x%) | XX (0 | $\overline{}$ | XX | (%x.xx) | X | (%x.xx) | XX | $\overline{}$ | (%x.xx |
| Moderate | xx. ( xx.x.%) | xx (0 | ( xx.x%) | XX | ( xx.xx %) | XX | (%x.xx) | XX | $\overline{}$ | (%x.xx |
| Moderately Severe | (%x.xx ) xx | xx (0 | $\overline{}$ | XX | (%x.xx) | XX | (%x.xx) | XX | $\overline{}$ | (%X.XX |
| Severe | (%x.xx) xx | xx (0 | $\overline{}$ | XX | ( xx.xx ) | X | (%x.xx) | X | $\smile$ | (%X.XX |
| | | | | | Week 12 | | | | | |
| aseline | None | | $\overline{\text{Mild}}$ | | <u>Moderate</u> | Mo | Moderately Severe | <u>ere</u> | | Severe |
| None | (%x.xx ) xx | xx (0 | ( xx.x%) | XX | ( xx.xx %) | XX | (%x.xx) | XX | $\overline{}$ | (%x.xx |
| Mild | xx ( xx.x%) | xx (0 | $\overline{}$ | XX | ( xx.xx %) | XX | (%x.xx) | XX | $\overline{}$ | (%x.xx |
| Moderate | xx ( xx.x%) | xx (0 | $\overline{}$ | XX | ( xx.xx %) | XX | (%x.xx ) | XX | $\overline{}$ | (%x.xx |
| Moderately Severe | xx ( xx.x%) | xx (0 | ( xx.x%) | XX | (%x.xx) | XX | (%x.xx ) | XX | $\overline{}$ | (%X.XX |
| Severe | xx (xx.x%) | xx (0 | ( xx.xx ) | XX | ( xx.xx ) | X | ( xx.xx ) | XX | $\overline{}$ | (%x.xx |
| | | | | | Week 24 | | | | | |
| aseline | None | | Mild | | Moderate | Mo | Moderately Severe | <u>sre</u> | | Severe |
| None | xx ( xx.x%) | xx (0 | (%x.xx ) | XX | (%x.xx) | XX | (%x.xx ) | XX | $\overline{}$ | (%X.XX |
| Mild | xx ( xx.x%) | xx (0 | $\overline{}$ | XX | (%x.xx) | XX | (%x.xx ) | XX | $\overline{}$ | (%X.XX |
| Moderate | xx ( xx.x%) | xx (0 | $\overline{}$ | XX | (%x.xx) | XX | (%x.xx ) | XX | $\overline{}$ | (%X.XX |
| Moderately Severe | xx ( xx.x%) | xx (0 | $\overline{}$ | XX | (%x.xx) | XX | (%x.xx ) | XX | $\overline{}$ | (%x.xx |
| Severe | (%x.xx) xx | xx (0 | ( xx.x%) | XX | (%x.xx) | X | (%x.xx ) | XX | $\overline{}$ | (%x.xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTYJOBNAME (DATE,TIME)

Table 14.3.1.3.3: Shift Summary of Patient Health Questionnaire Depression Scale Assessments (PHQ-8) by Treatment Group (Safety Population)


| eam) |
|--------------|
| umilast Cro |
| -201: Rofi |
| (ARQ-151-201 |
| PHQ-8 for |

| , | | | | | Week 36 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| <u>Baseline</u> | None | | Mild | | Moderate | Mo | Moderately Severe | <u>sre</u> | Severe |
| None | xx ( xx.x%) | ) xx | (%x.xx | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx) |
| Mild | xx ( xx.x%) | ) xx | (%x.xx) | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx ) |
| Moderate | xx ( xx.x%) | ) xx | (%x.xx | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx ) |
| Moderately Severe | xx ( xx.x%) | ) xx | (%x.xx | XX | (%x.xx) | XX | (%x.xx) | XX | (%x.xx) |
| Severe | xx ( xx.x%) | ) xx | xx.x%) | XX | (%x.xx) | XX | (%x.xx) | XX | ( xx.xx ) |
| | | | | | Week 52 | | | | |
| Baseline | None | | Mild | | Moderate | Mo | Moderately Severe | ere. | Severe |
| None | xx ( xx.x%) | ) xx | (%x.xx | XX | (%x.xx ) | XX | (%x.xx ) | XX | (%x.xx ) |
| Mild | xx ( xx.x%) | ) xx | (%x.xx | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx) |
| Moderate | xx ( xx.x%) | ) xx | (%x.xx | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx ) |
| Moderately Severe | xx ( xx.x%) | ) xx | (%x.xx | XX | (%x.xx) | XX | (%x.xx ) | XX | (%x.xx ) |
| Severe | xx ( xx.x%) | ) xx | (%x.xx | XX | (%x.xx ) | XX | (%x.xx ) | XX | (%x.xx) |

Note: None = Minimal Depression (0 to 4); Mild = Mild Depression (5 to 9); Moderate = Moderate Depression (10 to 14);

Moderately Severe = Moderately Severe Depression (15 to 19); Severe = Severe Depression (20 to 24).

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note to Programmer - Repeat for each treatment group (ARQ-151-201: Vehicle Cream and Cohort 2; Total)
Table 14.3.1.4.1.1: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Inurious Behavior without Suicidal Intent Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population: Cohort 1)

| | | | | ARQ-151-202: Roflumilast Cream 0.3% | oflumilast C | ream 0.3% | | |
|---|---|---|---|---|---|---|---|---|
| | A<br>Roffin | ARQ-151-201: ARQ-151-201: Refumiliset Cream 0 3% Refumiliset Cream 0 15% | A<br>Roflim | ARQ-151-201:<br>milast Cream 0 15% | ARQ-<br>Vebicl | ARQ-151-201:<br>Vehicle Cream | | Total |
| Events During Treatment | TOTAL | (N=XX) | | (N=xx) | (N | N=xx) | | (N=XX) |
| Suicidal Ideation (1-5) | ) XX | xx.x%) | ) xx | xx.x%) | xx ( xx.x%) | (0/X | ) xx | XX.X%) |
| 1) Wish to be dead | ) xx | (%X.XX | ) xx | (%X.XX | xx ( xx.) | xx.xx%) | ) xx | (%X.XX |
| 2) Non-specific active suicidal thoughts | ) XX | (%X.XX | ) XX | (%X.XX | xx ( xx | (%X.XX | ) xx | (%X.XX |
| 3) Active suicidal ideation with any methods | ) xx | (%X.XX | ) xx | (%X.XX | xx ( xx.) | xx.x%) | ) xx | (%X.XX |
| (not plan) without intent to act | , | | , | | | | , | |
| 4) Active suicidal ideation with some intent to | ) xx | xx ( xx.x%) | ) xx | (%x.xx | xx ( xx.x%) | (%X | ) xx | (%X.XX |
| act, without specific plan | | | | | | | | |
| 5) Active suicidal ideation with specific plan | ) xx | (%x.xx) | ) xx | (%X.XX) | xx ( xx.x%) | (%x | ) xx | XX.X% |
| and intent | | | | | | | | |
| Suicidal Behavior (6-10) | ) xx | xx.x%) | ) xx | XX.X%) | xx (xx.) | xx.x%) | ) xx | xx.x%) |
| 6) Preparatory acts or behavior | ) xx | (%X.XX | ) xx | (%X.XX | xx ( xx.) | (%X.XX | ) xx | xx.x%) |
| 7) Aborted attempt | ) xx | (%X.XX | ) xx | XX.X% | xx ( xx.) | (%X.XX | ) xx | xx.x%) |
| 8) Interrupted attempt | ) xx | XX.X%) | ) xx | XX.X% | xx ( xx.) | (%X.XX | ) xx | xx.x%) |
| 9) Non-fatal suicide attempt | ) xx | (%X.XX | ) xx | XX.X%) | xx ( xx.) | (%X.XX | ) xx | xx.x%) |
| 10) Completed Suicide | ) xx | (%X:XX | ) xx | XX.X%) | xx ( xx.x%) | (%x | ) xx | xx.x%) |
| Suicidal Ideation or Behavior (1-10) | ) xx | ( , xx.x ) xx | ) xx | xx ( xx.x%) | xx ( xx.x%) | (%x | ) xx | xx ( xx.x%) |
| Self-injurious behavior without suicidal intent | ) xx | xx ( xx.x%) | ) xx | xx ( xx.x%) | (%x.xx ) xx | (%x | ) xx | ( XX.X%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.4.1.2: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Inurious Behavior without Suicidal Intent Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population: Cohort 1)

| 9 | | | |
|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| Events During Treatment | Suicidal Ideation (1-5) 1) Wish to be dead 2) Non-specific active suicidal thoughts 3) Active suicidal ideation with any methods (not plan) without intent to act 4) Active suicidal ideation with some intent to act, without specific plan 5) Active suicidal ideation with specific plan and intent | Suicidal Behavior (6-10) 6) Preparatory acts or behavior 7) Aborted attempt 8) Interrupted attempt 9) Non-fatal suicide attempt 10) Completed Suicide | Suicidal Ideation or Behavior (1-10) Self-injurious behavior without suicidal intent |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.4.1.3: Number of Patients with Suicidal Ideation, Suicidal Behavior, and Self-Inurious Behavior without Suicidal Intent Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment (Safety Population)

| | | ARQ-151-201: | |
|---|---|---|---|
| | ARQ-151-201: | Vehicle Cream | , |
| | Roflumilast Cream | and Cohort 2 | Total |
| Events During Treatment | (N=xx) | (N=xx) | (N=xx) |
| Suicidal Ideation (1-5) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1) Wish to be dead | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 2) Non-specific active suicidal thoughts | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 3) Active suicidal ideation with any methods | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| (not plan) without intent to act | | | |
| 4) Active suicidal ideation with some intent to | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | xx ( xx.x%) |
| act, without specific plan | | | |
| 5) Active suicidal ideation with specific plan | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| and intent | | | |
| Suicidal Behavior (6-10) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 6) Preparatory acts or behavior | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 7) Aborted attempt | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x) |
| 8) Interrupted attempt | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x) |
| 9) Non-fatal suicide attempt | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ |
| 10) Completed Suicide | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Suicidal Ideation or Behavior (1-10) | XX ( XX.X%) | xx ( xx.x%) | XX (XX.X%) |
| Self-injurious behavior without suicidal intent | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.4.2.1: Number of Patients with Suicidal-Related Treatment-Emergent Events Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment

(Safety Population: Cohort 1)

| | provement in suicidal ideation at endpoint xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) | nergence of serious suicidal ideation | ARQ-151-202: Roflumilast Cream 0.3%<br>ARQ-151-201: ARQ-151-201: | , <u> </u> | z | 2-151-201: icle Cream N=xx) | | 151-201: 151-201: Cream 0.15% =xx) n <sup>a</sup> (%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | Roffum N | 151-201:<br>t Cream 0.3%<br>=xx) | Roflumilas (N XX | Treatment-Emergent (TE) Events TE suicidal ideation (1-5) compared to recent history <sup>b</sup> TE serious suicidal ideation (0-3 to 4-5) compared to recent history <sup>c</sup> Emergence of serious suicidal ideation (0 to 4-5) compared to recent history <sup>d</sup> Improvement in suicidal ideation at endpoint |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx | al ideation xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx it history d | mbared to recent history o | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | (X XX (XX.X%) | | (%x.xx) xx x | X | xx (xx.x%) | XX | xx ( xx.x%) | × | ent history <sup>b</sup> serious suicidal ideation (0-3 to 4-5) |
| idal ideation (0-3 to 4-5) $xx xx(xx.x\%)$ | idal ideation (0-3 to 4-5) $xx xx(xx.x\%)$ $xx xx(xx.x\%)$ $xx xx(xx.x\%)$ $xx xx(xx.x\%)$ $xx$ erious suicidal ideation $xx xx(xx.x\%)$ | idal ideation (0-3 to 4-5) $xx - xx (xx.x\%) = xx - xx (xx.x\%)$ $xx - xx (xx.x\%) = xx - xx (xx.x\%)$ | Roflumilast Cream 0.3% Roflumilast Cream 0.15% Vehicle Cream To $\frac{(N=xx)}{N}$ | (x x ( xx.x%) | | | XX | | XX | xx (xx.x%) | XX | suicidal ideation (1-5) compared to |
| ation (1-5) compared to xx | ation (1-5) compared to $xx xx(xx.x\%)$ | ation (1-5) compared to xx xx (xx.x%) xx xx (xx.x%) idal ideation (0-3 to 4-5) xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) xx xx (xx.x%) | Roflumilast Cream 0.15% Vehicle Cream | (N=xx)<br>n <sup>a</sup> (%) | Z | N=xx)<br>n <sup>a</sup> (%) | Z | =xx)<br>n <sup>a</sup> (%) | Z)<br>Z | =xx)<br>n <sup>a</sup> (%) | Z<br>Z | tment-Emergent (TE) Events |
| ed to $ \frac{(N=xx)}{N} = \frac{(N=xx)}{xx(xx.x\%)} = \frac{(N=xx)}{N} = \frac{(N=xx)}{xx(xx.x\%)} = \frac{(N=xx)}{N} = \frac{(N=xx)}{xx(xx.x\%)} = \frac{(N=xx)}{N} = ($ | ed to $ \frac{(N=xx)}{N} = \frac{(N=xx)}{xx} $ | ed to $ \frac{(N=xx)}{N} = \frac{(N=xx)}{xx} = (N=x$ | ANC-121-201: | Total | | <pre>&lt;-131-201. icle Cream</pre> | | Cream 0.15% | | t Cream 0.3% | Roflumilas | |

Note: Restricted to subjects with at least one post-treatment C-SSRS assessment.

- <sup>a</sup> Counts reflect numbers of subjects who experienced the event at least once post-treatment.
- <sup>b</sup> N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is non-missing and <5.
- N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is
  - d N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is
    - N=Number of subjects whose suicidal ideation score is non-missing and >0 just prior to treatment.
- <sup>f</sup> N=Number of subjects with at least one post-baseline C-SSRS assessment and who did not have suicidal behavior (6-10) prior to treatment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.1.4.2.2: Number of Patients with Suicidal-Related Treatment-Emergent Events Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment

(Safety Population: Cohort 2)

| Roflumilast Cream 0.3% $\frac{(N=xx)}{N}$ | XX (XX.X%) XX (XX.X%) | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) | xx xx (xx.x%) |
|---|---|---|---|---|---|
| Treatment-Emergent (TE) Events | TE suicidal ideation (1-5) compared to recent history <sup>b</sup> | TE serious suicidal ideation (0-3 to 4-5) compared to recent history $^{\circ}$ | Emergence of serious suicidal ideation (0 to 4-5) compared to recent history <sup>d</sup> | Improvement in suicidal ideation at endpoint compared with baselined <sup>e</sup> | Emergence of suicidal behavior (6-10) compared to all prior history <sup>f</sup> |

Note: Restricted to subjects with at least one post-treatment C-SSRS assessment.

- <sup>a</sup> Counts reflect numbers of subjects who experienced the event at least once post-treatment.
- <sup>b</sup> N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is non-missing and <5.
  - N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is
    - d N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is
- <sup>e</sup> N=Number of subjects whose suicidal ideation score is non-missing and >0 just prior to treatment.
- <sup>f</sup> N=Number of subjects with at least one post-baseline C-SSRS assessment and who did not have suicidal behavior (6-10) prior to treatment.

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.3.1.4.2.3: Number of Patients with Suicidal-Related Treatment-Emergent Events Based on the Columbia-Suicide Severity Rating Scale (C-SSRS) During Treatment

(Safety Population)

| Treatment-Emergent (TE) Events | ARQ-1<br>Roflumi | ARQ-151-201: Roflumilast Cream | ARQ-1<br>Vehicl | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: Vehicle Cream and Cohort 2 | | Total (N=xx) |
|---|---|---|---|---|---|---|
| | Z | n <sup>a</sup> (%) | z | n <sup>a</sup> (%) | z | n <sup>a</sup> (%) |
| TE suicidal ideation (1-5) compared to recent history <sup>b</sup> | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) |
| TE serious suicidal ideation (0-3 to 4-5) compared to recent history $^{\circ}$ | XX | xx xx (xx.x%) | XX | xx xx (xx.x%) | XX | xx xx (xx.x%) |
| Emergence of serious suicidal ideation (0 to 4-5) compared to recent history <sup>d</sup> | XX | xx xx (xx.x%) | XX | xx ( xx.x%) | XX | xx (xx.x%) |
| Improvement in suicidal ideation at endpoint compared with baselined ° | XX | xx xx (xx.x%) | XX | ( xx.x ) xx | XX | xx (xx.x%) |
| Emergence of suicidal behavior (6-10) compared to all prior history $^{\rm f}$ | XX | xx xx (xx.x%) | XX | xx xx (xx.x%) | XX | xx xx (xx.x%) |

Note: Restricted to subjects with at least one post-treatment C-SSRS assessment.

<sup>a</sup> Counts reflect numbers of subjects who experienced the event at least once post-treatment.

<sup>&</sup>lt;sup>b</sup> N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is non-missing and <5.

<sup>&</sup>lt;sup>d</sup> N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is c N=Number of subjects with at least one post-baseline suicidal ideation score and whose maximum C-SSRS suicidal ideation score during the past 6 months is

<sup>&</sup>lt;sup>e</sup> N=Number of subjects whose suicidal ideation score is non-missing and >0 just prior to treatment.

<sup>&</sup>lt;sup>f</sup> N=Number of subjects with at least one post-baseline C-SSRS assessment and who did not have suicidal behavior (6-10) prior to treatment. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.2.1.1.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population: Cohort 1)

| | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Creat (N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|
| Number (%) of Subjects Reporting At Least<br>One TEAE | XX ( XX.X <sup>9</sup> / <sub>0</sub> ) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of TEAEs | XX | XX | XX | XX |
| Number (%) of Subjects Reporting At Least<br>One Serious Adverse Event | (%X.XX ) XX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | XX | XX | XX | XX |
| Number (%) of Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects who Discontinued<br>Study Drug due to Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity by Subject | | | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | $(xx.x^{0})$ |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | | |
| Likely | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ |
| Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (xx.xx) xx |
| Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (XX,XX) |
| Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (XX,XX) |
| Unrelated | xx ( xx.x%) | xx ( xx.x%) | ( xx.xx ) xx | (XX,XX) |

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.1.1.2: Summary of Post Active Treatment-Emergent Adverse Events Characteristics (Safety Population: Cohort 1)


Table 14.3.2.1.2: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population: Cohort 2)

| | Roflumilast<br>(N= | Roflumilast Cream $0.3\%$ $(N=xx)$ |
|---|---|---|
| Number (%) of Subjects Reporting At Least<br>One TEAE<br>Number of TEAEs | xx ( xx.x%) xx | (x,x%) |
| Number (%) of Subjects Reporting At Least<br>One Serious Adverse Event<br>Number of Serious TEAEs | x ) xx | xx.x%) |
| Number (%) of Subjects who Died | x ) xx | xx.x%) |
| Number (%) of Subjects who Discontinued<br>Study Drug due to Adverse Event | xx ( xx.x%) | (X.X%) |
| Maximum Severity by Subject Grade 5 | $\sim$ | $\mathbf{x}\mathbf{x}.\mathbf{x}\%$ |
| Grade 3 | x ) xx | XX.X%) |
| Grade 2<br>Grade 1 | $\sim$ | xx.x%)<br>xx.x%) |
| Maximum Relationship by Subject Likely Probably Possibly Unlikely Unrelated | x x x x x x x x x x x x x x x x x x x | xx.x%) xx.x%) xx.x%) xx.x%) xx.x%) |

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.2.1.3.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population)

| | ARO-151 | ARO-151-202: Roflumilast Cream 0.3% | |
|---|---|---|---|
| | ARO-151-201: | ARQ-151-201:<br>Vehicle Cream | |
| | Roflumilast Cream | and Cohort 2 | Total |
| ļ | (N=xx) | (N=xx) | (N=xx) |
| Number (%) of Subjects Reporting At Least | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of TEAEs | XX | XX | XX |
| Number (%) of Subjects Reporting At Least<br>One Serious Adverse Event | xx ( xx.x <sup>0</sup> / <sub>0</sub> ) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | XX | XX | XX |
| Number (%) of Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects who Discontinued<br>Study Drug due to Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity by Subject | | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x <sup>0</sup> %) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | |
| Likely | xx ( xx.x%) | xx ( xx.x <sup>0</sup> %) | xx ( xx.x%) |
| Probably | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Possibly | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Unrelated | xx ( xx.x%) | (%X.XX ) XX | xx ( xx.x%) |

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Repeat Table 14.3.2.1.3.1.: Summary of Treatment Emergent Adverse Events Characteristics and update footnote to:

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.1.3.2: Summary of Post Active Treatment-Emergent Adverse Events Characteristics (Safety Population)

Table 14.3.2.2.1.1: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 1)


Note: MedDRA dictionary (Version xx)

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note to the programmer: Sort the table by descending total frequency of system organ class and descending total frequency of preferred terms within each system organ class. Sort all remaining AE tables in the same fashion.

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Table 14.3.2.2.1.2: Summary of Post Active Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 1)


| ARO-151-202: Roflumilast Cream 0.3% | ARQ-151-201: ARQ-151-201: ARQ-151-201: | Roflumilast Cream 0.3% Roflumilast Cream 0.15% Vehicle Cream | $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | lass |
|---|---|---|---|---|
| | | System Organ Class <sup>a</sup> | Preferred Term | System Organ Class<br>Preferred Term |

Note: MedDRA dictionary (Version xx)

Note: Post active treatment-emergent adverse event defined as event with an onset on or after the date of the first dose of active study drug application in either ARQ-151-201 or ARQ-151-202 study.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Table 14.3.2.2.: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 2)

| Roflumilast Cream $0.3\%$ $(N=xx)$ | xx ( xx.x%)<br>xx ( xx.x%) |
|---|---|
| System Organ Class <sup>a</sup> Preferred Term | System Organ Class<br>Preferred Term |

Note: MedDRA dictionary (Version xx)

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Table 14.3.2.2.3.1: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)


Note: MedDRA dictionary (Version xx)

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note to the programmer: Sort the table by alphabetical order of system organ class and descending total frequency of preferred terms within each system organ class. Sort all remaining AE tables in the same fashion.

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Repeat Table 14.3.2.2.3.1.: Summary of Treatment Emergent Adverse Events by MedDRA System Organ Class and Preferred Term and update footnote to:

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202..

For the following tables:

Table 14.3.2.2.3.2: Summary of Post Active Treatment-Emergent Adverse Events System Organ Class and Preferred Term (Safety Population)

Table 14.3.2.3.1.1: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population: Cohort 1)


| | | | ARQ-151-202: Kotlumilast Cream 0.5% | umilast Cream 0.5% | | |
|---|---|---|---|---|---|---|
| | | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | | |
| System Organ Class <sup>a</sup> | | Roflumilast Cream 0.3% | Roflumilast Cream 0.15% | Vehicle Cream | Tc | Total |
| Preferred Term | Severity | (N=XX) | (N=xx) | (N=xx) | N. | (N=xx) |
| System Organ Class | Grade 5 | xx ( xx.x%) | XX ( XX.X%) | xx ( xx.x%) | x ( x | xx.x%) |
| ) | Grade 4 | xx (xx.x%) | xx ( xx.x%) | (xx.x) xx. $(xx.x)$ | x ) xx | (%X.XX |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | (XX, XX) XX | x ( x | (%x.xx |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | (XX, XX, X) | x ) xx | xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | x ( x | xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | x ) xx | xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | x ) xx | xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | $XX (XX.X^{0})$ | x ) xx | xx.x%) |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | x ) xx | xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | x ) xx | (%x.xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study.

MedDRA dictionary (Version xx)

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in

either ARQ-151-201 or ARQ-151-202...

For the following tables:

Table 14.3.2.3.1.2: Summary of Post Active Treatment-Emergent Adverse Events by Severity (Safety Population: Cohort 1)


Table 14.3.2.3.2: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population: Cohort 2) (Page 1 of xx)

| .3% | | |
|---|---|---|
| Roflumilast Cream 0.3%<br>(N=xx) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| R Severity | Grade 5<br>Grade 4<br>Grade 3<br>Grade 2<br>Grade 1 | Grade 5<br>Grade 4<br>Grade 3<br>Grade 2<br>Grade 1 |
| System Organ Class <sup>a</sup><br>Preferred Term | System Organ Class | Preferred Term |

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application.

Table 14.3.2.3.3.1: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population) (Page 1 of xx)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study.


SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Repeat Table 14.3.2.3.3.1.: Summary of Treatment Emergent Adverse Events by Severity - and update footnote to:

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.3.3.2: Summary of Post Active Treatment-Emergent Adverse Events by Severity (Safety Population)

Table 14.3.2.4.1.1: Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population: Cohort 1) (Page 1 of xx)

| | | | ARQ-151-202: Roflumilast Cream 0.3% | umilast Cream 0.3% | |
|---|---|---|---|---|---|
| System Organ Class <sup>a</sup><br>Preferred Term | Relationship | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-201:<br>Roflumilast Cream 0.15%<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>(N=xx) | Total<br>(N=xx) |
| System Organ Class | Likely<br>Probably<br>Possibly<br>Unlikely | $\sim$ | | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx (x | |
| Preferred Term | Unrelated<br>Likelv | XX ( XX.X%) XX ( XX.X%) | xx ( xx.x%)<br>xx ( xx.x%) | XX ( XX.X%)<br>XX ( XX.X%) | XX ( XX.X%)<br>XX ( XX.X%) |
| | Probably Possibly Unlikely Unrelated | | x ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | x ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | |

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the strongest reported relationship.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study.

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.4.1.2: Summary of Post Active Treatment-Emergent Adverse Events by Relationship (Safety Population: Cohort 1)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.3.2.4.2: Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population: Cohort 2) (Page 1 of xx)

| Roflumilast Cream 0.3% (N=xx) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
|---|---|---|
| Relationship | Likely<br>Probably<br>Possibly<br>Unlikely<br>Unrelated | Likely<br>Probably<br>Possibly<br>Unlikely<br>Unrelated |
| System Organ Class <sup>a</sup><br>Preferred Term | System Organ Class | Preferred Term |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the strongest reported relationship.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application.

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.3.2.4.3.1: Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population) (Page 1 of xx)

| | | ARQ-15 | ARQ-151-202: Roflumilast Cream 0.3% | 0.3% |
|---|---|---|---|---|
| System Organ Class <sup>a</sup><br>Preferred Term | Relationship | ARQ-151-201:<br>Roflumilast Cream<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2<br>(N=xx) | Total (N=xx) |
| System Organ Class | Likely<br>Probably | (%x.xx ) xx (%x.xx) | $\begin{array}{ccc} XX.XX & XX \\ XX.XY & XX \end{array}$ | (%X.XX ) XX |
| | Possibly | , , | | |
| | Unlikely | xx ( xx.x <sup>0</sup> %) | xx (xx.x) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or

Preferred Term) subjects are counted once under the strongest reported relationship.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. MedDRA dictionary (Version xx)SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in

For the following tables:

either ARQ-151-201 or ARQ-151-202.:

Table 14.3.2.4.3.2: Summary of Post Active Treatment-Emergent Adverse Events by Relationship (Safety Population)


Table 14.3.2.5.1.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population: Cohort 1)

| | | ARQ-151-202: Roflumilast Cream 0.3% | ilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| | (N=xx) | (XX=N) | (N=xx) | (x = N) |
| Number (%) of Subjects Reporting At Least | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | XX | XX | XX | XX |
| Number (%) of Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects who Discontinued Study Drug due to Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Severity by Subject | | | | |
| Grade 5 | (xx.x) xx. $(xx.x)$ | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | (xx.x) xx.x | xx ( xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | (xx.x) xx.x | xx ( xx.x%) |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Grade 1 | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | | |
| Likely | (XX, XX, X) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Probably | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Possibly | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unrelated | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x <sup>0</sup> %) | xx ( xx.x%) |

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Repeat Table 14.3.2.5.1.1.: Summary of Treatment Emergent Serious Adverse Events Characteristics - and update footnote to:

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.5.1.2: Summary of Post Active Treatment-Emergent Serious Adverse Events Characteristics (Safety Population: Cohort 1)

Table 14.3.2.5.2: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population: Cohort 2)

| Roflumilast Cream 0.3% (N=xx) | xx ( xx.x%)<br>xx | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
|---|---|---|---|---|
| | Number (%) of Subjects Reporting At Least<br>One Serious Adverse Event<br>Number of Serious TEAEs | Number (%) of Subjects who Died | Number (%) of Subjects who Discontinued<br>Study Drug due to Adverse Event | Maximum Severity by Subject Grade 5 Grade 4 Grade 3 Grade 2 Grade 1 Maximum Relationship by Subject Likely Probably Possibly Unlikely Unrelated |

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.3.2.5.3.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)

| | ARO- | ARO-151-202: Roflumilast Cream 0.3% | .3% |
|---|---|---|---|
| | ARO-151-201: | ARQ-151-201:<br>Vehicle Cream | |
| | Roflumilast Cream | and Cohort 2 | Total |
| | (N=xx) | (N=XX) | (N=xx) |
| Number (%) of Subjects Reporting At Least<br>One Serious Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of Serious TEAEs | XX | XX | XX |
| Number (%) of Subjects who Died | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number (%) of Subjects who Discontinued<br>Study Drug due to Adverse Event | xx ( xx.x%) | ( , xx.x ) xx | xx ( xx.x%) |
| Maximum Severity by Subject | | | |
| Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Grade 3 | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ |
| Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Maximum Relationship by Subject | | | |
| Likely | xx ( xx.x%) | xx ( xx.x <sup>o</sup> %) | $xx (xx.x^{0})$ |
| Probably | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Possibly | xx ( xx.x%) | xx ( xx.x%) | $XX (XX.X^{0})$ |
| Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| Unrelated | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ |

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in

either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.5.3.2: Summary of Post Active Treatment-Emergent Serious Adverse Events Characteristics (Safety Population)

Table 14.3.2.6.1.1: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 1)


| n 0.3% Roflum xx | Roflu |
|-------------------|-------|
|-------------------|-------|

Note: MedDRA dictionary (Version xx)

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Repeat Table 14.3.2.6.1.1.: Summary of Treatment Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term- and update footnote to: Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.6.1.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 1)

Table 14.3.2.6.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population: Cohort 2)


| Roflumilast Cream 0.3% (N=xx) | xx ( xx.x%)<br>xx ( xx.x%) |
|---------------------------------|----------------------------|
| System Organ Class <sup>a</sup> | System Organ Class |
| Preferred Term | Preferred Term |

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once. Note: MedDRA dictionary (Version xx)

Table 14.3.2.6.3.1: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)


| | ARQ | ARQ-151-202: Rotlumilast Cream 0.3%<br>ARO-151-201· | n 0.3% |
|---|---|---|---|
| | ARQ-151-201: | Vehicle Cream | |
| System Organ Class <sup>a</sup> | Roflumilast Cream | and Cohort 2 | Total |
| Preferred Term | (xx=N) | (N=xx) | (N=xx) |
| System Organ Class<br>Preferred Term | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |

Note: MedDRA dictionary (Version xx)

Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

## 

Repeat Table 14.3.2.6.3.1: Summary of Treatment Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term- and update footnote to:

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.6.3.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)
Table 14.3.2.7.1.1: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population: Cohort 1) (Page 1 of xx)

| System Organ Class <sup>a</sup> Preferred Term Severity System Organ Class Grade 5 x | ABO-151-201 | | | | |
|---|---|---|---|---|---|
| Grade 5 | Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% $(N=xx)$ | ARQ-151-201:<br>Vehicle Cream | Total (N=xx) | <u> </u> |
| Grade 5 | (327, 11) | (222) | (333, 11) | 77 (1) | |
| | xx ( xx.x%) | xx ( xx.x <sup>0</sup> / <sub>0</sub> ) | xx ( xx.x%) | xx ( xx.x <sup>0</sup> %) | (%) |
| | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | xx ( xx.x%) | (%) |
| | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | xx ( xx.x%) | (%) |
| | (XX.XX) | xx ( xx.x%) | (%X.XX ) XX | (xx.x) | (%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (%) |
| Preferred Term Grade 5 x | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (%) |
| | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | xx ( xx.x%) | (%) |
| | XX (XX.X%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | $xx (xx.x^{0})$ | κ%) |
| | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ ) | xx ( xx.x%) | (%) |
| | xx ( xx.x%) | xx ( xx.x%) | (xx.x) ( $xx.x$ %) | xx ( xx.x%) | (%) |

Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization

<sup>(</sup>System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. MedDRA dictionary (Version xx)

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in

either ARQ-151-201 or ARQ-151-202..

For the following tables:

Table 14.3.2.7.1.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by Severity (Safety Population: Cohort 1)

Table 14.3.2.7.2: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population: Cohort 2) (Page 1 of xx)

| Roflumilast Cream $0.3\%$ $(N=xx)$ | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | XX ( XX.X%)<br>XX ( XX.X%)<br>XX ( XX.X%)<br>XX ( XX.X%)<br>XX ( XX.X%) |
|---|---|---|
| Severity | Grade 5<br>Grade 4<br>Grade 3<br>Grade 2<br>Grade 1 | Grade 5<br>Grade 4<br>Grade 3<br>Grade 2 |
| System Organ Class <sup>a</sup><br>Preferred Term | System Organ Class | Preferred Term |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application.


Table 14.3.2.7.3.1: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population) (Page 1 of xx)

| | | | ARO-151-201· | |
|---|---|---|---|---|
| System Organ Class <sup>a</sup> | Corrowity | ARQ-151-201:<br>Roflumilast Cream | Vehicle Cream and Cohort 2 | Total |
| rreierred Lerm | Severity | (XX=NI) | (XX=NI) | (XX=NI) |
| System Organ Class | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| | Grade 2 | XX ( XX.X%) | xx ( xx.x%) | (xx.xx) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Preferred Term | Grade 5 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 4 | XX ( XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 3 | xx ( xx.x%) | xx ( xx.x%) | $xx (xx.x^{0})$ |
| | Grade 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Grade 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study.

Repeat Table 14.3.2.7.3.1: Summary of Treatment Emergent Serious Adverse Events by Severity- and update footnote to:

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in

either ARQ-151-201 or ARQ-151-202.: For the following tables: Table 14.3.2.7.3.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by Severity (Safety Population)

Table 14.3.2.8.1.1: Summary of Treatment-Emergent Serious Adverse Events by Relationship (Safety Population: Cohort 1) (Page 1 of xx)

| | | | ARQ-151-202: Roflumilast Cream 0.3% | umilast Cream 0.3% | |
|---|---|---|---|---|---|
| 6 | | ARQ-151-201: | ARQ-151-201: | ARQ-151-201: | E |
| System Organ Class <sup>a</sup><br>Preferred Term | Relationship | Roflumilast Cream 0.3% (N=xx) | Rotlumilast Cream $0.15\%$<br>(N=xx) | Vehicle Cream<br>(N=xx) | Fotal (N=xx) |
| System Oroan Class | Likely | (%x xx ) xx | (%x xx ) xx | (%x xx ) xx | (%x xx ) xx |
| | Probably | _ ر | xx ( xx.x%) | () XX () XX () XX | xx ( xx.x%) |
| | Possibly | xx (xx.x%) | | | |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | | (xx.x) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | (%x.xx) xx | xx ( xx.x%) |
| Preferred Term | Likely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Probably | xx ( xx.x%) | xx ( xx.x%) | (xx.x) (xx.x/%) | xx ( xx.x%) |
| | Possibly | xx ( xx.x%) | xx ( xx.x%) | (xx.x) (xx.x/%) | xx (xx.x%) |
| | Unlikely | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Unrelated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the strongest reported relationship.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study.

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in

either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.8.1.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by Relationship (Safety Population: Cohort 1)


Table 14.3.2.8.2: Summary of Treatment-Emergent Serious Adverse Events by Relationship (Safety Population: Cohort 2) (Page 1 of xx)

| Roflumilast Cream 0.3% (N=xx) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
|---|---|---|
| Relationship | Likely<br>Probably<br>Possibly<br>Unlikely<br>Unrelated | Likely<br>Probably<br>Possibly<br>Unlikely<br>Unrelated |
| System Organ Class <sup>a</sup><br>Preferred Term | System Organ Class | Preferred Term |

SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the strongest reported relationship.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application.

Table 14.3.2.8.3.1: Summary of Treatment-Emergent Serious Adverse Events by Relationship (Safety Population) (Page 1 of xx)

| | | ARO | ARQ-151-202: Roflumilast Cream 0.3% | ım 0.3% |
|---|---|---|---|---|
| System Organ Class <sup>a</sup><br>Preferred Term | Relationship | ARQ-151-201:<br>Roflumilast Cream<br>(N=xx) | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2<br>(N=xx) | Total<br>(N=xx) |
| System Organ Class | Likely<br>Probably<br>Possibly<br>Unlikely | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| Preferred Term | Likely<br>Probably<br>Possibly<br>Unlikely | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | |

<sup>(</sup>System Organ Class or Preferred Term) subjects are counted once under the strongest reported relationship.

Note: Treatment-emergent adverse event defined as event with an onset on or after the date of the first study drug application in ARQ-151-202 study. <sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note: Post active treatment-emergent adverse event defined as event with an onset date on or after the date of first dose of active study drug in either ARQ-151-201 or ARQ-151-202.:

For the following tables:

Table 14.3.2.8.3.2: Summary of Post Active Treatment-Emergent Serious Adverse Events by Relationship (Safety Subjects)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.3.3.1.1.1: Summary of Chemistry Laboratory Results (Safety Population: Cohort 1) (Page 1 of xx)

| | | ARO-151-202: Roflumilast Cream 0.3% | milast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| <parameter> (<units>)</units></parameter> | (N=XX) | (XX=N) | (XX=N) | (N=XX) |
| Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XXX.X | XXX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Week 4 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XXX.X | XXX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.3.1.1.1: Summary of Chemistry Laboratory Results (Safety Population: Cohort 1) (Page 2 of xx)

| | | ARQ-151-202: Roflumilast Cream 0.3% | nilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| <parameter> (<units>)</units></parameter> | (N=xx) | (XX=N) | (N=XX) | (X=N) |
| Week 12 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Week 24 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

### CONFIDENTIAL

Table 14.3.3.1.1.1: Summary of Chemistry Laboratory Results (Safety Population: Cohort 1) (Page 3 of xx)

| | ARQ-151-201: | ARQ-151-202: Roflumilast Cream 0.3%<br>ARQ-151-201: ARQ-151-20 | nilast Cream 0.3%<br>ARQ-151-201: | |
|---|---|---|---|---|
| <parameter> (<units>)</units></parameter> | Roflumilast Cream 0.3% (N=xx) | Roflumilast Cream 0.15%<br>(N=xx) | Vehicle Cream<br>(N=xx) | Total<br>(N=xx) |
| Week 36 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XXX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Week 52 | | | | |
| u | XX | XX | XX | XX |
| Mean | XX.X | XXX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XXX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XXX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

For the following tables:

Table 14.3.3.1.2.1: Summary of Hematology Laboratory Results (Safety Population: Cohort 1) Table 14.3.3.1.3.1: Summary of Urinalysis Laboratory Results (Safety Population: Cohort 1)

Table 14.3.3.1.1.2: Summary of Chemistry Laboratory Results (Safety Population: Cohort 2) (Page 1 of xx)

| n 0.3% | | | |
|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | XX | XX | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.XX |
| <parameter> (<units>)</units></parameter> | Baseline<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. | Week 4 n Mean SD Median Min. to Max. | Change from Baseline<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. |

Table 14.3.3.1.1.2: Summary of Chemistry Laboratory Results (Safety Population: Cohort 2) (Page 2 of xx)

| Roflumilast Cream 0.3% (N=xx) | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX to XX | xx<br>xx.x<br>xx.xx<br>xx.xx<br>xx.x | xx<br>xx.x<br>xx.xx<br>xx.xx<br>xx.x | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX to XX |
|---|---|---|---|---|
| <parameter> (<units>)</units></parameter> | Week 12 n Mean SD Median Min. to Max. | Change from Baseline n Mean SD Median Min. to Max. | Week 24 n Mean SD Median Min. to Max. | Change from Baseline n Mean SD Median Min. to Max. |

Table 14.3.3.1.1.2: Summary of Chemistry Laboratory Results (Safety Population: Cohort 2) (Page 3 of xx)

| Roflumilast Cream 0.3% (N=xx) | XX<br>XX.XX<br>XX.XX<br>XX.XX | XXX<br>XX.XX<br>XX.XX<br>XX.XX | XXX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.X |
|---|---|---|---|---|
| <parameter> (<units>)</units></parameter> | Week 36 n Mean SD Median Min. to Max. | Change from Baseline n Mean SD Median Min. to Max. | Week 52 n Mean SD Median Min. to Max. | Change from Baseline n Mean SD Median Min. to Max. |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

### CONFIDENTIAL

### Repeat Table 14.3.3.1.1.2: Summary of Chemistry Laboratory Results

For the following tables:

Table 14.3.3.1.2.2: Summary of Hematology Laboratory Results (Safety Population: Cohort 2) Table 14.3.3.1.3.2: Summary of Urinalysis Laboratory Results (Safety Population: Cohort 2)

Table 14.3.3.1.1.3: Summary of Chemistry Laboratory Results (Safety Population)

| | ARQ-15 | ARQ-151-202: Roflumilast Cream 0.3% | 3% |
|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream | ARQ-151-201:<br>Vehicle Cream<br>and Cohort 2 | Total |
| <parameter> (<units>)</units></parameter> | (XX=N) | (XX=N) | (N=XX) |
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XXX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 4 | | | |
| u | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XXX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.3.1.1.3: Summary of Chemistry Laboratory Results (Safety Population)

| | ARQ-1 | ARQ-151-202: Roflumilast Cream 0.3% | .3% |
|---|---|---|---|
| | | ARQ-151-201: | |
| | ARQ-151-201:<br>Roflumilast Cream | Vehicle Cream<br>and Cohort 2 | Total |
| <parameter> (<units>)</units></parameter> | (N=xx) | (N=xx) | (N=xx) |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XXX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XXX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | XX to XX | xx to xx |
| Week 24 | | | |
| п | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XXX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XXX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XXX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.3.1.1.3: Summary of Chemistry Laboratory Results (Safety Population)

| | ARQ-1 | ARQ-151-202: Roflumilast Cream 0.3% | .3% |
|---|---|---|---|
| | | ARQ-151-201: | |
| | ARQ-151-201:<br>Roflumilast Cream | Vehicle Cream<br>and Cohort 2 | Total |
| <parameter> (<units>) Wood 36</units></parameter> | (N=xx) | (N=xx) | (N=xx) |
| n n | XX | XX | XX |
| Mean | X.X.X | xx.x | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 52 | | | |
| n | XX | xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XXXX | XX.X | xx.x |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

### Repeat Table 14.3.3.1.1.3: Summary of Chemistry Laboratory Results

For the following tables:

Table 14.3.3.1.2.3: Summary of Hematology Laboratory Results (Safety Population) Table 14.3.3.1.3.3: Summary of Urinalysis Laboratory Results (Safety Population)

Table 14.3.3.2.1.1: Shift Summary of Chemistry Lab Results (Safety Population: Cohort 1)

| <test name="">(<units>)</units></test> | | | | | Week 4 | | |
|---|---|---|---|---|---|---|---|
| , | | Rof | Roflumilast Cream 0.3% (N=xx) | .3% (N=xx) | Roffi | Roflumilast Cream 0.15% (N=xx) | 5% (N=xx) |
| | Baseline | BNL | WNL | ANL | BNL | MNL | ANL |
| | BNL | xx ( xx.x%) | (xx.x) | ( XX.X%) | (xx.x) | (XX) $(XX)$ | (xx)(x) |
| | WNL | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | ANL | xx( xx.x%) | xx(xx.xx) | xx(xx.x) | xx ( xx.x%) | $xx(xx.x^{0})$ | xx ( xx.x%) |
| | | | Vehicle Cream (N=xx) | N=xx) | | Total (N=xx) | |
| | Baseline | BNL | WNL | ANL | BNL | WNL | ANL |
| | BNL | xx ( xx.x%) | ( xx.x%) | ( XX.X. Xx) | ( xx.x%) | ( xx.x ) xx | ( xx.x%) |
| | WNL | xx ( xx.x%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | ANL | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

# Note to Programmer: Repeat for Visits: Week 12, Week 24, Week 36, Week 52

Repeat table 14.3.3.2.1.1 Shift Summary of Chemistry Lab Results

For the following tables:

Table 14.3.3.2.2.1: Shift Summary of Hematology Laboratory Results (Safety Population: Cohort 1) Table 14.3.3.2.3.1: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population: Cohort 1)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.3.2.1.2: Shift Summary of Chemistry Lab Results (Safety Population: Cohort 2)

| <units>)</units> |
|-----------------------|
| Name> ( |
| <test< td=""></test<> |

| =xx | ANL | xx.x% | xx.x% | xx.x% |
|---|---|---|---|---|
| .3% (N | | ) xx | ) xx | ) xx |
| oflumilast Cream 0.3% (N=xx) | WNL | xx.x% | xx.x% | xx.x% |
| lumila | ļ | ) xx | ) xx | ) xx |
| Rof | BNL | xx.x%) | xx.x% | (%X.XX |
| | | $\mathbf{x}\mathbf{x}$ | $\mathbf{x}\mathbf{x}$ | )xx |
| | Baseline | BNL | WNL | ANL |

Week 4

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Note to Programmer: Repeat for Visits: Week 12, Week 24, Week 36, Week 52

Repeat table 14.3.3.2.1.2 Shift Summary of Chemistry Lab Results

For the following tables:

Table 14.3.3.2.3.2: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population: Cohort 2) Table 14.3.3.2.2.2: Shift Summary of Hematology Laboratory Results (Safety Population: Cohort 2)

Table 14.3.3.2.1.3: Shift Summary of Chemistry Lab Results (Safety Population)

| ARQ-151-201: Vehicle ARQ-151-201: Vehicle ANL | <test name=""> (<units>)</units></test> | | | | • | Week 4 | | | |
|---|---|---|---|---|---|---|---|---|---|
| ARQ-151-201: Roflumilast Cream (N=xx) and Cohort 2 (N=xx) xx(xxxx%) xx(xxxxx%) xx(xxxxx%) xx(xxxxx%) xx | , | | | | | AR | Q-151-201: Vehic | sle Cream | |
| E BNL WNL ANL BNL WNL xx(xxx,%) | | | ARQ-151 | 1-201: Roflumila | st Cream (N=xx) | | and Cohort 2 (N | =xx | |
| xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) <th></th> <th>Baseline</th> <th></th> <th>MNL</th> <th>ANL</th> <th>BNL</th> <th>MNL</th> <th>ANL</th> <th></th> | | Baseline | | MNL | ANL | BNL | MNL | ANL | |
| xx( xx.x%) | | BNL | XX | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx ( xx.x%) | () |
| xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) Total (N=xx) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) | | WNL | xx(xx.x) | xx(xx) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx ( xx.x%) | () |
| Total (N=xx) BNL WNL WNL Xx ( xx.x%) xx ( xx.xx%) xx ( xx.xx% | | ANL | xx ( xx.x%) | | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | () |
| XX ( XX.X%) XX ( XX.X%) XX ( XX.X%) XX ( XX.X%) XX ( XX.X%) XX ( XX.X%) XX ( XX.X%) | | | | Total (N=x | x) | | | | |
| xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) xx( xx.x%) | | Baseline | | MNL | ANL | | | | |
| xx( xx.x%) xx( xx.x%)<br>xx( xx.x%) xx( xx.x%) | | BNL | xx ( | xx(xx.x) | xx ( xx.x%) | | | | |
| xx(xx.x%) xx(xx.x%) | | WNL | )xx | xx(xx.x) | xx(xx.x) | | | | |
| | | ANL | xx(xx.x) | xx(xx.x) | xx(xx.x) | | | | |

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

# Note to Programmer: Repeat for Visits: Week 12, Week 24, Week 36, Week 52

Repeat table 14.3.3.2.1.3 Shift Summary of Chemistry Lab Results

For the following tables:

Table 14.3.3.2.2.3: Shift Summary of Hematology Laboratory Results (Safety Population) Table 14.3.3.2.3.3: Shift Summary of Quantitative Urinalysis Laboratory Results (Safety Population)

Table 14.3.4.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population: Cohort 1)

| | | ARQ-151-202: Roflumilast Cream 0.3% | milast Cream 0.3% | |
|---|---|---|---|---|
| <parameter> (<units>)</units></parameter> | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-201:<br>Roflumilast Cream $0.15\%$ | ARQ-151-201: Vehicle Cream $(N=xx)$ | Total (N=xx) |
| | | (377) | (3777 ) 1 | (3747 ) 4 |
| Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | X.XX | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Week 24 | | | | |
| n | XX | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XXX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | X.XX | XX.X | X.XX | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.4.1: Summary of Electrocardiogram (ECG) Parameters (Safety Population: Cohort 1)

| | | ARQ-151-202: Roflumilast Cream 0.3% | ilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| <parameter> (<units>)</units></parameter> | (X=X) | (X=XX) | (N=xx) | (N=xx) |
| Week 52 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.4.2: Summary of Electrocardiogram (ECG) Parameters (Safety Population: Cohort 2)

| Roflumilast Cream $0.3\%$ (N=xx) | XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX XXX XXXX XXXX XXXX XXXX XXXX |
|---|---|---|---|
| <parameter> (<units>)</units></parameter> | Baseline n Mean SD Median Min. to Max. | Week 24 n Mean SD Median Min. to Max. | Change from Baseline n Mean SD Median Min. to Max. |

Table 14.3.4.2: Summary of Electrocardiogram (ECG) Parameters (Safety Population: Cohort 2) (Page 2 of xx)

| Roflumilast Cream 0.3% $(N=xx)$ | | XX | XX.X | XX.XX | XX.X | tx to xx | | XX | XX.X | XX.XX | XX.X | tx to xx |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Roflumila<br>(] | | | | | | | | | | | | |
| <parameter> (<units>)</units></parameter> | Week 52 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | u | Mean | SD | Median | Min. to Max. |

Table 14.3.4.3: Summary of Electrocardiogram (ECG) Parameters (Safety Population)

| | ARO-1 | ARO-151-202: Roflumilast Cream 0.3% | .3% |
|---|---|---|---|
| | ARO-151-201: | ARQ-151-201:<br>Vehicle Cream | |
| | Roflumilast Cream | and Cohort 2 | Total |
| <parameter> (<units>)</units></parameter> | (N=xx) | (N=xx) | (N=xx) |
| Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 24 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.4.3: Summary of Electrocardiogram (ECG) Parameters (Safety Population)

| ARQ-151-202: Roflumilast Cream 0.3% | ARQ-151-201:<br>Vehicle Cream | (N=xx) (N=xx) (N=xx) (N=xx) (N=xx) | | XX XX XX XX | XX.X XX.X | XX.XX XX.XX XX.XX | XX.X XX.X | xx to xx | | XX XX XX XX | XX.X XX.X XX.X | XX.XX XX.XX XX.XX | XX.X XX.X XX.X | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | <parameter> (<units>)</units></parameter> | Week 52 | п | Mean | SD | Median | Min. to Max. | Change from Baseline | n | Mean | SD | Median | Min to Mov |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.5.1.1: Summary of Vital Signs (Safety Population: Cohort 1) (Page 1 of xx)

| | | ARO-151-202: Roflumilast Cream 0.3% | nilast Cream 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-201:<br>Roffumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| <parameter> (<units>)</units></parameter> | (N=XX) | | | (N=XX) |
| Baseline | | | | |
| u | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Week 4 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | X.XX | XXX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.5.1.1: Summary of Vital Signs (Safety Population: Cohort 1) (Page 2 of xx)

| | ARO-151-201: | ARQ-151-202: Roflumilast Cream 0.3%<br>ARQ-151-201: ARQ-151-20 | nilast Cream 0.3%<br>ARO-151-201: | |
|---|---|---|---|---|
| <parameter> (<units>)</units></parameter> | Roflumilast Cream 0.3% (N=xx) | Roflumilast Cream 0.15% (N=xx) | Vehicle Cream<br>(N=xx) | Total (N=xx) |
| Week 12 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Week 24 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XXX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| u | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XXX.X | XXX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.5.1.1: Summary of Vital Signs (Safety Population: Cohort 1) (Page 3 of xx)

| | ARQ-151-201:<br>Roflumilast Cream 0.3% | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: ARQ-151-20 Roflumilast Cream 0.15% Vehicle Crean | nilast Cream 0.3% ARQ-151-201: Vehicle Cream | Total |
|---|---|---|---|---|
| <parameter> (<units>)</units></parameter> | (xx=N) | (xx=N) | (xx=N) | (x=N) |
| Week 36 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | X.X.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Week 52 | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | |
| n | XX | XX | XX | XX |
| Mean | XX.X | XXX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | X.XX | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.5.1.2: Summary of Vital Signs (Safety Population: Cohort 2) (Page 1 of xx)

| ream 0.3%<br>x) | XX | XX.XX<br>XX.XX | ) XX | | XX | XX.X | K.XX | XX.X | XX C | | XX | XX.X | K.XX | XX.X | XX C |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | | X | xx t | | | | X | | xx t | | | | CX | | XX tr |
| <parameter> (<units>)</units></parameter> | Baseline<br>n | Mean<br>SD<br>Medion | Min. to Max. | Week 4 | n | Mean | SD | Median | Min. to Max. | Change from Baseline | n | Mean | SD | Median | Min. to Max. |

Table 14.3.5.1.2: Summary of Vital Signs (Safety Population: Cohort 2) (Page 2 of xx)

| eam 0.3% | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.XX | xx<br>xx.x<br>xx.xx<br>xx.x xx xx.x xx.x xx.x xx | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.X | xx<br>xx.x<br>xx.xx<br>xx.xx<br>xx.x |
|---|---|---|---|---|
| Roflumilast Cream 0.3% (N=xx) | XX.X XX.XX XX.XX XX.XX | xx.x<br>xx.xx<br>xx.xx | XX.X XX.XX XX.XX XX.XX XX.XX | XX.X XX.XX XX.XX XX.XX |
| <parameter> (<units>)</units></parameter> | Week 12<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. | Change from Baseline<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. | Week 24<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. | Change from Baseline<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. |
Table 14.3.5.1.2: Summary of Vital Signs (Safety Population: Cohort 2) (Page 3 of xx)

| eam 0.3% | xx<br>xx.x<br>xx.xx<br>xx.xx<br>xx.xx | xx<br>xx.x<br>xx.xx<br>xx.x xx.x xx.x xx.x xx.x | XX<br>XX.X<br>XX.XX<br>XX.XX<br>XX.X | xx |
|---|---|---|---|---|
| Roflumilast Cream $0.3\%$ (N=xx) | XX.X XX.XX XX.XX XX.XX | xx.x<br>xx.xx<br>xx.xx | XX.XX XX.XX XX.XX XX.XX | XX.X XX.XX XX.XX XX.XX XX.X |
| <parameter> (<units>)</units></parameter> | Week 36<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. | Change from Baseline n Mean SD Median Min. to Max. | Week 52<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. | Change from Baseline<br>n<br>Mean<br>SD<br>Median<br>Min. to Max. |

TOOL. AN. 10-01.01 Statistical Analysis Plan Template

Table 14.3.5.1.3: Summary of Vital Signs (Safety Population)

| <pre><parameter> (<units>) Baseline</units></parameter></pre> | ARQ-151-201: Roflumilast Cream (N=xx) xx.x xx.x xx.x xx.x xx.x xx.x xx.x | ARQ-151-202: Roflumilast Cream 0.3% ARQ-151-201: Vehicle Cream and Cohort 2 (N=xx) xx xx.x | Total (N=xx) (N=xx) xxx xx.x xx.xx xx.x xx.x xx.x xx.x |
|---|---|---|---|
| nge from Baseline<br>n<br>Mean | XX XX XX | XX XXX | XX XXX |
| SD<br>Median<br>Min. to Max. | XX.XX<br>XX.X<br>XX to XX | XX.XX<br>XX.X<br>XX to XX | XX.XX<br>XX.X<br>XX to XX |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.3.5.1.3: Summary of Vital Signs (Safety Population)

| | ARQ-1 | ARQ-151-202: Roflumilast Cream 0.3% | .3% |
|---|---|---|---|
| | | ARQ-151-201: | |
| | ARQ-151-201:<br>Pofumilast Cream | Vehicle Cream | Total |
| <parameter> (<units>)</units></parameter> | | | (N=xx) |
| Week 12 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Week 24 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | |
| n | XX | XX | XX |
| Mean | XXXX | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XXXX | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.5.1.3: Summary of Vital Signs (Safety Population)

| <parameter> (<units>) Week 36 n</units></parameter> | | | |
|---|---|---|---|
| <units>)</units> | ARQ-151-201:<br>Roflumilast Cream | Vehicle Cream and Cohort 2 | Total |
| | (x = N) | (xx=N) | (N=xx) |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX |
| | XX.X | XX.X | XX.X |
| | xx to xx | xx to xx | xx to xx |
| Baseline | | | |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX |
| | XX.X | XX.X | XX.X |
| × | xx to xx | XX to XX | xx to xx |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX |
| | XX.X | XX.X | XX.X |
| | xx to xx | xx to xx | xx to xx |
| eline | | | |
| | XX | XX | XX |
| | XX.X | XX.X | XX.X |
| | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| ax. | xx to xx | xx to xx | xx to xx |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Table 14.3.5.2.1: Summary of Change in Body Weight Compared to Baseline (Safety Population: Cohort 1) 

| Change in Body Weight Compared to Baseline | ARQ-151-201:<br>Roflumilast Cream 0.3%<br>(N=xx) | ARQ-151-202: Ro<br>ARQ-151-201: ARQ-151-201:<br>Roflumilast Cream 0.3% Roflumilast Cream 0.15% (N=xx) | ARQ-151-202: Roflumilast Cream 0.3% Q-151-201: ARQ-151-201: st Cream 0.15% Vehicle Cream (N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Week 4 Lost >5% Body Weight Lost >10% Body Weight Maintained Body Weight Gained >5% Body Weight Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 12 Lost >5% Body Weight Lost >10% Body Weight Maintained Body Weight Gained >5% Body Weight Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 24 Lost >5% Body Weight Lost >10% Body Weight Maintained Body Weight Gained >5% Body Weight Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.3.5.2.1: Summary of Change in Body Weight Compared to Baseline (Safety Population: Cohort 1)


| | | | ARQ-151-202: Ro | ARQ-151-202: Roflumilast Cream 0.3% | |
|---|---|---|---|---|---|
| | ARQ-151-201:<br>Roflumilast Cream | -201:<br>ream 0.3% Rof | ARQ-151-201: ARQ-151-201: Roflumilast Cream 0.3% Roflumilast Cream 0.15% | ARQ-151-201:<br>Vehicle Cream | Total |
| Change in Body Weight Compared to Baseline | (X=X) | (X | (N=xx) | (xx=N) | (XX=N) |
| Week 36 | | | | | |
| Lost >5% Body Weight | (%x.xx) xx | | xx ( xx.x%) | ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | (%x.xx) xx | | xx ( xx.x%) | ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | (%x.xx) xx | | XX (XX.X%) | ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | | $(xx.x^{0})$ | (%X.XX ) XX | xx ( xx.x%) |
| Gained >10% Body Weight | (%x.xx ) xx | | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Week 52 | | | | | |
| Lost >5% Body Weight | (%x.xx) xx | | xx ( xx.x%) | ( xx.x%) | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | | ( XX.X <sup>0</sup> / <sub>0</sub> ) | xx ( xx.x%) | xx ( xx.x%) |
| Maintained Body Weight | (%x.xx) xx | | $(xx.x^{0})$ | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x, ) xx | | $(xx.x^{0})$ | xx (xx.x) | xx ( xx.x%) |
| Gained >10% Body Weight | (%x.xx ) xx | | ( xx.x%) | ( xx.x. ) xx | (xx.x) xx.x% |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECTJOBNAME (DATE,TIME)

Table 14.3.5.2.2: Summary of Change in Body Weight Compared to Baseline (Safety Population: Cohort 2) 

| Roflumilast Cream 0.3% $(N=xx)$ | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
|---|---|---|---|---|
| Change in Body Weight Compared to Baseline | Week 4 Lost >5% Body Weight Lost >10% Body Weight Maintained Body Weight Gained >5% Body Weight Gained >10% Body Weight | Week 12 Lost >5% Body Weight Lost >10% Body Weight Maintained Body Weight Gained >5% Body Weight Gained >10% Body Weight | Week 24 Lost >5% Body Weight Lost >10% Body Weight Maintained Body Weight Gained >5% Body Weight Gained >10% Body Weight | Week 36 Lost >5% Body Weight Lost >10% Body Weight Maintained Body Weight Gained >5% Body Weight Gained >10% Body Weight |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Table 14.3.5.2.2: Summary of Change in Body Weight Compared to Baseline (Safety Population: Cohort 2)

| | |
|---------------|--|

| Roflumilast Cream 0.3% $N=xx$ | | XX (XX.X%) | XX ( XX.X%) | XX ( XX.X%) | $XX (XX.X^{0})$ | xx ( xx.x%) |
|---|---|---|---|---|---|---|
| Change in Body Weight Compared to Baseline | Week 52 | Lost >5% Body Weight | Lost >10% Body Weight | Maintained Body Weight | Gained >5% Body Weight | Gained >10% Body Weight |

Table 14.3.5.2.3: Summary of Change in Body Weight Compared to Baseline (Safety Population)


| | ARO- | ARO-151-202: Roflumilast Cream 0.3% | am 0.3% | |
|---|---|---|---|---|
| | ARQ-151-201:<br>Roflimilast Cream | ARQ-151-201:<br>Vehicle Cream | | Total |
| Change in Body Weight Compared to Baseline | (N=XX) | | | N=XX) |
| Week 4 | _ | | _ | |
| Lost $>$ 5% Body Weight | _ \ | _ \ | _ \ | (%) |
| Lost >10% Body Weight | XX ( XX.X%) | (0,XX.XX) XX | XX ( XX.X%) | (%) |
| Maintained Body Weight | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (% |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (%) |
| Week 17 | | | | |
| WOCN 12 | | : | | |
| Lost >5% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (% |
| Lost>10% Body Weight | $xx (xx.x^{0})$ | xx ( xx.x%) | xx ( xx.x%) | (%) |
| Maintained Body Weight | xx (xx.x%) | xx ( xx.x%) | xx (xx.x) | (% |
| Gained >5% Body Weight | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) | (%) |
| Gained >10% Body Weight | xx ( xx.x%) | ( xx.x%) | xx ( xx.x%) | (%) |
| Week 24 | | | | |
| Lost >5% Body Weight | xx ( xx.x%) | $xx (xx.x^{0})$ | xx ( xx.x%) | (%) |
| Lost>10% Body Weight | $xx (xx.x^{0})$ | xx (xx.x) | xx ( xx.x%) | (% |
| Maintained Body Weight | $xx (xx.x^{0})$ | $xx (xx.x^{0})$ | xx ( xx.x%) | (% |
| Gained >5% Body Weight | $xx (xx.x^{0})$ | XX (XX.X) | xx ( xx.x%) | (% |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | (%) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.5.2.3: Summary of Change in Body Weight Compared to Baseline (Safety Population)


| | ARO- | ARQ-151-202: Roflumilast Cream 0.3% | am 0.3% |
|---|---|---|---|
| | ARQ-151-201: | ARQ-151-201:<br>Vehicle Cream | F |
| Change in Body Weight Compared to Baseline | Kollumlast Cream<br>(N=xx) | and Conort 2<br>(N=xx) | 1 Otal $(N=xx)$ |
| Week 36 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | (%X.XX ) XX | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | (xx.x) xx.x | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | (xx.x) xx.x | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | (xx.x) xx | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | XX ( XX.X%) |
| Week 52 | | | |
| Lost >5% Body Weight | xx ( xx.x%) | (xx.x) xx.x | xx ( xx.x%) |
| Lost >10% Body Weight | xx ( xx.x%) | (xx.x) xx.x | xx ( xx.x%) |
| Maintained Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Gained >5% Body Weight | xx ( xx.x%) | xx (xx.x) | xx ( xx.x%) |
| Gained >10% Body Weight | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.5.3.1: Shift Summary of Body Mass Index (BMI) Results (Safety Population: Cohort 1) 

| <b>Body Mass Index</b> | | | | | | | | | Last BMI Record | /II Rec | ord | | | | | | ĺ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Roflu | Roflumilast Cream 0.3% (N=xx) | $0.3^{\circ}$ | % (N=xx) | | | | | Roflu | Roflumilast Cream 0.15% (N=xx) | m0.15 | % (N=xx) | | |
| | <b>Baseline</b> | ר | Under | | Normal | | Over | Į | Obese | | Under | | Normal | | Over | | Obese |
| | Under | $\mathbf{x}$ $\mathbf{x}$ | (%x.x | x )xx | (%x.x | $\mathbf{x}\mathbf{x}$ | ( xx.xx%) | )xx | (%x.xx | )xx | XX.X% | )xx | (%X.XX | )xx | (%X.XX | )xx | xx( xx.x%) |
| | Normal | $\mathbf{x}$ $\mathbf{x}$ | (%x.x | x ) $xx$ | (%x.x | $\mathbf{x}\mathbf{x}$ | (%x.xx) | )xx | (%x.xx | )xx | (%x.xx | )xx | xx(xx.x) | )xx | xx(xx.x) | )xx | (%x.xx |
| | Over | $\mathbf{x}$ $\mathbf{x}$ | (%x.x | x ) $xx$ | (%x.x | $\mathbf{x}\mathbf{x}$ | ( xx.xx ) | )xx | xx ( xx.x%) | )xx | xx(xxx) | )xx | xx(xx.x) | )xx | xx(xx.x%) | )xx | xx(xx.x) |
| | Opese | xx (x | xx(xx.x%) $xx(x.x%)$ | x )xx | (%x.x | ( ) xx | xx ( xx.x%) | )xx | xx ( xx.x%) | )xx | (%x.xx) | )xx | xx( xx.x%) | )xx | (%X.XX | )xx | (%x.xx |
| | | | | > | Vehicle Cream (N=xx) | am (N | =xx) | | | | | | Total (N=xx) | N=xx) | | | |
| | Baseline | | Under | Z | Normal | | Over | | Obese | | Under | | Normal | | Over | | Obese |
| | Under | $\mathbf{x}$ $\mathbf{x}$ | xx(xx.x%) $xx(xx.x%)$ | x )xx | (%x.x | $\mathbf{x}\mathbf{x}$ | (x.xx) (xx) | )xx | (x.xx.)x; | )xx | ( xx.x%) | )xx | (xx.x%) | )xx | ( xx.x %) | )xx | (xx.xx) |
| | Normal | $\mathbf{x}$ $\mathbf{x}$ | (%x.x | x )xx | (%x.x | $\mathbf{x}\mathbf{x}$ | (%x.xx) | )xx | xx ( xx.x%) | )xx | xx.x% | $\mathbf{x}\mathbf{x}$ | (%x.xx) | )xx | ( xx.x%) | )xx | (%x.xx) |
| | Over | $\mathbf{x}$ $\mathbf{x}$ | (%x.x | x )xx | (%x.x | | (%x:xx) | )xx | xx.x%) | )xx | ( xx.xx ) | )xx | xx ( xx.x%) | )xx | xx(xx.x%) | )xx | (%x.xx) |
| | Opese | $\mathbf{x}$ $\mathbf{x}$ | (%x.x | x ) $xx$ | (%x.x | $\mathbf{x}\mathbf{x}$ | xx(xx.x) | )xx | ( xx.x%) | )xx | (xx.xx) | )xx | xx( xx.x%) | )xx | xx.x%) | )xx | xx(xx.x) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Note To Programmer: Repeat this page, with Highest BMI Record and Lowest BMI Record

Table 14.3.5.3.2: Shift Summary of Body Mass Index (BMI) Results (Safety Population: Cohort 2)

| <b>Body Mass Index</b> | | | | | Roflumilast Cr | Roflumilast Cream 0.3% (N=xx) | | | |
|---|---|---|---|---|---|---|---|---|---|
| • | • [ | | Lowest BMI Record | 3MI Record | | | Highest B | Highest BMI Record | |
| | Baseline | Under | Normal | Over | Opese | Under | Normal | Over | Obese |
| | Under xx | ( xx.xx ): | xx(xx.x) | xx(xx.x%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Normal xx | ( xx.x%) | xx(xx.x) | xx(xx.x%) | xx(xx.x%) | xx(xx.x) | xx(xx.x%) | xx(xx.x) | xx(xx.x) |
| | Over xx | ( xx.x%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| | Obese xx | ( xx.xx%) | xx(xx.x%) xx(xx.x%) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x%) |
| | | | Last BMI Record | Al Record | | | | | |
| | Baseline | Under | Normal | Over | Obese | | | | |
| | Under xx | ( xx.xx ): | xx(xx.x) | xx(xx.x) | xx(xx.x) | | | | |
| | Normal xx | ( xx.xx%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | | | | |
| | Over xx | ( xx.xx%) | xx(xx.x) | xx(xx) | xx(xx.x) | | | | |
| | Obese xx | ( xx.xx ): | xx(xx.x%) $xx(x.x%)$ | xx(xx.x) | xx ( xx.x%) | | | | |

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.5.3.3: Shift Summary of Body Mass Index (BMI) Results (Safety Population) 

| <b>Body Mass Index</b> | | | | | | Last BMI Record | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Al | RQ-151-201: Rof | ARQ-151-201: Roflumilast Cream (N=xx) | (=XX) | | AF | Q-151-201: V | ARQ-151-201: Vehicle Cream (N=xx) | (xx) | |
| | <b>Baseline</b> | Ü | Normal | Over | | Ü | Jnder | Normal | Over | | Obese |
| | Under x | (xx.xx) | $xx(xx.x^{0})$ | xx(xx.x) | xx(xx.x%) | XX XX. | (%x.xx) | xx(xx.x%) | xx(xx.x%) | ) XX | |
| | Normal x | (xx.xx) | xx(xx.x) | xx(xx.x) | xx(xx.x) | XX XX. | xx.x%) | xx(xx.x%) | xx(xxx) | )xx | (%x.xx |
| | Over x | (xx.xx) | xx(xx.x%) | xx(xx.x) | xx(xx.x) | xx(xx) | (%x: | xx(xx.x%) | xx(xxx) | | xx(xx.x) |
| | Obese | ( xx.x ) xx | xx(xx.x%) $xx(xx.x%)$ | xx( xx.x%) | xx(xx.x) | xx (xx. | xx.x%) | xx( xx.x%) | xx(xx) | | (%X.XX |
| | | | Total | Total $(N=xx)$ | | | | | | | |
| | Baseline | Under | Normal | Over | Obese | | | | | | |
| | Under x | (xx.xx) | xx(xx.x%) xx(xx.x%) | xx(xx.x) | xx(xx.x) | | | | | | |
| | Normal x | (xx.xx) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | | | | | |
| | Over | (xx.xx) | xx(xx.x%) | xx(xx.x) | xx(xx.x) | | | | | | |
| | Obese x | (xx.xx) | xx(xx.x) | xx(xx.x) | xx(xx.x) | | | | | | |

Note: BNL=Below Normal Limit, WNL=Within Normal Limit, ANL=Above Normal Limit.

Baseline is defined as the last observation prior to the first dose of Roflumilast cream in either the ARQ-151-201 or ARQ-151-202 study. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Note To Programmer: Repeat this page, with Highest BMI Record and Lowest BMI Record

#### 11. INDEX OF PLANNED LISTINGS

| Listing 16.2.1.1: End of Study Information | 304 |
|---|---|
| Listing 16.2.1.2: Discontinued Subjects | 305 |
| Listing 16.2.2.1: Inclusion/Exclusion Criteria Violations | 306 |
| Listing 16.2.2.2: Protocol Deviations | 307 |
| Listing 16.2.3: Analysis Populations | 308 |
| Listing 16.2.4.1: Subject Demographic Information | 309 |
| Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System O and Preferred Terms | _ |
| Listing 16.2.4.2.2: Medical/Surgical History | 311 |
| Listing 16.2.4.3.1: Unique Medication Names Coded to WHO-DD ATC Level 2 T Preferred Names | |
| Listing 16.2.4.3.2: Prior and Concomitant Medications | 313 |
| Listing 16.2.4.4.1: Unique Therapies and Procedures Coded to MedDRA System Cand Preferred Terms | _ |
| Listing 16.2.4.4.2: Prior and Concomitant Therapies and Procedures | 315 |
| Listing 16.2.4.5: Physical Examination | 316 |
| Listing 16.2.5.1: Study Visit Compliance | 317 |
| Listing 16.2.5.2: Drug Accountability | 318 |
| Listing 16.2.5.3: Study Drug Application | 319 |
| Listing 16.2.5.4: Dosing Compliance | 320 |
| Listing 16.2.5.5: Dosing Deviations | 321 |
| Listing 16.2.6.1: Investigator Global Assessment (IGA) | 322 |
| Listing 16.2.6.2: Body Surface Area (BSA) Involved with Psoriasis | 323 |
| Listing 16.2.6.3: Psoriasis Area and Severity Index (PASI) | 324 |
| Listing 16.2.6.7: Columbia-Suicide Severity Rating Scale (C-SSRS) | 325 |
| Listing 16.2.6.8.1: Patient Health Questionnaire Depression Scale (PHQ-8) Question Descriptions | |
| Listing 16.2.6.8.2: Patient Health Questionnaire Depression Scale (PHQ-8) | 327 |
| Listing 16.2.7.1.1: Investigator Local Tolerability Assessment | 328 |
| Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Class Preferred Terms | |
| Listing 16.2.7.2.2: Treatment-Emergent Adverse Events | 330 |
| TOOL.AN.10-01.01 Statistical Analysis Plan Template | Page <b>302</b> of <b>337</b> |

| Listing 16.2.7.2.3: Serious Adverse Events | 331 |
|---|---|
| Listing 16.2.7.2.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse Events | 332 |
| or Exeprienced an Adverse Event Resulting in Death | 332 |
| Listing 16.2.8.1: Urine Pregnancy Test Results | 333 |
| Listing 16.2.8.2: 12-lead Electrocardiogram Test Results | 334 |
| Listing 16.2.8.3.1: Vital Signs | 335 |
| Listing 16.2.8.3.2: Weight Loss/Gain >5% | 336 |

Listing 16.2.1.1: End of Study Information Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | F: Date of First Dose of Drug<br>L: Date of Last Dose of Drug | Primary Reason for Study<br>Completion/Discontinuation | Date of Completion/Discontinuation |
|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | F: xxxxxxxxx<br>L: xxxxxxxxxx | *************************************** | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| S: | F: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | *************************************** | xxxx xxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxxxxxxx<br>L: xxxxxxxxxxxxxxxxxxxxxxxxx | ***** **** **** **** | xxxx xxxxxxxx |

Note to programmer: concatenate 'Describe' text onto Primary Reason where applicable.

Listing 16.2.1.2: Discontinued Subjects Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | F: Date of First Dose of Drug<br>L: Date of Last Dose of Drug | Primary Reason for Study<br>Completion/Discontinuation | Date of Completion/Discontinuation |
|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | F: xxxxxxxxx<br>L: xxxxxxxxxx | *************************************** | XXXXXXXXXX |
| S: xxxxxx<br>A: xxxxx<br>E: xxxxxxxxx | F: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | *************************************** | xxxx xxxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | F: xxxxxxxxx<br>L: xxxxxxxxxxxxxxxxxxxxxxxxx | ***** **** **** **** | xxxx xxxxxxxx |

Listing 16.2.2.1: Inclusion/Exclusion Criteria Violations
Treatment Group

| YY) |
|----------|
| of<br>Of |
| e xx |
| (Page |

| | XXXXXXXX XXX XX XX XXXXXXXX XX XXXXXXXX | XXXXXXX XXXXXXXX X XXXXXXXXXX X X XXXXXX | XXXXXXX XXXX XXXX X XXXXXXXXX XX X XXXXX | XXXXXXXX XXXX XXXXX XXXXXXXXXXX XXXXXXX | XXX XXX XXXXXXXX X XX XXXXXXXXX X XX XX | XXXXXXX XXXX XXXX X X XXXXXXXXX XX X XXXX |
|---|---|---|---|---|---|---|
| Description | ****** * ***** *********************** | XXXXXX X XXXX XXXXXX | XXXXXX XXXX XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX XXXXXX XXXX XXXXXXXXXXXXXXXXXXXXX | XXXXX X XXXX XXXXXXXX | XXXXXX XXXX XXXX XXXX XXXX XXXX XXXX XXXX |
| Criterion<br>Identifier | × | × | × | ×× | × | ×× |
| Criterion<br>Category | ×××××××××××××××××××××××××××××××××××××× | ×××××××× | ××××××××××××××××××××××××××××××××××××××× | xxxxxxxx | XXXXXXXX | ××××××× |
| Eval | ××××××××××××××××××××××××××××××××××××××× | | ××××××××××××××××××××××××××××××××××××××× | | XXXXXXXX | |
| Age/Sex Eval | ×××× | | ×××× | | XXXX | |
| Subject | ××××× | | ××××× | | XXXXXX | |

Listing sorted by Subject, Criterion Category, and Criterion Identifier.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.2.2: Protocol Deviations Treatment Group (Page xx of yy)

TOOL. AN. 10-01.01 Statistical Analysis Plan Template

Listing 16.2.3: Analysis Populations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Population | Included | Reason(s) Excluded |
|---------|---------|------------|----------|-----------------------------|
| XXXXXX | XXXX | Safety | XX | XXXXXXX X XXXXXXX X XXXXXXX |
| ××××× | XXXX | Safety | ××× | |
| XXXXXX | ×××× | Safety | xxx | |

Listing sorted by Subject, and Population.

Listing 16.2.4.1: Subject Demographic Information (Page xx of yy)

| <pre>C: Childbearing Potential B: Birth Control Method</pre> | C: xx<br>B: | C: xxx<br>B: xxxxxxxxx xxxxxxxx | C: xxx<br>B: xxxx xxxxxxxxxxxxxxxxxxxxxxxxxx |
|---|---|---|---|
| R: Race<br>E: Ethnicity | R: XXXXX XX XXXXXXX<br>E: XXX XXXXXXXX XX | R: xxxxx<br>E: xxx xxxxxxxx xx | R: xxxxx<br>E: xxx xxxxxxx xx |
| Date/Time of<br>Informed Consent<br>Age at Consent | XXXX-XX-XXTXX:XX:XX | XXXX-XX-XXTXX:XX:XX | xxxx-xx-xxTxx:xx |
| D:<br>B: Date of Birth<br>S: Sex A: | B: xxxxxxxxx D:<br>S: xxxx A: | B: xxxxxxxxx D:<br>S: xxxxxx A: | B: xxxxxxxxx D:<br>S: xxxxxx A: |
| | xxxxxxx | ××××××××××××××××××××××××××××××××××××××× | xxxxxxx |
| Subject Eval | ××××× | ××××× | ××××× |

Listing 16.2.4.2.1: Unique Medical/Surgical History Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Condition/Surgery Verbatim Term |
|---|---|---|
| x xxx xxxxx | xxxx xxx xxxx | XXXX XXXXXXXX XX XXXXXX |
| | | XX XXXX XXX XXX |
| XXXXXXXX X XXXX | XXXXXXXX XXXXXXXX | XXXX XX XXXXXXXXX XXXXX |
| XXXX XXX XXX | XXXX XXX XXXX | XXXX XXXXXXX |
| | | XXXXXX XXXXXXXXXX |
| | | XXXXXX XX XXXXXXX XXXXXX |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by System Organ Class, Preferred Term, and Verbatim Term.

Listing 16.2.4.2.2: Medical/Surgical History Treatment Group (Page xx of yy)

| Subject Age/ | Age/Sex Eval | Condition/Surgery<br>Verbatim Term | P: MedDRA Preferred Term<br>S: MedDRA System Organ Class | S: Onset Date<br>E: End Date |
|---|---|---|---|---|
| ×××× | xxxxxxx | (***** ************ | P: xxxxxx xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | S: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | XXXXXXXX XXXXXXXX | P: xxxxxx xxxxxxxx<br>S: xxxxx xxxxxxxxxxxxx | S: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Medical Condition/Surgery, Start Date, and End Date.

Listing 16.2.4.3.1: Unique Medication Names Coded to WHO-DD ATC Level 2 Terms and Preferred Names (Page xx of yy)

| ATC Level 2 Term | Preferred Name | Medication Name | I: Indication<br>R: Route |
|---|---|---|---|
| XXXXXX XXXXXX | XXXXXXXXX | XXXXXXXXX | I: XXXXXXX XXXXXXXX R: XXXX |
| | × ××××××× | ×××××× | I: XXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | ××××××××××××××××××××××××××××××××××××××× | ××××××××××××××××××××××××××××××××××××××× | I: XXXXXXX XXXXXXXX XXXX XXXX XXXXX XXXXX XXXX |

Note: Preferred Name and ATC Level 2 Term map to the WHO-DD (Version March 1, 2018). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by ATC Level 2 Term, Preferred Name, Medication Name, Indication, and Route.

TOOL.AN.10-01.01 Statistical Analysis Plan Template


Listing 16.2.4.3.2: Prior and Concomitant Medications Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | M: Medication Name P: Preferred Name A: AIC Level 2 Term I: Indication | F: Date of First Dose<br>S: Start Date (Day) <sup>1</sup><br>E: End Date (Day) <sup>1</sup> | D: Dose<br>U: Units<br>F: Frequency<br>R: Route |
|---|---|---|---|---|---|
| ××××× | ×××× | ××××××××××××××××××××××××××××××××××××××× | M: xxxxxxxxxxxxxxx P: xxxxxxxxxxxxxxxxxx | F: xxxxxxxxxx<br>S: xxxxxxxxxxx<br>E: xxxxxxxxxxxxxxxxxxxxxxx | D: xx<br>U: xx<br>F: xxxx<br>R:xxxx |
| | | | M: xxxxxxxxxxxxxxx P: xxxxxxxxxxxxxxxxxx | F: XXXXXXXXXXXXXX S: XXXXXXXXXXXXXXXXXXX | D: xxxxx<br>U: xx<br>F: xx<br>R:xxxx |
| ××××× | ×<br>×<br>× | ××××××××××××××××××××××××××××××××××××××× | M: xxxxxxxxxxxxxxxx P: xxxxxxxxxxxxxxxxx | F: xxxxxxxxxx S: xxxxxxxxxx E: xxxxxxxxxxxxxxxxxxxxxxxx | D: xxx<br>U: xx<br>F: xx<br>R:xxxx |

Listing sorted by Subject, Start Date, End Date, Medication Name, Indication, and Route. If ongoing, include 'Ongoing' in place of End Date. Concatenate Topical Area Treated onto route where applicable.

¹ Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of dose + 1 for dates on or after first dose.
Note: Preferred Name and ATC Level 2 Term map to the WHO-DD (Version March 1, 2018).
SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.4.4.1: Unique Therapies and Procedures Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Procedure/Therapy Verbatim Term |
|---|---|---|
| XXXX XXX XXX | xxxx xxx xxxxx | xxxx |
| | | xxxxxx xx xxxxxxx |
| | | XXXXXX XX XXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| xxxx xxx xxxx | xxxx xxx xxxxx | XXXX |
| | | XXXXXX XXXXXXXXX |
| | | XXXXXX XXXXXXXXX |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, MedDRA Preferred Term, and Procedure/Therapy Verbatim Term.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Start Date, End Date, Procedure/Therapy, Indication. If ongoing, include 'Ongoing' in place of End Date.

Listing 16.2.4.5: Physical Examination Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | Visit | Date | Body System Assessed | Finding | Abnormal Finding<br>Specification |
|---|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXX | Heart<br>Lungs<br>Skin (Other than Psoriasis)<br><other, specify=""></other,> | XXXXXXXXX<br>XXXXX XXXXXX<br>XXXXXXXXX | ****** |
| | XXXXXXXXXX | XXXXXXXX | Heart<br>Lungs<br>Skin (Other than Psoriasis) | ************************************** | |
| | xx xxxx | XXXXXXXX | Heart<br>Lungs<br>Skin (Other than Psoriasis) | XXXXXXXXX<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| S: xxxxxx A: xxxxx E: xxxxxxxx | ****** | XXXXXXXX | Heart<br>Lungs<br>Skin (Other than Psoriasis) | ************************************** | ×××××× |
| | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXX | Heart<br>Lungs<br>Skin (Other than Psoriasis) | XXXXX XXXXX<br>XXXXXXXX<br>XXXXXXXXX | |
| | ×× ×××× | ×××××××××××××××××××××××××××××××××××××× | Heart<br>Lungs<br>Skin (Other than Psoriasis) | XXXXXXXX<br>XXXXX XXXXXXX | |

Listing sorted by Subject, Visit, Date, Body System Assessed.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.5.1: Study Visit Compliance Treatment Group (Page xx of yy)

| Subject Age/Sex | Eval | Visit | Visit Date | Study<br>Day¹ | Within Visit<br>Window | Days Out of<br>Window <sup>2</sup> | Reason<br>Not Done |
|---|---|---|---|---|---|---|---|
| | ××××××× | ****** | XXXXXXXXX | × × | XXX<br>XXX | | ×××××× |
| | | x xxxx | XXXXXXXXX | ×× | xxx | XXXX | |
| | XXXXXXXX | XXXXXXXXX | xxxxxxxxx to xxxxxxxxx | × | XXX | | |
| | | XXXXXXXX | XXXXXXXXX | × | XXX | | |
| | | x xxxx | XXXXXXXXX | ×× | ××× | | XX XXXXXXXX |
| | | × ×××× | ×××××××× | XX | XXX | | |
| | XXXXXXX | ×××××××× | ×××××××× | ×× | ××× | | |
| | | XXXXXXXX | XXXXXXXXX | × | ××× | | |
| | | X XXXX | XXXXXXXXX | ×× | XXX | | |

TOOL.AN.10-01.01 Statistical Analysis Plan Template

¹ Day is calculated as date - baseline date for dates prior to baseline visit. Otherwise, day is calculated as
date - baseline date + 1 for dates on or after baseline visit.
² Populated only for post baseline visits that are planned and out of window.
source: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Subject, Visit, Visit Date.

Listing 16.2.5.2: Drug Accountability
Treatment Group
(Page xx of yy)

| Subject | Age/Sex | Evaluable | Kit Number | Date<br>Dispensed | Date<br>Returned | Tube ID | Dispensed<br>Weight (g) | Returned<br>Weight (g) |
|---|---|---|---|---|---|---|---|---|
| ××××× | ×××× | XXXXXXX | XXXXX | XXXXXXXX | XXXXXXXX | × × × | × | × |
| | | | ×××× | XXXXXXXXX | XXXXXXXXX | ××× | × × × × × | × |
| | | | ××××× | ×<br>×<br>×<br>×<br>× | ××××××××××××××××××××××××××××××××××××××× | × × × × × | × | × |
| ×××××× | ×××× | ××××××××××××××××××××××××××××××××××××××× | ××××× | ××××××××××××××××××××××××××××××××××××××× | xxxxxxxx | < ×××× | : | : |
| | | | ××××× | ××××××××××××××××××××××××××××××××××××××× | ×××××××××××××××××××××××××××××××××××××× | × × × × | × | × |

Listing sorted by Subject, Kit Number, Date Dispensed, Date Returned, and Tube ID.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.5.3: Study Drug Application Treatment Group (Page xx of yy)

| Subject | Age/Sex | Evaluable | Visit | Date/Time of Study<br>Drug Application | Study Drug<br>Applied in Clinic? | Pre-Dose<br>Weight (g) | Post-Dose<br>Weight (g) | Reason<br>Not Done |
|---|---|---|---|---|---|---|---|---|
| ××××× | xxxx | XXXXXXX | XXXXX<br>XXXXX | XXXXXTXXXX<br>XXXXXTXXXX<br>XXXXXTXXXX | ***<br>*** | × | x . x x x x x x x x x x x x x x x x x x | |
| ××××× | ×××× | ××××××× | ×××××<br>××××× | XXXXXTXXXX<br>XXXXXTXXXX<br>XXXXXTXXXX | ×××<br>××× | × × × × | × × × | ***** *** |
| ×<br>×<br>×<br>×<br>× | ×<br>×<br>×<br>× | ×××××× | ×××××<br>××××× | XXXXXTXXXX<br>XXXXXTXXXX<br>XXXXXTXXXX | ×××<br>××× | × × ×<br>× × × | × × × × × | |
| ××××× | ×××× | XXXXXXX | XXXXX<br>XXXXX<br>XXXXX | XXXXXTXXXX<br>XXXXXTXXXX<br>XXXXXTXXXX | × | x : | x : x x x x x x x x x x x x x x x x x x | XXX XXX XXX |

Listing sorted by Subject, Date/Time of Study Drug Application, Visit.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.5.4: Dosing Compliance Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | D: Date of First Dose<br>R: Date of Last Dose | Number of<br>Days of<br>Exposure | Calculated¹<br>Number of<br>Doses | Amount of<br>Study Drug<br>Used (g) | Maximum Number<br>of Missed<br>Consecutive Doses | Percent<br>Compliant | Compliant?² |
|---|---|---|---|---|---|---|---|
| S: XXXXXXX A: XXXXX E: XXXXXXXXX | D: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | × | × | ×<br>×<br>× | × | ×<br>× | × |
| S: xxxxxx A: xxxxx E: xxxxxxxxx | D: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | × | ×× | ×××× | × | ××× | × |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | D: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | × | ×× | XXXX | | XXXX | ××× |

<sup>1</sup> The total number of doses was calculated from the date of first dose and the date of last known dose minus the missed doses plus

additional dose deviations.

2 A subject was considered compliant with the dosing regimen if the subject applied at least 80% of the expected doses during the study drug application period and did not miss more than 3 consecutive doses.

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.5.5: Dosing Deviations Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Date of First Dose | Date of Dosing Deviation | Number of Doses Applied |
|---|---|---|---|---|---|
| xxxxxx | ×××× | xxxxxxxx | XXXXXXXX | XXXXXXXXX<br>XXXXXXXXXX<br>XXXXXXXXXX | * * * |
| XXXXX | ×××× | XXXXXXXX | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXXXX | ×× |
| ××××× | ×××× | XXXXXXXX | XXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ×× |

Listing sorted by Subject, and Date of Dosing Deviation.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.6.1: Investigator Global Assessment (IGA)
Treatment Group
(Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | Visit | Date of<br>Assessment | Whole Body<br>Investigator Global<br>Assessment Score | Does the Subject<br>have Intertriginous<br>Area involvement? | Intertriginous<br>Investigator Global<br>Assessment Score | Evaluator<br>Initials | Was<br>Dosing<br>Stopped |
|---|---|---|---|---|---|---|---|
| S: XXXXXX A: XXXXXXX E: XXXXXXXXX | SCREENING BASELINE WEEK 2 WEEK 4 WEEK 6 WEEK 8 WEEK 12 | XXXXXXXXX<br>XXXXXXXXXXX<br>XXXXXXXXXXXXXX | XXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXX<br>XXXXXXXX | × ×××××××××××××××××××××××××××××××××××× | × | × ×××××××××××××××××××××××××××××××××××× | ××× |
| S: XXXXXX A: XXXX E: XXXXXXXX | SCREENING BASELINE WEEK 2 WEEK 6 WEEK 8 WEEK 12 WEEK 12 | XXXXXXXXX<br>XXXXXXXXXX<br>XXXXXXXXXX<br>XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | * **** | | × ××××××<br> | ×× |

Listing sorted by Subject, Visit, and Date of Assessment.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.6.2: Body Surface Area (BSA) Involved with Psoriasis Treatment Group (Page xx of yy)

| Subject | Subject Age/Sex Eval | Eval | Visit | Date of Assessment | BSA <sup>1</sup> (%) | Evaluator Initials |
|---|---|---|---|---|---|---|
| xxxx xxxxxxx | ×××× | ×<br>×<br>×<br>×<br>×<br>×<br>× | ×××××××××××××××××××××××××××××××××××××× | ************************************** | *<br>* | * * * * * * * |
| ××××××× | ×××× | ××××××××××××××××××××××××××××××××××××××× | ×××××××××××××××××××××××××××××××××××××× | XXXXXXXXX<br>XXXXXXXXXX<br>XXXXXXXXXX | × | ××× × |
| | | | XXXX X XXXX X X X X X X X X X X X X X | XXXXXXXXX<br>XXXXXXXXXX | : | <br> |

## Listing sorted by Subject, Visit, Date of Assessment.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

<sup>&</sup>lt;sup>1</sup> Body Surface Area (BSA) involved with psoriasis (excluding the scalp, palms and soles). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.6.3: Psoriasis Area and Severity Index (PASI)
Treatment Group
(Page xx of yy)

| S: Subject<br>A: Age/Sex | V: Visit<br>D: Date<br>E: Evaluator | P: PASI | Affected Area | | Parameter Score | |
|---|---|---|---|---|---|---|
| E: Eval | Initials | M: mPASI | (% Involved) | Erythema (redness) | Induration (thickness) | Desquamation (scaling) |
| S: XXXXXX A: XXXXXX E: XXXXXXXX | V: SCREENING D: XXXXXXXXXX E: XXX | P: xx.x<br>M: x.x | Arms (xx-xx%) | XXXXXXX XXXXXX = X | xxxxxxx xxxxxxxx | XXXXXXXX - X |
| | | | Head (xx-xx%) Legs (xx-xx%) Trunk(x%) | X - XXXXXXX XXXXXXXX | X - XXXXXXX XXXXXXXX X X - X X X X X X | x - xxxxxxx xxxxxxx - x |
| | V: BASELINE D: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | P: x : x | Arms (x%) | × | × | × |
| | | | Head (x%)<br>Legs (xx-xx%)<br>Trunk(xx-xx%) | x - xxxxxx xxxxxxx x x x x x x x x x x | XXXXXXXX XXXXXXXX | × |
| | V: WEEK 2 D: xxxxxxxxxx E: xxx | P. X X X X X X X X X X X X X X X X X X X | | | | |
| | | | Trunk (xx-xx%) | XXXX - X | XXXX - X | ×××× - × |
| | V: WEEK 6 D: XXXXXXXXXX E: XXX | P: x.x<br>M: x.x | Arms (xx-xx%) | ×××× - × | xxxx - x | × |
| | | | Head (xx-xx%) Legs (x.x%) Trunk(xx-xx%) | XXXX - X<br>XXXX - X | × | XXXX - X<br>XXX - X<br>XXX - X |

Listing sorted by Subject, Visit, Date, and Affected Area. If < 10% of skin involved, present actual percent involved.

TOOL.AN.10-01.01 Statistical Analysis Plan Template
Listing 16.2.6.7: Columbia-Suicide Severity Rating Scale (C-SSRS) Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | V: Visit<br>D: Date | Question | Time Period | Response |
|---|---|---|---|---|
| S: xxxxxxx<br>A: xxxx | V: SCREENING<br>D: XXXXXXXXX | xxx xx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX<br>XXX XXXX |
| E: XXXXXXXX | | XXXXXXX XXXXXXX XXXXXXX XXXXXXX | ××××××× | XXX |
| | | | xxxxx x xxxxx | ×× |
| | | xxx xxxxxxx xxxxx xxxxxxx xxxxxxx xxx | ****** | × × × |
| | | XXXXXX XXXXXXXX XXXXXXX XXXXXX | XXXXXXX | XX |
| | | XX XXX XXXXXXX XXXXXX XXXX | XXXXX X XXXXX | XX |
| | | XXXXXX XXXXXXXX XXXXXXX | XXXXXXX | XXX |
| | | XXXX XXX XXXXXX | XXXXXX X XXXX | XX |
| | | XXXX XXXXXXX | XXXXXXX | × |
| | | | XXXXXX X XXXX | xxx xxx |
| | | XXX XXXX XXXX XXXX XXXX XXXX | XXXXXXXX | X XXX XXXX |
| | | | XXXXXX X XXXXX | XXX XXXX |
| | | XXXX XX XXXX XXXXX XXXXXXX | XXXXXXXX | x x xx xx xx xx |
| | | XXX XXXX XXXX XXXX XXXX | XXXXX X XXXXX | XXX XXXX |
| | | XXXXXXX XXXXXXX | XXXXXXXX | XX |
| | | | XXXXXX X XXXXX | XXX XXXX |
| | | XXX XXX XXX XXX XXX XXXXXXX | XXXXXXXX | XX |
| | | XXXXXXXXXX XXXXXXXX | XXXXX X XXXXX | XX |
| | | XXXXXXXX XXXXXXX | XXXXXXX | XXX XXXXX |
| | | | XXXXX X XXXXX | xxx xxxx |
| | V: BASELINE<br>D: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXX XX XXXXX | XXXXX XXXX | XX |
| | | XXX XXXXXXX XXXXXXXX XXXXXXXX XXXXXXX XXXX | XXXXX XXXXX XXXXX | XX<br>XX |

Listing sorted by Subject, Visit, Date, Question (in order in CRF), and Time Period (in order in CRF). All additional information (such as description, number of attempts) will be concatenated onto the response for the main question.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

## Number PHQ-8 Question

- How often during the past 2 weeks were you bothered by: Little interest or pleasure in doing things?  $\vdash$
- How often during the past 2 weeks were you bothered by: Feeling down, depressed, or hopeless?  $\sim$
- How often during the past 2 weeks were you bothered by: Trouble falling or staying asleep, or sleeping too much?  $\sim$
- How often during the past 2 weeks were you bothered by: Feeling tired or having little energy? 4
- How often during the past 2 weeks were you bothered by: Poor appetite or overeating? Ŋ
- How often during the past 2 weeks were you bothered by: Feeling bad about yourself, or that you are a failure, or have let yourself or your family down? 9
- Or How often during the past 2 weeks were you bothered by: Trouble concentrating on things, such as reading the newspaper watching television? \_
- How often during the past 2 weeks were you bothered by: Moving or speaking so slowly that other people could have noticed. Or the opposite being so fidgety or restless that you have been moving around a lot more than usual? ω

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by Question Number.

Listing 16.2.6.8.2: Patient Health Questionnaire Depression Scale (PHQ-8) Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date of<br>Assessment | г | 7 | т | 4 | 22 | 9 | | 80 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ××××× | ×××× | XXXXXXX | XXXXXXXX<br>XXXX X<br>XXXX X<br>XXXX X | XXXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXXX | × × × × × | × × × × × | × × × × × | × × × × × | ×××× | * * * * * | × × × × × | * * * * * |
| ××<br>××<br>××<br>×× | ×××× | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXXX<br>XXXXXXXX<br>XXXX XX<br>XXXX XX | ************************************** | × × × × × | × × × × × | × × × × × | × × × × × | × × × × × | * * * * * | × × × × × | * * * * * |
| ××<br>××<br>××<br>×× | ×××× | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXXX<br>XXXXXXXXX<br>XXXXX XXXXXXXXXXXX | XXXXXXXXXX<br>XXXXXXXXXX<br>XXXXXXXXXXXXXXXX | × × × × × | × × × × × | × × × × × | × × × × × | × × × × × | * * * * * | * * * * * | * * * * * |

Note: For all Questions: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day, ND = Not Done. SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

# Listing sorted by Subject, Visit, and Date of Assessment.

Listing 16.2.7.1.1: Investigator Local Tolerability Assessment Treatment Group (Page xx of yy)

| fects Locations where Other Effects are Present | XXXXXX XXXX XXXX XXXX XXXXX XXXXX XXXXX XXXX | XXXXXXX XXXX XXXX XXX | XXXX XXXXXXX XX | XXXX XXXXXXXX | XXXXX XXXX XXXXX XXXXX XXXXX XXXXX XXXXX | XXXX XXXXXXX XX |
|---|---|---|---|---|---|---|
| Other Effects<br>Present | , xxxxxx | xxx xxxxx | XXX XXXXX | ×<br>×<br>×<br>×<br>×<br>×<br>× | · ×××××× | xxx xxxxx |
| Other Effects<br>Assessed? | ××× | ××× | ××× | ××× | ××× | ××× |
| Dermal Response | ***** ******* | XXXX XXXXXXX XXXXXXX XXXXXXX XXXXXXX XXXX | ***** ******************************** | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ***** ******* | XXXX XXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXX |
| V: Visit<br>D: Date<br>E: Evaluator Initials | V: xxxxxxx<br>D: xxxxxxxxx xxxx<br>E: xxx | V: xxxxxxxx<br>D: xxxxxxxxx xxx<br>E: xxx | V: xxxxxxxx<br>D: xxxxxxxxx xxx<br>E: xxx | V: xxxxxxxx<br>D: xxxxxxxxx xxxx<br>E: xxx | V: xxxxxxxx<br>D: xxxxxxxxxx xxxx<br>E: xxx | V: XXXXXXX<br>D: XXXXXXXXX XXXX |
| S: Subject V A: Age/Sex D E: Eval | S: xxxxxx V A: xxxx D E: xxxxxxxx E | > □ □ | > □ 回 | > U E | S: xxxxxx V A: xxxx D E: xxxxxxxx E | > 11 |

Listing sorted by Subject, Visit, and Date.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.7.2.1: Unique Adverse Events Coded to MedDRA System Organ Classes and Preferred Terms (Page xx of yy)

| MedDRA System Organ Class | MedDRA Preferred Term | Adverse Event |
|---|---|---|
| ****** ******************************** | ×××××× | XXXXXX |
| | | XXXXXX |
| | XXXXXXXXXX | XXXXXXXXXX |
| XXX XXX XXXXXXXX XXX | XXXXXXX | XXXXXX |
| XXX XXXXXXXX | XXXXXX XXXXXXX | XXXXXXX XXXXXX |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXX | XXXXXXXXX XXXX |
| | XXXXXXXXX XXXXXXXXXXX | XXXXX XXXXXXXXXX XXXXXXXXXX |

Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing sorted by MedDRA System Organ Class, MedDRA Preferred Term, and Adverse Event.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.7.2.2: Treatment-Emergent Adverse Events Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | A: Adverse Event<br>C: System Organ Class<br>P: Preferred Term | F: Date of First Dose<br>S: Start Date (Day) <sup>1</sup><br>E: End Date (Day) <sup>1</sup> | G: Grade <sup>2</sup> R: Relationship to Study Drug O: Outcome | S: Serious Event? A: In Treatment Area? T: Action Taken with Study Drug E: Action Taken to Treat Event |
|---|---|---|---|---|
| S: XXXXXX A: XXXX E: XXXXXXXX | A: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | F: XXXXXXXXXX S: XXXXXXXXX XXXX E: XXXXXXXXXX XXXX | G: xxxx R: xxxxxxxxx O: xxxxxxxxxx | S: XX A: XXXX T: XXX E: XXXXXXXX |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxxx | A: XXXXXXXXXXXXXXXC: XXXXXXXXXXXXXXXXXXX | F: XXXXXXXXXX S: XXXXXXXXX XXXX E: XXXXXXXXX XXXX | G: xxxx R: xxxxxxxxxx O: xxxxxxxxxxx | S: xx A: xxxx T: xxx E: xxxxxxx |
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | A: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | F: XXXXXXXXXX S: XXXXXXXXXX XXXX E: XXXXXXXXXXXXXXXXXXX | G: xxxx<br>R: xxxxxxxxxx<br>O: xxxxxxxxxxx | S: xx<br>A: xx<br>T: xxx<br>E: xxxxxxx |

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death. Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.7.2.3: Serious Adverse Events Treatment Group (Page xx of yy)

| S: Subject<br>A: Age/Sex<br>E: Eval | A: Adverse Event<br>C: System Organ Class<br>P: Preferred Term | F: Date of First Dose<br>S: Start Date (Day) <sup>1</sup><br>E: End Date (Day) <sup>1</sup> | G: Grade <sup>2</sup><br>R: Relationship to<br>Study Drug<br>O: Outcome | S: Serious Evemt? A: In Treatment Area? T: Action Taken with Study Drug E: Action Taken to Treat Event |
|---|---|---|---|---|
| S: xxxxxx<br>A: xxxx<br>E: xxxxxxxx | A: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | F: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | G: xxxx<br>R: xxxxxxxx<br>O: xxxxxxxxx | S: xxx A: xxxx T: xxxx E: xxxxxxxx |
| S: XXXXXX A: XXXX E: XXXXXXXX | A: xxxxxxxxxxxxxxxxx C: xxxxxxxxxxxxxxxx | F: XXXXXXXXXX S: XXXXXXXXX XXXX E: XXXXXXXXX XXXX | G: xxxx R: xxxxxxxxx O: xxxxxxxxxx | S: xxx A: xxxx T: xxx E: xxxxxxxx |
| S: XXXXXX A: XXXX E: XXXXXXXX | A: xxxxxxxxxxxxxxxxx C: xxxxxxxxxxxxxxxx | F: XXXXXXXXXXX S: XXXXXXXXXXXXXXXXXXXXXX | G: xxxx<br>R: xxxxxxx<br>O: xxxxxxxxx | S: xxx A: xx T: xxx E: xxxxxxx |

Listing sorted by Subject, Start Date, End Date, and Adverse Event.

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death. Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.7.2.4: Subjects Who Permanently Discontinued Study Drug Due to Adverse Events or Exeprienced an Adverse Event Resulting in Death

Treatment Group (Page xx of yy)

| S: Start Date (Day) 1<br>E: End Date (Day) 1 | S: XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|
| Adverse Events G: Grade <sup>2</sup> R: Relationship to Study Drug A: Action Taken | G: xxxxx x R: xxxxxxxxx A: xxxxxxxxx xxxxxxxxxxxxxxx |
| Adverse Events A: Adverse Event Description R: Relationship to System Organ Class P: Preferred Term A: Action Taken | A: xxxxxxx xxx C: xxxxxxxx xxxx P: xxxxxxxx xxxx xxxxxxxx xxxxxxxxxx |
| R: Primary Reason for Study Completion/Discontinuation S: Date of Study Completion/Discontinuation (Day) 1 C: System Organ Class V: Last Visit Attended P: Preferred Term | R: xxxxxx xxxxx<br>S: xxxxxxxxx xxxx<br>V: xxxx x |
| S: Subject A: Age/Sex Completion/Discontin E: Eval S: Date of First Dose Completion/Discontin L: Date of Last Dose V: Last Visit Attended | S: xxxxxx |

<sup>&</sup>lt;sup>1</sup> Day is calculated as date - date of first dose for dates prior to first dose. Otherwise, day is calculated as date - date of first dose + 1 for dates on or after first dose.

<sup>&</sup>lt;sup>2</sup> Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life Threatening; Grade 5 = Death. Note: System Organ Class and Preferred Term map to the MedDRA dictionary (Version 21.1). SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE, TIME)

Listing 16.2.8.1: Urine Pregnancy Test Results Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date | Result |
|---|---|---|---|---|---|
| ××××× | ×<br>×<br>× | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXX<br>XXXX X<br>XXXX X<br>XXXX X | XXXXXXXXX<br>XXXXXXXXXX<br>XXXXXXXXXX | XXXXXXXX<br>XXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXX |
| ××××× | ××× | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXX<br>XXXX X<br>XXXX X<br>XXXX X<br>XXXX X | ************************************** | XXXXXXX<br>XXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXX |
| ×××××× | ×××× | ×<br>×<br>×<br>×<br>×<br>× | XXXXXXXXX<br>XXXXXXXX<br>XXXX X<br>XXXX X<br>XXXX X<br>XXXXXX | ************************************** | XXXXXXXX XXXXXXXX XXXXXXX XXXXXXX XXXX |

Listing sorted by Subject, Visit, and Date.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

| Subject | Age/Sex | Eval | V: Visit<br>D: Date/Time of ECG | ECG Parameter | Result (Units) | ECG Interpetation | Abnormal |
|---|---|---|---|---|---|---|---|
| XXXXXXXX | ×××× | ××××××× | V: xxxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx | XXXXXXXX<br>XXXXXXXXX<br>XXXXXXXXXX<br>XXXXXXX | XX XXXXX XXXX XXXX XXXX XXXX XXXX XXXX XXXX | ************************************** | ××× × |
| | | | V: XXXXXXXXX D: XXXX-XX-XXTXX:XX | X X X X X X X X X X X X X X X X X X X | X X X X X X X X X X X X X X X X X X X | | |
| XXXXXXX | ×××× | ××××××××××××××××××××××××××××××××××××××× | V: xxxxxxxxx<br>D: xxxx-xx-xxTxx:xx:xx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX XXXXX XXXX XXXX XXXX XXXX XXXX XXXX XXXX | *************************************** | |

Listing sorted by Subject, Visit, Date/Time, Category, and ECG Parameter.

TOOL.AN.10-01.01 Statistical Analysis Plan Template

Listing 16.2.8.3.1: Vital Signs Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date | Vital Sign | Result | Units |
|---|---|---|---|---|---|---|---|
| ××××× | ×××× | ××××××××××××××××××××××××××××××××××××××× | SCREENING | ××××××××××××××××××××××××××××××××××××××× | Temperature<br>Heart Rate<br>Systolic Blood Pressure<br>Diastolic Blood Pressure<br>Weight | ××××<br>×××<br>××××<br>×××× | ×××××××××××××××××××××××××××××××××××××× |
| | | | BASELINE | ××××××××××××××××××××××××××××××××××××××× | Temperature Heart Rate Systolic Blood Pressure Diastolic Blood Pressure Height | ×××× ××× ×××× | ×××××<br>××××<br>××××<br>××××<br>××××<br>×××× |
| | | | × ×××× | XXXXXXXXX | Temperature<br>Heart Rate<br>Systolic Blood Pressure<br>Diastolic Blood Pressure<br>Weight | X X X X X X X X X X X X X X X X X X X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | ×<br>×<br>×<br>×<br>×<br>× | XXXXXXXXX | Temperature<br>Heart Rate<br>Systolic Blood Pressure<br>Diastolic Blood Pressure<br>Weight | × | xxxxxxxx<br>xxxx<br>xxxx<br>xxxx |

Listing sorted by Subject, Visit, Date, and Vital Sign (in the order displayed in the CRF).

Listing 16.2.8.3.2: Weight Loss/Gain >5% Treatment Group (Page xx of yy)

| Subject | Age/Sex | Eval | Visit | Date | Weight (kg) | Baseline<br>Weight(kg) | Baseline % Change<br>Weight(kg) Weight(kg) from Baseline | Reason |
|---|---|---|---|---|---|---|---|---|
| XXXXX | ×××× | XXXXXXX | × ×××× | ××××××××× | XXX | ××× | ××× | ** *** |
| | | | X XXXX | XXXXXXXXX | ××× | ××× | ××× | ***** *** |

Listing sorted by Subject, Visit, Date.

TOOL.AN.10-01.01 Statistical Analysis Plan Template



### **Certificate Of Completion**

Envelope Id: CDEB1B02388C4970A7D23284343C98D6

Subject: Arcutis ARQ-151-202 Finalized SAP

Source Envelope:

Document Pages: 337 Signatures: 4 Initials: 0 Certificate Pages: 5

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed



### **Record Tracking**

Status: Original

10/22/2020 12:23:58 PM

Location: DocuSign



### Signature

### **Timestamp**

Sent: 10/22/2020 12:39:01 PM Viewed: 10/23/2020 3:36:38 PM Signed: 10/23/2020 7:58:10 PM



With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

### **Electronic Record and Signature Disclosure:**

Accepted: 10/23/2020 3:36:38 PM

ID: a7419f37-d2a5-45b2-904d-cfd5cf1ff84b

Sent: 10/23/2020 7:58:13 PM Viewed: 10/23/2020 8:14:07 PM Signed: 10/23/2020 8:14:29 PM



With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 10/23/2020 8:14:07 PM ID: 6ff260db-7ba0-4f4a-a0a7-0b3f069a889b Signer Events Signature

Sent: 10/23/2020 8:14:32 PM Viewed: 10/25/2020 9:59:44 PM Signed: 10/25/2020 10:00:38 PM

**Timestamp** 

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I am the author of this document

### Electronic Record and Signature Disclosure:

Not Offered via DocuSign



Sent: 10/25/2020 10:00:42 PM Viewed: 10/26/2020 7:41:01 AM Signed: 10/26/2020 7:42:02 AM

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I have reviewed this document

### Electronic Record and Signature Disclosure: Not Offered via DocuSign

| isclosure | |
|---|---|
| Status | Timestamps |
| Security Checked | 10/26/2020 7:42:02 AM |
| Security Checked | 10/26/2020 7:42:02 AM |
| Security Checked | 10/26/2020 7:41:01 AM |
| Hashed/Encrypted | 10/25/2020 10:00:42 PM |
| Status | Timestamps |
| Signature | Timestamp |
| Signature | Timestamp |
| Status | Timestamp |
| Status | Timestamp |
| Status | Timestamp |
| Status | Timestamp |
| Status | Timestamp |
| Signature | Timestamp |
| | Status Status Status Status Status Signature Signature Status Hashed/Encrypted Security Checked Security Checked Security Checked |

### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Abond CRO (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### **How to contact Abond CRO:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by phone call: 616-892-3704

To contact us by email send messages to: helpdesk@abondcro.com

### To advise Abond CRO of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at HelpDesk@abondcro.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

### To request paper copies from Abond CRO

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to jproos@abondcro.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

### To withdraw your consent with Abond CRO

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to helpdesk@abondcro.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Abond CRO as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Abond CRO during the course of your relationship with Abond CRO.